### PROTOCOL PS0008 AMENDMENT 2

BY A DOSE-BLIND MAINTENANCE

INCALMENT PERIOD TO EVALUATE THE EFFICACY AND

SAFETY OF BIMEKIZUMAB IN ADULT SUBJECTS WITH

MODERATE TO SEVERE CHRONIC PLAQUE PSORIAGE

PHASE A PHASE 3, MULTICENTER, RANDOMIZED, DOUBLE-BLIND STUDY WITH AN ACTIVE-CONTROLLED INITIAL TREATMENT TREATMENT PERIOD TO EVALUATE THE EFFICACY AND MODERATE TO SEVERE CHRONIC PLAQUE PSORIASIS EudraCT Number: 2016-003392-22 and any extension
IND Number: 128707

Sponsor:
UCB Biopharma SPDJ
A112

Allée de la Recherche 60

1070 Brussels

| Protocol/Amendment number | Date | Type of amendment |
|---------------------------|-------------|-------------------|
| Final Protocol | 15 Aug 2017 | Not applicable |
| Protocol Amendment 1 | 15 Oct 2017 | Not applicable |
| Protocol Amendment 2 | 06 Apr 2018 | Substantial |

### **Confidential Material**

### **Confidential**

This document is the property of UCB and may not – in full or in part – be passed on, reproduced, published, or otherwise used without the express permission of UCB.


## STUDY CONTACT INFORMATION

### **Sponsor**

UCB Biopharma SPRL

Allée de la Recherche 60

1070 Brussels

**BELGIUM** 

## **Sponsor Study Physician**

| Name: | Nancy Cross, MD |
|----------|-----------------------------------------------------------------|
| Address: | UCB Biosciences, 8010 Arco Corporation Drive, Raleigh, NC 27617 |
| Phone: | +1 919 767 1060 |
| Fax: | +1 919 767 2570 |

## **Clinical Project Manager**

| Name: | Petrina Wall |
|----------|-----------------------------------------------------------------|
| Address: | UCB Biosciences, 8010 Arco Corporation Drive, Raleigh, NC 27617 |
| Phone: | +1 919 767 2613 |
| Fax: | +1 919 767 2570 |

# Clinical Trial Biostatistician

| Name: | Maggie Wang |
|----------|-----------------------------------------------------------------|
| Address: | UCB Biosciences, 8010 Arco Corporation Drive, Raleigh, NC 27617 |
| Phone: | +1 919 767 2877 |
| Fax: US | +1 919 767 2570 |

# Clinical Monitoring Contract Research Organization

| Name: | PAREXEL International (IRL) Limited-Ireland |
|----------|-------------------------------------------------------------------|
| Address: | Ireland Limited at 70 Sir John Rogerson's Quay, Dublin 2, Ireland |
| Phone: | +353 (1) 477 3171 |
| Fax: | +353 (1) 477 3308 |


| Serious adverse event reporting (24h) | |
|---|---|
| Fax | Europe and Rest of the World: +32 2 386 24 21 |
| | USA and Canada: +1 800 880 6949 or +1 866 890 3175 |
| Email | Global: DS_ICT@ucb.com |

The accuracy taken to support any new area and a support and the support of the s


# **TABLE OF CONTENTS**

| LIS | T OF A | BBREVIATIONS | 10 |
|-----|----------------------|---------------------------------------|-----|
| 1 | SUMN | 1ARY | 14 |
| 2 | INTRO | DDUCTION | 15 |
| 2.1 | Psorias | sis | 15 |
| 2 | .1.1 | Global epidemiology of psoriasis | 15 |
| 2 | .1.2 | Current treatments for psoriasis | 16, |
| 2.2 | Bimek | izumab | 48 |
| 2 | 2.1 | Clinical | |
| | 2.2.1. | 1 Completed studies | 18 |
| | 2.2.1. | 2 Ongoing studies | |
| 2 | 2.2 | Nonclinical | 20 |
| 3 | STUD | Y OBJECTIVE(S) | 21 |
| 3.1 | Primar | y objective | 21 |
| 3.2 | Second | dary objectives | 21 |
| 3.3 | Other of | objectives | 21 |
| 4 | STUD | Y VARIABLES | 22 |
| 4.1 | Primar | y efficacy variable | 22 |
| 4.2 | Second | Clinical | 22 |
| 4 | .2.1 | Secondary efficacy variables | 22 |
| 4 | .2.2 | Secondary safety variables | 22 |
| 4.3 | Other v | variables | 22 |
| 4 | .3.1 | Other efficacy variables | 22 |
| 4 | 3.2 | Other safety variables | 24 |
| 4 | .3.3 | Pharmacokinetic variable | 24 |
| 4 | .3.4 | Pharmacogenomic variables | 24 |
| 4 | .3.5 | Immunological variable | 24 |
| 5 | STUD | Y DESIGN | 24 |
| 5.1 | | description | |
| 5.2 | Study | periods | 25 |
| 5 | 21 | Screening Period | |
| 5 | .2.2<br>.2.4<br>.2.5 | Double-blind Initial Treatment Period | 25 |
| 5 | .2.4 | Safety Follow-Up Period | 26 |
| Q5 | .2.5 | Premature End of Treatment | 26 |
| | | duration per subject | 27 |
| 5.4 | | d number of subjects and site(s) | |
| 5.5 | | pated regions and countries | |
| 5.6 | | ile of study assessments | |

| 5.7 | Schematic diagram | 33 |
|---|---|---|
| 5.8 | Rationale for study design and selection of dose | 34 |
| 5 | 5.8.1 Study design | 34 |
| 5 | 5.8.2 Dose selection | 34 |
| 6 | SELECTION AND WITHDRAWAL OF SUBJECTS | 34 |
| 6.1 | Inclusion criteria | 34 |
| 6.2 | Exclusion criteria | |
| 6.3 | Withdrawal criteria | 38100 |
| 6 | Potential drug-induced liver injury IMP discontinuation criteria | |
| 7 | STUDY TREATMENT(S) | 41 |
| 7.1 | Description of investigational medicinal product(s) | .xe41 |
| 7.2 | Treatment(s) to be administered | 42 |
| 7.3 | Packaging | 44 |
| 7.4 | Labeling | 44 |
| 7.5 | Handling and storage requirements | 44 |
| 7.6 | Drug accountability | 44 |
| 7.7 | Procedures for monitoring subject compliance | 45 |
| 7.8 | Concomitant medication(s)/treatment(s) | 45 |
| 7 | Withdrawal criteria 3.3.1 Potential drug-induced liver injury IMP discontinuation criteria STUDY TREATMENT(S) Description of investigational medicinal product(s) Treatment(s) to be administered Packaging Labeling Handling and storage requirements Drug accountability Procedures for monitoring subject compliance Concomitant medication(s)/treatment(s) 7.8.1 Permitted concomitant treatments (medications and therapies) 7.8.1.1 Topical medications | 45 |
| | 7.8.1.1 Topical medications | 45 |
| | 7.8.1.2 Other medications | 45 |
| 7 | 7.8.2 Prohibited concomitant treatments (medications and therapies) | 46 |
| | 7.8.2 Prohibited concomitant treatments (medications and therapies) | 47 |
| 7.9 | Blinding | 47 |
| 7 | Procedures for maintaining and breaking the treatment blind | 48 |
| | 7.9.1.1 Maintenance of IMP blind | 48 |
| | 7.9.1.2 Breaking the treatment blind in an emergency situation | 48 |
| 7.10 | 0 Randomization and numbering of subjects | 48 |
| 8 | STUDY PROCEDURES BY VISIT | 48 |
| 8.1 | Screening Visit (2 to 5 weeks) | 49 |
| 8.2 | Initial Treatment Period | 50 |
| | 3.2.1 Baseline Visit | 50 |
| 8 | 3.22 Week 1 (±3 days) | 51 |
| 8 | 2.2.4 Week 3 (±3 days) | 52 |
| 8 | 3.2.4 Week 4 (±3 days) | |
| 8 | 3.2.5 Week 5 and 7 (±3 days) | 53 |
| 8 | 3.2.6 Week 8 (±3 days) | 54 |
| 8 | 2.7.7 Week 9 and 11 (+3 days) | 55 |

| 8 | .2.8 | Week 12 (±3 days) | 55 |
|---|---|---|---|
| 8 | .2.9 | Week 13 and 15 (±3 days) | 56 |
| 8 | .2.10 | Week 16 (±3 days) | 56 |
| 8.3 | Dose-b | lind Maintenance Treatment Period | 57 |
| 8 | .3.1 | Week 17 and 19 (±3 days) | 57 |
| 8 | .3.2 | Week 20 (±3 days) | 58 |
| 8 | .3.3 | Week 21 and 23 (±3 days) | 59 |
| 8 | .3.4 | Week 24 (±3 days) | 59 <sup>10</sup> |
| 8 | .3.5 | Week 28 (±7 days) | 60 |
| 8 | .3.6 | Week 32 (±7 days) | 61 |
| 8 | .3.7 | Week 36 (±7 days) | 61 |
| 8 | .3.8 | Week 40 (±7 days) | 62 |
| 8 | .3.9 | Week 44 (±7 days) | 63 |
| 8 | .3.10 | Week 48 (±7 days) | 63 |
| 8 | .3.11 | Week 52 (±7 days) | 64 |
| 8 | .3.12 | Week 56 (±7 days) | 65 |
| 8.4 | Premat | ure End of Treatment Visit | 66 |
| 8.5 | Safety | Week 24 (±3 days) Week 28 (±7 days) Week 32 (±7 days) Week 36 (±7 days) Week 40 (±7 days) Week 44 (±7 days) Week 48 (±7 days) Week 52 (±7 days) Week 56 (±7 days) ure End of Treatment Visit Follow-Up Visit (20 weeks after final dose ±7 days) eduled Visit SSMENT OF EFFICACY sis Area and Severity Index gator's Global Assessment tology Life Quality Index | 67 |
| 8.6 | Unsche | eduled Visit | 67 |
| 9 | ASSES | SSMENT OF EFFICACY | 67 |
| 9.1 | Psorias | sis Area and Severity Index | 68 |
| 9.2 | Investi | gator's Global Assessment | 68 |
| 9.3 | Dermat | tology Life Quality Index | 69 |
| 9.4 | Patient | Health ()nectionnaire U a'U' | 6u |
| 9.5 | Scalp I | GAx | 69 |
| 9.6 | | | |
| 9.7 | pp-IGA | Quality of Life 5-Dimensions, 3-Level | <del>70</del> |
| 9.8 | Euro Q | uality of Life 5-Dimensions, 3-Level | 71 |
| 9.9 | Short F | Form 36 Item Health Survey | 71 |
| 9.10 | | Global Assessment of psoriasis | |
| 9.11 | Patient | Symptom Diary responses | 72 |
| 9.12 | e s <mark>PAS</mark> E | questionnaire | 72 |
| 9.13 | PGAD. | A for the arthritis visual analog scale | 72 |
| 9.14 | WPAI- | SHP V2.0 | 73 |
| 10 | ASSES | SSMENT OF PHARMACOKINETIC AND PHARMACOGENOMIC | |
| | | ABLE(S) | |
| | | acokinetic variables | 73 |
| 10.3 | Dharma | acogenomic variables | 73 |

| 11 | ASSE | SSMENT OF IMMUNOLOGICAL VARIABLE(S) | 74 |
|---|---|---|---|
| 12 | ASSE | SSMENT OF SAFETY | 74 |
| 12 | 1 Adver | rse events | 74 |
| | 12.1.1 | Definitions | 74 |
| | 12.1. | 1.1 Adverse event | 74 |
| | 12.1. | 1.2 Serious adverse event | 75 |
| | 12.1. | 1 | |
| | 12.1. | 1.4 Other safety topics of interest | |
| | 12.1.2 | Procedures for reporting and recording adverse events | 5. 76 |
| | 12.1. | 2.1 Description of adverse events | |
| | 12.1. | 2.2 Rule for repetition of an adverse event | 77 |
| | 12.1. | .2.3 Additional procedures for reporting serious adverse events | 77 |
| | 12.1.3 | Follow up of adverse events | 78 |
| | 12.1.4 | Pregnancy | 78 |
| | 12.1.5 | Sugnosted transmission of an intentious agent was a medicinal product | 1/0 |
| | 12.1.6 | Overdose of investigational medicinal product | 79 |
| | 12.1.7 | Overdose of investigational medicinal product | 79 |
| 12 | 2 Labora | atory measurements | 80 |
| | 12.2.1 | Evaluation of PDILI | 81 |
| | 12.2. | 11.1 Consultation with Medical Mountof and local nepatologist | |
| | 12.2. | | |
| | 12.2. | | 85 |
| | 12.2. | 1 | |
| 12 | 3 Other | safety measurements | |
| | 12.3.1 | Assessment and management of TB and TB risk factors | |
| | 12.3. | | |
| | 12.3. | .1.2 Chest x-ray for tuberculosis | |
| | 12.3. | ¥O 1 | |
| | 12.3. | . 010 | |
| | 12.3.2 | Pregnancy testing | |
| | | ∜ital signs | |
| | 12.3.4 | | |
| | 12.3.5 | Physical examination | |
| | 12.3.6 | Height and body weight | |
| | 12.3.7 | Assessment of suicidal ideation and behavior | |
| | | study measurements | |
| | 12.4.1 | Demographic information | 93 |
| | 1242 | Medical History | 93 |

| 12.4.3 Psoriasis History | 93 |
|---|---|
| 12.4.4 Data Monitoring and Adjudication Committees | 93 |
| 13 STUDY MANAGEMENT AND ADMINISTRATION | 94 |
| 13.1 Adherence to protocol | 94 |
| 13.2 Monitoring | 94 |
| 13.2.1 Definition of source data | 94 |
| 13.2.2 Source data verification | 95 |
| 13.3 Data handling | |
| 13.3.1 Case Report Form completion | |
| 13.3.2 Database entry and reconciliation | 95 |
| 13.3.3 Subject Screening and Enrollment log/Subject Identification Code list | 96 |
| 13.4 Termination of the study | 96 |
| 13.5 Archiving and data retention | 96 |
| 13.6 Audit and inspection | 96 |
| 13.7 Good Clinical Practice | 97 |
| 14 STATISTICS | 97 |
| 14.1 Definition of analysis sets | 97 |
| 14.2 General statistical considerations | 97 |
| 14.3 Planned efficacy analyses | 99 |
| 13.3.3 Subject Screening and Enrollment log/Subject Identification Code list2 | 99 |
| 14.3.1.1 Sensitivity analyses | 99 |
| 14.3.2 Other efficacy analyses | 100 |
| 14.3.2.1 Analysis of the secondary efficacy variables | 100 |
| 14.4 Subgroup analyses | |
| 14.5 Planned safety and other analyses | |
| 14.5.1 Safety analyses | |
| 14.5.2 Pharmacokinetic analyses | |
| 14.5.3 Immunogenicity analyses | |
| 14.6 Handling of protocol deviations | |
| 14.7 Handling of dropouts or missing data | 103 |
| 14.8 Planned interim analysis and data monitoring | |
| 14.9 Determination of sample size | |
| 15 ETHICS AND REGULATORY REQUIREMENTS | |
| 15.1 Informed consent | 105 |
| 15.2 Subject identification cards | |
| 15.3 Institutional Review Boards and Independent Ethics Committees | 106 |
| 15.4 Subject privacy. | 106 |

| 15.5 Protocol | amendments | 107 |
|---|---|---|
| 16 FINANC | CE, INSURANCE, AND PUBLICATION | 107 |
| 17 REFERI | ENCES | 107 |
| 18 APPENI | DICES | 110 |
| 18.1 Protocol | Amendment 1 | 110 |
| | Amendment 2 | |
| 19 DECLA | RATION AND SIGNATURE OF INVESTIGATOR | 189 |
| 20 SPONSO | OR DECLARATION | 190 |
| | | ons |
| | LIST OF TABLES | |
| Table 5–1: | Schedule of study assessments. | 28 |
| Table 7–1: | Dosing scheme | 43 |
| Table 7–2: | Prohibited psoriasis medications | 46 |
| Table 9–3: | LIST OF TABLES Schedule of study assessments. Dosing scheme. Prohibited psoriasis medications. Body areas for calculation of percent BSA for PASIO. | 68 |
| Table 9–4: | Five-point IGA | 69 |
| Table 9–5: | Scalp IGA | 70 |
| Table 9–6: | Five-point IGA Scalp IGA pp-IGA | 71 |
| Table 12.1: | Anticipated serious adverse events for the population of subjects with moderate to severe chronic plaque psoriasis | |
| Table 12–2: | Laboratory measurements | |
| Table 12–3: | Required investigations and follow-up for PDILI | |
| Table 12–4: | PDILI laboratory measurements | 86 |
| Table 12–5: | PDILI information to be collected | 87 |
| | LIST OF FIGURES | |
| Figure 5–1: | Schematic diagram of PS0008 | 33 |
| Figure 12-1: | Schematic diagram of TB test results and study eligibility | 90 |
| Figure 144: | Sequence of testing | 98 |

PS0008

### LIST OF ABBREVIATIONS

AE

**AESI** 

**ALP** 

**ALT** 

**AST** 

axSpA **AUC** 

BA

**BKZ Set BMI** 

BP

**BSA** 

cAMP

CAT

CDC

**CDMS** 

CI

**CMH CPM** 

**CPMP** 

**CRO** Contract Research Organization

Clinical Study Report **CSR** 

**CTCAE** Common Terminology Criteria for Adverse Events

CVcardiovascular

**DLOI** Dermatology Life Quality Index **DMC Data Monitoring Committee** 

**ECG** electrocardiogram

**eCRF** electronic Case Report Form

eC-SSRS electronic Columbia Suicide Severity Rating Scale

Electronic Data Capture

This document ePRO electronic Patient-Reported Outcome

EQ-5D-3L Euro-Quality of Life 5-Dimensions, 3-Levels

**Enrolled Set** ES

**FAS** Full Analysis Set

**FDA** Food and Drug Administration

**GCP** 

GeoMean

...cy virus
...ar **GMP HBcAb HBsAg HCP** 

**HCV HCV Ab** 

HIV

HLT

IΒ **IBD ICF** 

**ICH** 

**IEC** 

Ig

**IGA IGRA** 

IL

investigational medicinal product **IMP** 

Institutional Review Board **IRB IRT** interactive response technology

Intravenous iv

**LOCF** last observation carried forward

LTB latent tuberculosis

**LTBI** latent tuberculosis infection

mAb monoclonal antibody MAR missing at random

minimal clinically important difference

His documer. **MCMC** Markov-Chain Monte Carlo Mental Component Summary

MedDRA Medical Dictionary for Regulatory Activities MI multiple imputation

**MID** minimally important difference

**mNAPSI** Modified Nail Psoriasis Severity Index Score

NRI nonresponder imputation

**NSAID** nonsteroidal anti-inflammatory drug nontuberculous mycobacterium **NTMB** 

**PASE** Psoriatic Arthritis Screening and Evaluation

**PASI** Psoriasis Area and Severity Index **PCS** Physical Component Summary

PD pharmacodynamics PDE4 phosphodiesterase 4

**PDILI** potential drug-induced liver injury

**PEOT** Premature End of Treatment

PFS prefilled syringe

tion and any extensions of variations thereof. Patient's Global Assessment of Disease Activity **PGADA** 

Patient Health Questionnaire PHQ-9

PK pharmacokinetics

PK-PPS Pharmacokinetics Per-Protocol Set

palmoplantar Investigator's Global Assessment pp-IGA

Per-Protocol Set PPS

patient-reported outcome **PRO** 

PS Patient Safety psoriatic arthritis **PsA** 

**PSO Psoriasis** 

Q2W every 2 weeks Q4W every 4 weeks Q8W every 8 weeks QOL quality of life RS Randomized Set

serious adverse event statistical analysis plan

subcutaneous

scalp IGA scalp-specific IGA SD standard deviation


### 1 SUMMARY

PS0008 is a Phase 3, multicenter, randomized, double-blind, active-comparator-controlled, parallel-group study to evaluate the efficacy, safety, and pharmacokinetics (PK) of bimekizumab (also known as UCB4940) compared with adalimumab in adult subjects with moderate to severe chronic plaque psoriasis (PSO).

The study population consists of adult subjects (≥18 years of age) with a diagnosis of moderate to severe chronic plaque PSO (Baseline Psoriasis Area and Severity Index [PASI] ≥12 and body surface area [BSA] affected by PSO ≥10% and Investigator's Global Assessment [IGA] score ≥3 [on a 5-point scale]) who are candidates for adalimumab or for systemic PSO therapy and/or phototherapy.

Approximately 600 subjects will be screened in order to have a total of 450 subjects randomized in the study. For each subject, the study will last a maximum of 77 weeks and will consist of 4 periods, a Screening Period (2 to 5 weeks), a double-blind, active comparator-controlled Initial Treatment Period (16 weeks), a dose-blind Maintenance Treatment Period (40 weeks), and a Safety Follow-Up (SFU) Period (20 weeks after the final dose of the investigational medicinal product [IMP]). After completion of the 40-week Maintenance Treatment Period, eligible subjects will be allowed to enroll in an open-label study.

Eligible subjects will be randomized 1:1:1 to receive the following blinded IMP regimens subcutaneously (sc):

- Bimekizumab 320mg every 4 weeks (Q4W) administered throughout the study (150 subjects)
- Bimekizumab 320mg administered Q4W/every 8 weeks (Q8W) (ie, bimekizumab 320mg Q4W will be administered until Week 16, then bimekizumab 320mg Q8W from Week 16 through Week 52 (150 subjects)
- Adalimumab 80mg administered as an initial dose, followed by 40mg every 2 weeks (Q2W) starting 1 week after the initial dose (ie, adalimumab will be administered according to the labeling recommendations) until Week 24, then bimekizumab Q4W from Week 24 to Week 52 (150 subjects)

At Week 56, all subjects enrolling in the open-label study will undergo the Week 56 study assessments before receiving their first open-label study dose of IMP. All subjects not enrolling in the open-label study will have the Week 56 study assessments and will enter the 20-week SFU Period.

Subjects withdrawing early from the study will undergo the Premature End of Treatment (PEOT) Visit assessments and will enter the 20-week SFU Period.

The primary objective of the study is to compare the efficacy of bimekizumab administered sc for 16 weeks versus adalimumab in the treatment of subjects with moderate to severe chronic plaque PSO. The secondary objectives of the study are listed in Section 3.2.

The co-primary efficacy variables are the PASI90 response (defined as a subject that achieves 90% reduction from Baseline in the PASI score) at Week 16 and the IGA response (defined as


PS0008

Clear or Almost Clear with at least a 2-category improvement relative to Baseline) at Week 16. The secondary efficacy variables are listed in Section 4.2.1.

Safety variables to be assessed are adverse events (AEs), vital signs, electrocardiograms (ECGs), and measurements of laboratory parameters.

2 INTRODUCTION

2.1 Psoriasis

Psoriasis

Psoriasis is a common, chronic inflammatory disease characterized by a series changes in the skin: hyperplasia of epidermal keratinosyte infiltration of T lymphocytes pour he nather. the pathophysiology of PSO is not fully understood, the importance of T-cells and inflammatory cytokines has been demonstrated by the clinical benefit provided by therapies directed at these targets (Krueger and Ellis, 2005).

There are a variety of forms including plaque, guttate, inverse, pustular, and erythrodermic. Plaque PSO is the most common, comprising approximately 80% to 90% of all cases. Approximately 17% of those with PSO have moderate to severe disease (Kurd et al., 2008).

In addition to the impact on skin, PSO has a multitude of psychosocial and emotional effects on patients, including increased self-consciousness, frustration, fatigue, depression, and suicidal ideation. As a result, patients frequently report sleeping problems, difficulties at work, problems interacting with family members, disrupted leisure activities, and sexual difficulties (Dowlatshahi et al, 2014; Gottlieb, 2005; Mukhtar et al, 2004; Ortonne, 2004; Krueger et al, 2001).

A number of comorbidities have been associated with PSO, especially with more severe PSO. Psoriatic arthritis (PsA), cardiovascular (CV) disease, metabolic syndrome, chronic pulmonary disease, peptic ulcer disease, renal disease, and diabetes have all been demonstrated to have an increased prevalence in PSO patients (Yeung et al, 2013; Christophers et al, 2010; Gisondi et al, 2007; Gelfand et al, 2006).

### Global epidemiology of psoriasis 2.1.1

Psoriasis affects approximately 3% of the US adult population (Rachakonda et al, 2014; Kurd and Gelfand, 2009) and its onset can begin at any age (Augustin et al, 2010; Icen et al, 2009). The reported worldwide incidence and prevalence of PSO varies greatly depending on age, the disease, therefore reported estimates of the magnitude of this condition are likely weighted heavily by this subtype. Both the incidence and prevalence of PSO are higher amount. gender, ethnicity, and geography primarily due to genetic and environmental factors. Estimates of incidence and prevalence include all types of PSO. Plaque PSO is the most common form of heavily by this subtype. Both the incidence and prevalence of PSO are higher among Caucasians and those living in higher latitudes. Psoriasis affects approximately 2% to 4% of the population of western countries. Geographical differences are also influenced by case definition, study


design, and the definition of prevalence (Parisi et al, 2013; Langley et al, 2005; Raychaudhuri and Gross, 2000).

### 2.1.2 Current treatments for psoriasis

Therapy for patients with PSO varies according to the severity of disease. Limited or mild disease is often treated with topical therapies such as corticosteroids and vitamin D analogs. Patients with more severe disease are often treated with phototherapy, methotrexate, cyclosporine, the oral phosphodiesterase 4 (PDE4) inhibitor apremilast, or biologic agents, such as tumor necrosis factor (TNF) antagonists, interleukin (IL)-12/23 inhibitors, IL-23p19 inhibitors and IL-17A inhibitors. The effectiveness of TNF inhibitors in the treatment of PSO has been demonstrated in many Phase 3 clinical studies and has led to the approval of multiple TNF inhibitors for use in patients with moderate to severe PSO. Interleukin inhibitors approved for this indication include the IL-12/23 antagonist ustekinumab, the IL-23p19 antagonist guselkumab, the IL-17A inhibitors secukinumab and ixekizumab, and the IL-17 receptor antagonist brodalumab.

Standard therapies for PSO are listed below:

- Topical steroids (eg, triamcinolone, mometasone, clobetasol, betamethasone, hydrocortisone) are generally used as first-line treatment of PSO. High-strength steroids are typically reserved for use on the arms and legs. Areas such as the face and skin folds (axillary, inguinal regions, etc) are usually treated with a low potency steroid. Chronic use of topical steroids can lead to corticosteroid-related side effects and is generally discouraged.
- Vitamin D analogs (eg, calcipotriol and tacalcitol) are commonly used to treat mild to moderate PSO, and work best within the mild patients. They are safe but lack efficacy for more severe disease.
- Phototherapy is a frequent option for moderate to severe patients, but the inconvenience of multiple treatment visits and varying efficacy limits its use in the market.
- Methotrexate is a systemic immunosuppressant and is used in moderate to severe PSO patients. Toxicity concerns, particularly in older patients, are a major drawback.
- Cyclosporine is a systemic immunosuppressant used in patients with severe, recalcitrant, PSO who have failed at least one systemic therapy or in whom other systemic therapies are contraindicated. In recommended dosages cyclosporine can cause systemic hypertension and nephrotoxicity, therefore, renal function must be monitored during therapy.
- Apremilast is an oral small-molecule inhibitor of PDE4 that is also approved for treatment of adults with moderate to severe plaque PSO. Phosphodiesterase 4 inhibitors work intracellularly to modulate a network of proinflammatory and anti-inflammatory mediators. Phosphodiesterase 4 is a cyclic adenosine monophosphate (cAMP)-specific PDE and the dominant PDE in inflammatory cells. Phosphodiesterase 4 inhibition elevates intracellular cAMP levels, which in turn down-regulates the inflammatory response by modulating the expression of TNFα, IL-23, IL-17, and other inflammatory cytokines.
- Biologics, including TNFα inhibitors (adalimumab, etanercept, and infliximab), IL-12/23 inhibitors (ustekinumab), the IL-23p19 antagonist (guselkumab), the IL-17A inhibitors (secukinumab and ixekizumab), and the IL-17 receptor antagonist brodalumab are

Bimekizumab

the treatment options of choice for patients with moderate to severe plaque PSO who are candidates for systemic therapy or phototherapy. These products are injected sc or delivered via intravenous (iv) infusion. Different from the traditional systemic drugs that impact the entire immune system, biologics target specific parts of the immune system and offer reduced multi-organ toxicity and adverse effects associated with traditional treatments.

- TNFα inhibitors, while effective, come with boxed warnings including the risk of serious infections and reports of lymphoma and malignancy in children and adolescent patients. The efficacy of TNFα inhibitors in treating PSO is attributed to their inhibition of Th17-T cells.
- Ustekinumab has been approved in the US and the EU for the treatment of patients with moderate to severe plaque PSO who are candidates for phototherapy or systemic therapy. Ustekinumab is a human immunoglobulin (Ig) G1κ monoclonal antibody that binds with specificity to the p40 protein subunit used by both the IL-12 and IL-23 cytokines, naturally occurring cytokines that are involved in inflammatory and immune responses, such as natural killer cell activation and CD4+ T-cell differentiation and activation.
- Secukinumab and ixekizumab have been approved in the US and the EU for the treatment of moderate to severe plaque PSO in adult patients who are candidates for systemic therapy or phototherapy. Secukinumab is a human IgG1 monoclonal antibody that selectively binds to the interleukin-17A (IL-17A) cytokine and inhibits its interaction with the IL-17 receptor. Ixekizumab is a humanized IgG4 monoclonal antibody that selectively binds with the interleukin 17A (IL-17A) cytokine and inhibits its interaction with the IL-17 receptor. IL-17A is a naturally occurring cytokine that is involved in normal inflammatory and immune responses. Both drugs inhibit the release of proinflammatory cytokines and chemokines.
- Guselkumab has been approved in the US and the EU for the treatment of adult patients with moderate to severe plaque PSO who are candidates for systemic therapy or phototherapy. It is a human monoclonal IgG1λ antibody that selectively binds to the p19 subunit of interleukin 23 (IL-23) and inhibits its interaction with the IL-23 receptor. IL-23 is a naturally occurring cytokine that is involved in normal inflammatory and immune responses. Guselkumab inhibits the release of proinflammatory cytokines and chemokines.
- Brodalumab has been approved in the US for the treatment of moderate to severe plaque psoriasis in adult patients who are candidates for systemic therapy or phototherapy and have failed to respond or have lost response to other systemic therapies. In the EU, brodalumab is indicated for the treatment of moderate to severe plaque PSO in adult patients who are candidates for systemic therapy. Brodalumab is a human monoclonal IgG2 antibody that selectively binds to human IL-17RA and inhibits its interactions with cytokines IL-17A, IL-17F, IL-17C, IL-17A/F heterodimer and IL-25. Blocking IL 17RA inhibits IL-17 cytokine-induced responses including the release of proinflammatory cytokines and chemokines. Brodalumab has a black box warning regarding suicidal ideation and behavior.

### 2.2 Bimekizumab

Bimekizumab (UCB4940) is an engineered, humanized full-length monoclonal antibody (mAb) of immunoglobulin (Ig) G1 subclass of approximately 150,000 Daltons which is expressed in a genetically engineered Chinese hamster ovary cell line. Bimekizumab has high affinity for human IL-17A and human IL-17F and selectively and potently inhibits the activity of both isoforms in vitro. Interleukin-17A and IL-17F are key proinflammatory cytokines believed to play important roles in autoimmune and inflammatory diseases. Bimekizumab is being developed for the treatment of patients with inflammatory diseases such as PsA, PSO, and axial spondyloarthritis (axSpA).

While anti-IL-17A antibodies have demonstrated efficacy in patients with PSO PsA ankylosing spondylitis, as yet, no therapeutic approach activity of both II 17A

While anti-IL-17A antibodies have demonstrated efficacy in patients with PSO, PsA, and ankylosing spondylitis, as yet, no therapeutic approach selectively and potently inhibits the activity of both IL-17A and IL-17F isoforms in vitro. Bimekizumab is an engineered, humanized, full-length IgG1 mAb which has been designed to inhibit the activity of IL-17A and IL-17F subtypes of IL-17. This property makes bimekizumab distinct from the other IL-17-targeting agents like secukinumab and ixekizumab (selective anti-IL-17-A mAb), or brodalumab (anti-IL-17 receptor mAb).

Overexpression of IL-17A, IL-17C, and IL-17F in lesion tissue suggests that broader IL-17 blockade may be more beneficial in the treatment of plaque PSO. However, blocking all IL-17 isoforms (including the IL-17E isoform, also known as IL-25) may not be the optimal approach. The role of IL-25 in PSO and other IL-17 mediated diseases has not been well established, however it has been suggested that IL-25 may play a beneficial role in inflammatory conditions associated with type 1 T helper (Th-1) mediated immune responses, such as PSO (as opposed to type 2 T helper [Th-2) mediated) (Valizadeh et al., 2015). Thus, it can be hypothesized that inhibition of both IL-17A and IL-17F is associated with additional benefits in PSO compared to the selective IL-17A inhibition or a broader IL-17 blockade.

### 2.2.1 Clinical

### 2.2.1.1 Completed studies

Five clinical studies of bimekizumab have been completed: UP0008 in 39 subjects with mild to moderate plaque PSO, RA0124 in 30 healthy volunteers, PA0007 in 53 subjects with PsA, UP0031 in 12 healthy volunteers, and UP0042 in 48 healthy volunteers.

UP0008 was a Phase ¶, single ascending dose study in adults with mild to moderate PSO affecting ≤5% BSA. In this blinded study, single doses of up to 640mg (approximately 8mg/kg in an 80kg adult) were evaluated without any safety concerns. A total of 26 subjects with PSO with less than 5% of body surface involvement were treated with a range of single iv doses from 8 to 640mg. There were no clinically relevant safety findings identified at any dose and all doses were well tolerated. The pre-specified exploratory assessment of disease activity showed clinically relevant and statistically significant improvements at the higher doses studied.

RA0124 was a Phase 1, open-label, parallel-group, single-dose study in healthy subjects. The primary objective of this study was to determine the absolute bioavailability (BA) of single sc doses of bimekizumab (80mg and 160mg). The secondary objectives were to evaluate the dose proportionality of bimekizumab 80mg and 160mg sc, and to evaluate the safety and tolerability of these sc doses and 160mg given by iv infusion. In RA0124, the absolute BA was similar for


Bimekizumab

the 2 doses tested (0.656 and 0.631 for the bimekizumab 80mg and 160mg sc doses, respectively). The PK of bimekizumab was linear in the tested dose range and the median  $t_{1/2}$ following sc administration was similar to that following iv administration (27.81 days and

a rnase 1b, proof of concept, randomized, placebo concept, randomized, randomized, placebo concept, randomized, placebo concept, randomized, placebo concept, randomized, randomized, randomiz and any extension

- 160mg loading dose followed by 80mg at Weeks 3 and 6
- 240mg loading dose followed by 160mg at Weeks 3 and 6
- 560mg loading dose followed by 320mg at Weeks 3 and 6

The results of this study demonstrated that all doses of bimekizumab were well tolerated and there were no unexpected clinically relevant safety findings.

Infections (mostly nasopharyngitis) were the most commonly reported events in both the active treatment and the placebo group. None of the infections were considered serious or required treatment with antibiotics. Two subjects in the active treatment group experienced 1 local candida infection each (oropharhyngitis and vulvovaginitis, respectively) that were non-serious and resolved with topical therapy. There was a potential reduction in mean neutrophil count in the active treatment group, although this drop was not clinically relevant and a clear relationship with dose or time was not evident. Some increases in liver function tests were reported, but none had a convincing relationship to exposure to IMP. The exploratory analysis showed clinically relevant improvement in activity of PsA and in skin involvement in those subjects with concomitant active psoriatic lesions.

UP0031 was a Phase 1, open-label, parallel-group, randomized, single-dose study to evaluate the BA, PK, and tolerability of 2 different formulations of bimekizumab in healthy subjects. Subjects receiving Formulation A (histidine-based) were administered two 1mL injections of 80mg each of bimekizumab and subjects receiving Formulation B ) were administered a single injection of bimekizumab 160mg given as a 1mL injection. Six subjects were randomized to each bimekizumab formulation. The geometric means (GeoMeans) for area under the curve (AUC) were similar between bimekizumab 2x80mg and 1x160mg groups and the relative BA for Formulation B vs Formulation A was 96.1% (95% confidence interval [CI]: 72.7%, 127.0%). Administration of the 2 formulations of bimekizumab used in this study identified no new safety experienced by more than 1 subject in either treatment group was injection site pain (5 subjects [83.3%] and 3 subjects [50.0%] in the 2x80mg and 1x160mg groups, respectively. The frequently reported TEAE considered related to the subjects [50.0%] in the 2x80mg and 1x160mg groups, respectively. frequently reported TEAE considered related to the IMP was injection site pain, experienced by 5 subjects [83.3%] and 3 subjects [50.0%] in the 2x80mg and 1x160mg groups, respectively. There were no clinically significant laboratory values reported in the study.

UP0042 was a randomized double-blind, placebo-controlled, single-dose, parallel-group study to evaluate the safety, tolerability, and PK of bimekizumab administered as an sc injection to Eighs of Variations thereof Japanese and Caucasian healthy subjects. This study demonstrated that the PK profiles following single administration of 80mg, 160mg, and 320mg with an sc injection were dose proportional with a linear elimination in both Japanese and Caucasian subjects and that the PK profiles of Japanese and Caucasian subjects were considered to be generally similar. A single dose of bimekizumab (80mg, 160mg, or 320mg) administered as an sc injection was generally safe and well tolerated in healthy Japanese and Caucasian subjects and no major differences in safety findings were observed between Japanese and Caucasian subjects.

#### 2.2.1.2 **Ongoing studies**

Four additional studies of bimekizumab in the treatment of PSO are ongoing.

- PS0010 is a Phase 2b, double-blind, placebo-controlled, dose ranging study to evaluate the safety, efficacy, PK, and pharmacodynamics (PD) of bimekizumab in adult subjects with moderate to severe chronic plaque PSO.
- PS0011 is a long-term extension study for subjects who completed PS0010 to assess the long-term safety, tolerability, and efficacy of bimekizumab.
- PS0016 is a Phase 2a, subject-blind, Investigator-blind study to evaluate the time course of PD response, safety, and PK of bimekizumab in adult subjects with moderate to severe chronic plaque PSO.
- PS0018 is a long-term extension study for eligible subjects from PS0016 to assess the safety, tolerability, and efficacy of bimekizumab.

Bimekizumab is also being evaluated in the treatment of other indications (eg, PsA, axSpA, hidradenitis suppurativa). Additional information on the clinical data for bimekizumab is available in the current version of the Investigator's Brochure (IB).

#### 2.2.2 **Nonclinical**

Parallel inhibition of IL-17A and IL-17F has been shown to be efficacious in a variety of animal models of inflammatory disease. Intravenously administered bimekizumab was well tolerated in repeat dose toxicology studies in Cynomolgus monkeys with a no adverse effect level of 200mg/kg/week. The findings of note in toxicity studies were diarrhea related to infectious enteritis (observed in the single dose study) and asymptomatic mild colonic ulceration in a proportion of animals (in the repeat dose study); this latter finding was not associated with hematology abnormalities. Data suggest that bimekizumab has induced primary lesions to the mucosa associated lymphoid tissue via a pharmacologically-related mechanism. In a second repeat-dose study, none of the minor apoptosis/necrosis findings observed in gut associated lymph nodes were revealed. In animals given the highest dose of bimekizumab in the study (20mg/kg/week), a slightly higher number of protozoa (Balantidium coli) was observed in the secum and colon as compared to the control animals and low dose animals. Therefore, gut associated lymph node lesions observed in the first study are considered to be accidental and/or linked to exaggerated pharmacology and proliferation of Balantidium coli and is considered the consequence of a change in local mucosal immunity. To date, similar findings have not been seen in studies in humans.

Additional information on the nonclinical data for bimekizumab is available in the current version of the IB.

## 3 STUDY OBJECTIVE(S)

### 3.1 Primary objective

The primary objective of the study is to compare the efficacy of bimekizumab administered sc for 16 weeks versus adalimumab in the treatment of subjects with moderate to severe chronic plaque PSO.

### 3.2 Secondary objectives

The secondary objectives of the study are to:

- Evaluate the efficacy of bimekizumab compared to adalimumab after 4, 16, and 24 weeks of treatment
- Evaluate the efficacy of bimekizumab compared to adalimumab at achieving complete clearance (PASI100) after 16 weeks and 24 weeks of treatment
- Assess the maintenance of efficacy of bimekizumab dosing Q4W versus Q8W at Week 56
- Assess TEAEs, SAEs, and TEAEs leading to withdrawal adjusted by duration of subject exposure to study treatment

### 3.3 Other objectives

The other objectives of the study are to demonstrate the effects of bimekizumab on aspects of the disease:

- Assess the maintenance of efficacy of bimekizumab dosing Q4W versus Q8W during the Maintenance Treatment Period
- Assess the efficacy of bimekizumab over time
- Assess the change of skin-related quality of life (QOL)
- Assess the change of general health-related QOL
- Assess the change in hail PSO over time in subjects with nail PSO at Baseline
- Assess the change in scalp PSO over time in subjects with scalp PSO at Baseline
- Assess the change in palmoplantar PSO over time in subjects with palmoplantar PSO at Baseline
- Assess the symptoms of PsA as measured by the Psoriatic Arthritis Screening and Evaluation (PASE) questionnaire
- Assess the change of patient-reported joint symptoms in subjects with PsA at Baseline
- Assess the change in symptoms of PSO as reported by subjects using the Patient Symptom Diary (all items) through Week 24
- Assess depression
- Assess the PK of bimekizumab

- Assess the immunogenicity of bimekizumab
- Assess work productivity
- isions or variations thereof. Assess the effect of bimekizumab on gene and protein expression, and explore the relationship between genomic, genetic, and proteomic biomarkers and disease biology, drug treatment and inflammatory and immune responses (from consenting subjects who agree to participate in the biomarker substudy)
- Assess the safety and tolerability of bimekizumab

#### 4 STUDY VARIABLES

#### 4.1 Primary efficacy variable

The co-primary efficacy variables are the PASI90 response (defined as a subject that achieves 90% reduction from Baseline in the PASI score) at Week 16 and the IGA response (defined as Clear or Almost Clear with at least a 2-category improvement relative to Baseline) at Week 16.

#### 4.2 Secondary variables

#### 4.2.1 Secondary efficacy variables

The secondary efficacy variables are:

- PASI90 response at Week 24
- IGA response (Clear or Almost Clear with at least 2-category improvement relative to Baseline) at Week 24
- PASI75 response at Week 4
- PASI100 response at Week 16 and 2
- PASI90 response at Week 56
- IGA response at Week 56

#### 4.2.2 Secondary safety variables

- TEAEs adjusted by duration of subject exposure to study treatment
- SAEs adjusted by duration of subject exposure to study treatment
- TEAEs leading to withdrawal adjusted by duration of subject exposure to study treatment

#### 4.3 **⊘Other variables**

The other variables are listed below and will be evaluated according to the planned assessments Table 5–1.

### 423.1 Other efficacy variables

The other efficacy variables are listed below and will be evaluated according to the planned assessments Table 5–1. This excludes the time points for the primary and secondary variables specified above in Section 4.1 and Section 4.2.1, respectively.

Change from Baseline variables evaluated are relative to the Baseline (first dose) Visit. In addition, for subjects who start with adalimumab and switch treatment at the Week 24 Visit, , or variations thereof change from Baseline variables during the Maintenance Treatment Period may be evaluated relative to both the Baseline (first dose) Visit and the Week 24 Visit. For simplicity, "change from Baseline" is used below for all such variables. Greater detail on the definition of Baseline for different summaries will be provided in the Statistical Analysis Plan (SAP). Unless otherwise stated PASI responder rates will be calculated relative to the Baseline Visit (first dose).

Bimekizumab

The other efficacy variables are:

- PASI50, PASI75, PASI90, and PASI100 response
- Time to PASI50, PASI75, PASI90, and PASI100 response during the Initial Treatment Period
- Absolute and percent change from Baseline in PASI score
- IGA response (Clear)
- IGA response (Clear or Almost Clear with at least 2-category improvement relative to Baseline)
- Shift from Baseline in IGA score
- Absolute and percent change from Baseline in the BSA affected by PSO
- Absolute and percent change from Baseline in the product of IGA and BSA (IGAxBSA)
- Change from Baseline in the Dermatology Life Quality Index (DLQI)
- Percent of subjects achieving a DLQI total score of 0 or 1
- Percentage of subjects achieving a minimal clinically important difference (MCID) (improvement from Baseline of 4 or more) in the DLQI
- Change from Baseline in Patient's Global Assessment of Disease Activity (PGADA) for the arthritis visual analog scale (VAS) in subjects with PsA as defined by PASE score at Baseline
- Change from Baseline in Patient Global Assessment of PSO score
- Change from Baseline in the Patient Symptom Diary responses
- Scalp-specific Investigator's Global Assessment (scalp IGA) response (Clear or Almost Clear) for subjects with scalp PSO at Baseline
- Change from Baseline in modified Nail Psoriasis Severity Index (mNAPSI) score for subjects with nail PSO at Baseline
- Palmoplantar Investigator's Global Assessment (pp-IGA) response (Clear or Almost Clear) for subjects with palmoplantar PSO at Baseline
- Change from Baseline in the PASE questionnaire scores (function score, symptom score, and total score)
- Shift from Baseline in PASE score suggestive of PsA (<47 versus ≥47)

- Change from Baseline in Short Form 36-item Health Survey (SF-36) Physical Component Summary (PCS) score, and Mental Component Summary (MCS) score, and individual domains

- Lagrand baseline in Patient Health Questionnaire-9 (PHQ-9) scores

  Change from Baseline in Work Productivity and Activity Impairment Questionnaire-specific health problem (WPAI-SHP) V2.0 adapted to PSO scores

  Other safety variables

  ety variables to be assessed are: and any extensions of

### 4.3.2

Safety variables to be assessed are:

- Severity and frequency of AEs
- Change from Baseline in vital signs
- ECG results
- Change from Baseline in clinical laboratory values (chemistry, hematology, and urinalysis)

Physical examination findings considered clinically significant changes since the physical examination at the Screening Visit will be recorded as AEs

#### Pharmacokinetic variable 4.3.3

The PK variable is the plasma concentration of bimekizumab.

### Pharmacogenomic variables 4.3.4

Additional blood samples will be collected from subjects who consent to participate in the substudy at specific time points and stored at -80°C for up to 20 years.

Genomic, genetic, epigenetic, proteins, and metabolite biomarkers may be measured to evaluate the relationship with response to treatment with bimekizumab, PSO disease biology, and inflammatory and immune response processes. The nature and format of these tentative substudy analyses will be determined when the results of the main study are made available.

The candidate exploratory variables are the blood or blood derivative (eg., serum) concentrations of cytokines and chemokines of relevance to IL-17A/F signaling pathway and PSO biology. Additional variables may include but will not be limited to serum complement concentrations.

### ,,⊘lĭmmunological variable 4.3.5

The immunological variable is the anti-bimekizumab antibody level prior to and following IMP.

## STUDY DESIGN

## **Study description**

PS0008 is a Phase 3, multicenter study consisting of a 16-week, randomized, double-blind, parallel-group, active-comparator-controlled Initial Treatment Period followed by a 40-week, Maintenance Treatment Period to evaluate the efficacy and safety of bimekizumab in adult subjects with moderate to severe chronic plaque PSO. To be eligible to participate in this study, subjects must be adults with a diagnosis of moderate to severe PSO (Baseline PASI ≥12 and BSA affected by PSO  $\geq$ 10% and IGA score  $\geq$ 3 [on a 5-point scale]) who are candidates for systemic PSO therapy and/or phototherapy. Adalimumab will be administered per the local label.

Study periods

This study will include 4 periods, a Screening Period (2 to 5 weeks), an Initial Treatment Period (16 weeks), a Maintenance Treatment Period (40 weeks), and a SFU Period (20 weeks after the final dose of IMP). After completion of the Maintenance Treatment Period be allowed to enroll in an open-label study of the PS0000 GPT. have the PS0008 SFU Visit.

#### 5.2.1 Screening Period

The Screening Period will last 2 weeks, but can be extended up to a total of 5 weeks in cases where a laboratory assessment needs to be repeated or to allow washout of prohibited medications. During this time, eligible subjects will be informed about the study and sign the Informed Consent Form (ICF), laboratory data (hematology, urine, and biochemistry tests) will be obtained, and the doses of medications used to treat PsA, will be verified as stable. The Screening Period will also enable washout of any medications not permitted for use during the study. Subjects who require prophylaxis for latent tuberculosis (LTB) infection must be on treatment for at least 8 weeks prior to their first dose of IMP. These subjects may be rescreened once they have completed the first 8 weeks of prophylaxis treatment.

One rescreening may be allowed after consultation with the Medical Monitor.

The assessments to be performed at the Screening Visit are presented in Table 5–1.

#### 5.2.2 **Double-blind Initial Treatment Period**

During the active-controlled 16-week initial Treatment Period, approximately 450 subjects will be randomized 1:1:1 to receive the following blinded IMP regimens:

- Bimekizumab 320mg administered Q4W throughout the study (150 subjects)
- Bimekizumab 320mg administered Q4W until Week 16 (150 subjects)
- Adalimumab 80mg administered as an initial dose, followed by 40mg Q2W starting 1 week after the initial dose (ie, adalimumab will be administered according to the labeling recommendations) until Week 24 (150 subjects)

Investigational medicinal products will be administered in the clinic by sc injection at the time points specified in the schedule of study assessments (Table 5–1).

The active comparator-controlled The efficacy of 1. Subjects will be followed in a double-blind fashion. Subjects may receive placebo injections at certain visits in order to blind the IMP. The assessments to be performed at each Initial

The active comparator-controlled Initial Treatment Period will be used to demonstrate the efficacy of bimekizumab versus adalimumab. Efficacy of bimekizumab versus adalimumab will be measured at Week 16 because it was the time point for the primary endpoint in prior pivotal studies of adalimumab in PSO where efficacy was demonstrated.

**UCB** 

Subjects withdrawing early from the study will undergo the PEOT Visit assessments and will enter the SFU Period. Subjects withdrawing early from the study will not be eligible for inclusion in the open-label study.

#### 5.2.3 **Dose-blind Maintenance Treatment Period**

After the 16-week Initial Treatment Period, subjects will enter the 40-week Maintenance Treatment Period. Treatment during the Maintenance Treatment Period will start at Week 16 and subjects will return to the clinic Q4W or Q8W through Week 56. The IMP will be administered in the clinic by sc injection at the time points specified in the schedule of study assessments (Table 5–1). Treatment during the Maintenance Treatment Period will be based on initial treatment per the following:

- Subjects in the bimekizumab 320mg Q4W treatment arm will continue to receive bimekizumab 320mg Q4W.
- Subjects in the bimekizumab 320mg Q4W/Q8W treatment arm will receive bimekizumab Q8W from Week 16 through Week 52.
- Subjects in the adalimumab treatment arm will receive bimekizumab 320mg Q4W from Week 24 to Week 52.

Subjects may receive placebo injections at certain visits in order to blind the IMP (see Section 7.2).

At the end of the Maintenance Treatment Period, all subjects enrolling in the open-label study will, after signing a new ICF, undergo the Week 56 study assessments and then receive their first dose of bimekizumab in the open-label study. All subjects not enrolling in the open-label study will have the Week 56 study assessments and will enter the SFU Period.

The assessments to be performed at each visit of the Maintenance Treatment Period are presented in Table 5–1.

#### Safety Follow-Up Period 5.2.4

All subjects not continuing in the open-label study, including those withdrawn from IMP, will have a SFU Visit 20 weeks after their final dose of IMP.

The assessments for the SFU Visit are presented in in Table 5–1.

#### 5.2.5 **Premature End of Treatment**

Subjects withdrawing early from the study will undergo the PEOT Visit assessments (see Section 8.4) and will enter the SFU Period.

#### 5.3 Study duration per subject

For each subject, the study will last a maximum of up to 77 weeks, as follows:

Safety Follow-Up Period: a SFU Visit is planned 20 weeks after the final dose of IMP (for subjects not enrolling in the open-label study)

er the 40-week Maintenance Treatment Period, subjects will be all el study, in which case subjects will undergo de r first open-label IMP 1 After the 40-week Maintenance Treatment Period, subjects will be allowed to enroll in an openlabel study, in which case subjects will undergo the Week 56 study assessments before receiving their first open-label IMP dose. The SFU Visit will not be required for subjects who enroll in the open-label study.

The end of the study is defined as the date of the last visit of the last subject in the study.

#### Planned number of subjects and site(s) 5.4

Approximately 600 subjects will be screened in order to have 450 subjects randomized in the study. There will be approximately 150 subjects per treatment arm. The planned number of study sites is approximately 100. Every eligible subject who signs an ICF will be expected to be randomized.

#### 5.5 Anticipated regions and countries

The regions planned for study conduct are North America, Western Europe, Central/Eastern Europe, and Asia/Australia, with possible extension to other regions and countries.

### 5.6 Schedule of study assessments

The schedule of study assessments for all subjects enrolled in the study is presented in andy and support and the used to support and the support and t Table 5–1. At each visit, all study assessments should be performed prior to administration of



 Table 5–1:
 Schedule of study assessments

| Clinical Study Prot | | | | | | | | | | | | | | | | | | | | | | | PS00 | _ |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Table 5–1: S Visit <sup>a</sup> / Week | Double-blind Initial Treatment Period (weeks after first dose) Dose-blind Maintenance Treatment Period (weeks after first dose) | | | | | | | | | | | | | | t Per | iod | | W56/PEOT | SET IS | | | | | |
| Protocol<br>activity | | Baseline (first dose) | 1 | 3 | 4 | 5,<br>7 | 8 | 9,<br>11 | 12 | 13,<br>15 | 16 | 17,<br>19 | 20 | 21, 23 | 242 | 40 | 32 | 36 | 40 | 44 | 48 | 52 | 56 | |
| Informed consent <sup>c</sup> | X | | | | | | | | | | | | | ijo | | | | | | | | $X^{d}$ | | |
| Inclusion/exclusion | X | X | | | | | | | | | | 7 | Slic | | | | | | | | | | | |
| Urine drug screen | X | | | | | | | | | | 0 | 2 | 3% | | | | | | | | | | X | |
| Demographic data | X | | | | | | | | | | ) , 19 | ijo | | | | | | | | | | | | |
| Psoriasis history | X | | | | | | | | | C, 's | Office | | | | | | | | | | | | | |
| Significant past<br>medical history and<br>concomitant<br>diseases | X | Xe | | | | | | < | ZED! | Oan | | | | | | | | | | | | | | |
| Physical examination <sup>f,g</sup> | X | X | | | | | | 11/1/2 | X | | | | | | X | | | X | | | X | | X | X |
| Height | | X | | | | | XO | | | | | | | | | | | | | | | | | |
| Body weight | | X | | | | 10, | 0, | | X | | | | | | X | | | X | | | X | | X | |
| Vital signs <sup>h</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Hematology and biochemistry | X | X | X | X | SAS I | | X | | X | | X | | X | | X | X | X | | X | | X | | X | X |
| Urinalysis | X | X | | be, | | | | | | | X | | | | X | | X | | X | | X | | X | X |
| ECG | X | | 2170 | | | | | | X | | | | | | X | | | X | | | X | | X | |
| Pregnancy testing <sup>i</sup> | X | X C | 3 | | X | | X | | X | | X | | X | | X | X | X | X | X | X | X | X | X | X |

 Table 5–1:
 Schedule of study assessments

| UCB<br>Clinical Study Prot | CB Inical Study Protocol Bimekizumab able 5–1: Schedule of study assessments | | | | | | | | | | | | | | | , S | 06 A | Apr 20<br>PS00 | 18<br>08 | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Table 5–1: | ble 5–1: Schedule of study assessments | | | | | | | | | | | | | | | | | | .6 | ailail | 0, | | | |
| Visit <sup>a</sup> /<br>Week | Screening | | | | nitial<br>rst dos | | ment | Perio | d | | | Dose-blind Maintenance Treatment Period (weeks after first dose) | | | | | | | | | | | | SFU |
| Protocol<br>activity | | Baseline (first dose) | 1 | 3 | 4 | 5,<br>7 | 8 | 9,<br>11 | 12 | 13,<br>15 | 16 | 17,<br>19 | 20 | 21, 23 | 24 | 40 | 32 | 36 | 40 | 44 | 48 | 52 | 56 | |
| Hepatitis B and C testing <sup>j</sup> | X | | | | | | | | | | | | · · · C | dilor | | | | | | | | | | |
| HIV testingk | X | | | | | | | | | | | 24 0 | 166 | | | | | | | | | | | |
| Chest x-ray <sup>l</sup> | X | | | | | | | | | | S | ijon | | | | | | | | | | | | |
| IGRA Tuberculosis<br>test | X | | | | | | | | | | 01/19 | | | | | | | | | | | X | | |
| Tuberculosis questionnaire | X | X | | | | | | | XOP | dani | | | | | X | | | X | | | X | | X | X |
| Blood sample for<br>bimekizumab<br>plasma<br>concentrations <sup>m</sup> | | X | X | X | X | | X | 1108 | X | | X | | X | | X | | | X | | | X | | X | X |
| Blood sample for anti-bimekizumab antibodies <sup>m</sup> | | X | | | X | a ( | OK O | | X | | X | | X | | X | | | X | | | X | | X | X |
| Blood sample<br>genomic,<br>proteomic, and<br>metabolomics, and<br>candidate<br>biomarker<br>analyses <sup>c,m</sup> | | X | X | , oe u | edic | SUR | X | | X | | X | | | | | | | | | | | | X | |

Table 5–1: Schedule of study assessments

| Clinical Study Pro Table 5–1: | | | e of | stud | v ass | sessr | nent | | | | | | | | | | | | | | | | | _ |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit <sup>a</sup> /<br>Week | Screening | | ıble-b | olind I | nitial | Treat | | | d | | | Dose-blind Maintenance Treatment Period (weeks after first dose) | | | | | | | | | | | | |
| Protocol<br>activity | | Baseline<br>(first dose) | 1 | 3 | 4 | 5,<br>7 | 8 | 9,<br>11 | 12 | 13,<br>15 | 16 | 17,<br>19 | 20 | 21, 23 | 240 | 70 | 32 | 36 | 40 | 44 | 48 | 52 | 56 | SFU |
| Blood sample<br>genetic/epigenetic<br>analyses <sup>c,m</sup> | | X | | | | | | | | | | 1 | oolic | atilot | | | | | | | | | X | |
| PASI | X | X | X | X | X | | X | | X | | XO | | Χ | | X | X | X | X | X | X | X | X | X | X |
| IGA | X | X | X | X | X | | X | | X | / | X | ijo, | X | | X | X | X | X | X | X | X | X | X | X |
| Percentage of BSA | X | X | X | X | X | | X | | X | C. | A | | X | | X | X | X | X | X | X | X | X | X | X |
| DLQI | | X | X | X | X | | X | | X | Sil | X | | X | | X | | X | | X | | X | | X | |
| PHQ-9 | X | X | | | X | | X | < | X | (9) | X | | X | | X | X | X | X | X | X | X | X | X | |
| eC-SSRS | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Patient Symptom<br>Diary (daily) | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | | | | | | | | | |
| scalp IGA | | X | X <sup>n</sup> | Xn | Xn | | X'n | | Xn | | Xn | | Xn | | Xn | | Xn | | Xn | | Xn | | Xn | |
| mNAPSI | | X | | | Xº | SUR | Xº | | Xº | | Xº | | Xº | | Xº | | Xº | | Xº | | Xº | | Xº | |
| pp-IGA | | X | | | X <sup>p</sup> . | ) | Xp | | Xp | | Xp | | Xp | | Xp | | X <sup>p</sup> | | Xp | | Xp | | Xp | |
| EQ-5D-3L | | X | | | X | | X | | X | | X | | | | X | | | | X | | | | X | |
| SF-36 | | X | | Pe | X | | X | | X | | X | | | | X | | | | X | | | | X | |
| Patient global<br>assessment of<br>psoriasis <sup>q</sup> | | . 0 | SINIC | | | | | | | | | | | | X | | X | | X | | X | | X | |

Table 5–1: Schedule of study assessments

| Visit <sup>a</sup> /<br>Week | Screening | Double-blind Initial Treatment Period (weeks after first dose) | | | | | | | | | | | | Dose-blind Maintenance Treatment Period (weeks after first dose) | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Protocol activity | | Baseline (first dose) | 1 | 3 | 4 | 5,<br>7 | 8 | 9,<br>11 | 12 | 13,<br>15 | 16 | 17,<br>19 | 20 | 21, 23 | 240 | 28 | 32 | 36 | 40 | 44 | 48 | 52 | 56 | |
| PASE | | X | | | | | | | | | | | | ijO) | | | | | | | | | X | |
| PGADA <sup>r</sup> | | X | | | X | | | | X | | X | 7 | olic | | X | | X | | X | | X | | X | |
| WPAI-SHP V2.0 | | X | | | | | | | | | X | | 36, | | X | | | | X | | | | X | |
| Concomitant medication | X | X | X | X | X | X | X | X | X | X | X<br>X | iX) | X | X | X | X | X | X | X | X | X | X | X | X |
| Adverse events | X | X | X | X | X | X | X | X | X | X | Ø | X | X | X | X | X | X | X | X | X | X | X | X | X |
| IRT <sup>s</sup> | X | X | X | X | X | X | X | X | XO V | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Bimekizumab,<br>adalimumab, or<br>placebo<br>administration <sup>s</sup> | | X | X | X | X | X | X | X | X | X | X | Х | X | X | X | X | X | X | X | X | X | X | | |

BSA=Body Surface Area; CV=cardiovascular; DLQI=Dermatology Life Quality Index; ECG=electrocardiogram; eCRF=electronic Case Report Form; eC-SSRS=electronic Columbia Suicide Severity Rating Scale; EQ-5D-3L=Euro-Quality of Life 5-Dimensions 3 Levels; GI=gastrointestinal; HCV=hepatitis C virus; HIV=human immunodeficiency virus; ICF=Informed Consent Form; IGA=Investigator's Global Assessment; IGRA=interferon-gamma release assay; IMP=investigational medicinal product; IRT=interactive response technology; mNAPSI=Modified Nail Psoriasis Severity Index Score; PASE=Psoriatic Arthritis Screening and Evaluation; PASI=psoriasis area severity index; PEOT=Premature End of Treatment Visit; PGADA=Patient Global Assessment of Disease Activity; PHQ-9=Patient Health Questionnaire-9; pp-IGA=palmoplantar Investigator's Global Assessment; PsA=psoriatic arthritis; SF-36=Short Form 36-item Health Survey; SFU=Safety Follow-Up; scalp IGA=scalp-specific Investigator's Global Assessment; TB=tuberculosis; WPAI-SHP=Work Productivity and Activity Impairment Questionnaire-specific health problem

<sup>&</sup>lt;sup>a</sup> Visit windows of ±3 days from the first dose to the Week 24 visit. Visit windows of ±7 days from the Week 28 visit to the Week 52 visit. The SFU Visit window is ±7 days from final dose.

<sup>&</sup>lt;sup>b</sup> The SFU Visit will occur 20 weeks after the final dose for subjects who do not enroll in the open-label study.

<sup>&</sup>lt;sup>c</sup> All genomic, proteomic, and metabolomics samples will be stored at -80°C at the central biorepository for up to 20 years.

<sup>&</sup>lt;sup>d</sup> A separate ICF is required to be completed for the open-label study.

<sup>&</sup>lt;sup>e</sup> Ensure no significant changes in medical history.

### Table 5-1: Schedule of study assessments

| Visit <sup>a</sup> /<br>Week | Screening | Double-blind Initial Treatment Period (weeks after first dose) | | | | | | | | | | | Dose-blind Maintenance Treatment Period (weeks after first dose) | | | | | | | | | | SFU <sup>5</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Protocol activity | | Baseline<br>(first dose) | 1 | 3 | 4 | 5,<br>7 | 8 | 9,<br>11 | 12 | 13,<br>15 | 16 | 17,<br>19 | 20 | 21, 23 | 240 28 | 32 | 36 | 40 | 44 | 48 | 52 | 56 | |

- <sup>f</sup> Includes evaluation of signs and symptoms of active TB and risk for exposure to TB.
- <sup>g</sup> The physical examination will be performed as per Section 12.3.5.
- h Vital signs (sitting systolic and diastolic blood pressure, pulse rate, and body temperature) are to be measured prior to blood sampling, and prior to dosing, where applicable.
- i Pregnancy testing will consist of serum testing at the Screening. The pregnancy test will be urine at all other visits.
- Subjects who have evidence of or test positive for hepatitis B by any of the following criteria: 1) positive for hepatitis B surface antigen (HBsAg+); 2) positive for anti-hepatitis B core antibody (HBcAb+) are excluded. A positive test for HCV is defined as: 1) positive for hepatitis C antibody (anti-HCV Ab), and 2) positive via a confirmatory test for HCV (for example, HCV polymerase chain reaction) are also excluded. Subjects will also be tested for anti-hepatitis B surface antibody.
- <sup>k</sup> The HIV test results will not be recorded in the eCRF.
- <sup>1</sup> Screening chest x-ray must occur within 3 months prior to Screening Visit.
- <sup>m</sup> All blood samples taken prior to dosing.
- <sup>n</sup> The scalp IGA will only be assessed for those subjects with scalp involvement (scalp IGA score >0) at Baseline.
- <sup>o</sup> The mNAPSI will be assessed only in subjects with nail involvement (mNAPSI score >0) at Baseline.
- <sup>p</sup> The pp-IGA will only be assessed in subjects with palmoplantar involvement (pp-IGA score >0) at Baseline.
- <sup>q</sup> The Patient Global Assessment of psoriasis will be performed as part of the patient symptoms diary on a weekly basis from Screening through the Initial Treatment Period at the specified clinic visits. During the Maintenance Treatment Period this assessment will be completed at the specified clinic visits.
- The PGADA is assessed for all subjects at Baseline At all subsequent visits, the PGADA is only for subjects with PsA at Baseline (defined as a past medical history of PsA or PASE ≥47).
- s IMP administration is based on randomization. The dosing window is ±3 days relative to the scheduled dosing visit through Week 24. The dosing window is ±7 days from Week 28 through the end of the study.

### 96 Apr 2018 PS0008

## 5.7 Schematic diagram

The study schematic diagram for PS0008 is presented in Figure 5–1.

Figure 5-1: Schematic diagram of PS0008



IGA=Investigator's Global Assessment; IMP=investigational medicinal product; N=number; PASI=Psoriasis Area and Severity Index; Q4W=every 4 weeks; Q8W=every 8 weeks; SFU=Safety Follow-Up

Note: Refer to Section 5.2.2 for treatments during the Initial Treatment Period and to Section 5.2.3 for treatments during the Maintenance Treatment Period.

Note: At Week 28 and all following visits, subjects on continuous treatment with the same IMP for at least 12 weeks with a persistent IGA score ≥3 over at least a 4-week period are defined as nonresponders and should discontinue IMP.

### 5.8 Rationale for study design and selection of dose

### 5.8.1 Study design

A randomized, active-controlled study design has been selected to demonstrate efficacy and safety of bimekizumab for regulatory approval. The study population will include adults with moderate to severe chronic plaque PSO and allow subjects who have received previous biologic treatment as well as those who are biologic treatment naïve. The primary efficacy outcome measures (based on PASI and IGA) and other efficacy assessments included in this study are consistent with those used for other PSO studies and are considered appropriate for establishing efficacy of bimekizumab. An Initial Treatment Period of 16 weeks will be used to demonstrate the efficacy of bimekizumab compared with adalimumab. The study duration extends beyond the Initial Treatment Period (to 56 weeks) to allow for collection of long-term safety and efficacy data.

At Week 24, subjects on adalimumab treatment are re-allocated to treatment with bimekizumab 320mg Q4W. This allows for a controlled evaluation of the safety and efficacy of switching from a product with one mechanism of action to another, which is known to occur in clinical practice due to either loss of response or access. In a recent PSO study in which subjects were switched from adalimumab to a treatment with a different mechanism of action, there was no evidence of an increased safety risk following the switch without washout (Reich et al, 2017).

### 5.8.2 Dose selection

Bimekizumab doses ranging from 64mg to 480mg were evaluated in the Phase 2b multicenter, randomized, double-blind, placebo-controlled, parallel-group, dose-ranging study PS0010. Bimekizumab 320mg was found to have an acceptable safety profile, only required 2 injections per treatment administration, and achieved significant PASI responses at Week 12 (summarized in the IB). Furthermore, data from the Phase 2a multicenter, randomized, subject-blind, Investigator-blind study PS0016 and PK/PD modeling in this PSO population indicates improved responses through Week 16. Therefore, a bimekizumab dose of 320mg (Q4W initial and Q4W or Q8W maintenance) was selected for this study.

# 6 SELECTION AND WITHDRAWAL OF SUBJECTS

## 6.1 Inclusion criteria

To be eligible to participate in this study, all of the following criteria must be met at Screening and at the Baseline Visit:

- 1. Subject has provided informed consent.
- 2. Subject is considered reliable and capable of adhering to the protocol (eg, able to understand and complete diaries), visit schedule, or medication intake according to the judgment of the Investigator.
- 3. Male or female at least 18 years of age.
- 4. Chronic plaque PSO for at least 6 months prior to the Screening Visit.
- 5. PASI ≥12 and BSA affected by PSO ≥10% and IGA score ≥3 on a 5-point scale.
- 6a. Subject is a candidate for systemic PSO therapy and/or phototherapy.


- 7. Subject must be considered, in the opinion of the Investigator, to be a suitable candidate for treatment with adalimumab per regional labeling and has no contraindications to receive adalimumab as per the local label.
- 8. Female subjects must be:
  - Postmenopausal. Menopause is defined as 12 consecutive months of amenorrhea, for which there is no other obvious pathological or physiological cause.
  - Permanently sterilized (eg, tubal occlusion, hysterectomy, bilateral salpingectomy).
  - Or, if of childbearing potential (and engaged in sexual activity that could result in procreation), must be willing to use a highly effective method of contraception throughout the duration of the study until 20 weeks after last administration of MMP, and have a negative pregnancy test at Visit 1 (Screening) and immediately prior to first dose. The following methods are considered highly effective when used consistently and correctly:
    - o Combined (estrogen and progestogen) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, or transdermal)
    - o Progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable).

    - Intrauterine hormone-releasing system
      Vasectomised partner

    - vasectomised partier.
       Abstinence as a form of birth control is generally not allowed in the study unless abstinence is in accordance with a subject's preferred and common lifestyle. Study personnel must confirm the continued use of abstinence is still in accordance with the subject's lifestyle at regular intervals during the study.
- 9. Subject agrees not to change their usual sun exposure during the course of the study and to use ultraviolet A/ultraviolet B sunscreens if unavoidable exposure occurs.

#### 6.2 **Exclusion criteria**

Subjects are not permitted to enroll in the study if any of the following criteria are met:

- 1. Female subject who is breastfeeding, pregnant, or plans to become pregnant during the study or within 20 weeks following the final dose of IMP.
- 2. Subject has previously participated in a bimekizumab clinical study who received at least 1 dose of the IMP (including placebo).
- 3a Subject is currently participating in another study of a medication (systemic) under investigation. Subject must be washed out of the medication for 12 weeks or at least 5 halflives prior to the Baseline Visit, whichever is greater.
- 4a. Subject is currently participating in another study of a topical medication under investigation. Subject must be washed out of the medication for 4 weeks prior to the Baseline Visit.

- 5a. Subject is currently, or was within the 4 weeks prior to the Baseline Visit, participating in another study of a medical device under investigation.
- 6. Subject has a known hypersensitivity to any excipients of bimekizumab or adalimumab.
- , variations thereof 7. Subject has a form of PSO other than chronic plaque-type (eg, pustular, erythrodermic and guttate PSO, or drug-induced PSO).
- 8. Subject has an active infection or history of infection(s) as follows:
  - Any active infection (except common cold) within 14 days prior to Baseline.
  - A serious infection, defined as requiring hospitalization or iv anti-infective(s) within 2 months prior to the Baseline Visit.
  - A history of opportunistic, recurrent or chronic infections that, in the opinion of the Investigator, might cause this study to be detrimental to the subject. Opportunistic infections are infections caused by uncommon pathogens (eg, pneumocystis jirovicii, cryptococcosis) or unusually severe infections caused by common pathogens (eg, cytomegalovirus, herpes zoster).
- 9. Subject has concurrent acute or chronic viral hepatitis B or C or Ruman immunodeficiency virus (HIV) infection. Subjects who have evidence of, or tested positive for hepatitis B or hepatitis C are excluded. A positive test for the hepatitis Byirus is defined as: 1) positive for hepatitis B surface antigen (HBsAg+) or 2) positive for anti-hepatitis B core antibody (HBcAb+). A positive test for the hepatitis C virus (HCV) is defined as: 1) positive for hepatitis C antibody (anti-HCV Ab) and 2) positive via a confirmatory test for HCV (for example, HCV polymerase chain reaction).
- 10. Subject has received any live (includes attenuated) vaccination within the 8 weeks prior to the Baseline visit (eg., inactivated influenza and pneumococcal vaccines are allowed but nasal influenza vaccination is not permitted).
- 11. Subject has received Bacillus Calmette-Guerin vaccinations within 1 year prior to the Baseline Visit.
- 12. Subject has known tuberculosis (TB) infection, is at high risk of acquiring TB infection, or has current or history of nontuberculous mycobacterium (NTMB) infection. A subject with LTB (a positive interferon-gamma release assay [IGRA] and diagnosis confirmed by TB specialist) may be rescreened once and enrolled after receiving at least 8 weeks of appropriate LTB infection therapy and if no evidence of therapy-related hepatotoxicity has occurred prior to the first injection (alanine aminotransferase [ALT]/aspartate aminotransferase [AST] remain  $\leq 3$  times upper limit of normal [ULN]).
  - Subject has a past history of active TB involving any organ system unless adequately treated according to World Health Organization/Centers for Disease Control (CDC) therapeutic guidance and proven to be fully recovered upon consult with a TB specialist.
  - Refer to Section 12.3.1 for details on determining full TB exclusion criteria.
- 13. Subject has a history of a lymphoproliferative disorder including lymphoma or current signs and symptoms suggestive of lymphoproliferative disease.
- 14a. Subject has any active malignancy or history of malignancy within 5 years prior to the Screening Visit EXCEPT treated and considered cured cutaneous squamous or basal cell carcinoma, or in situ cervical cancer.
- 15. Subject has a diagnosis of inflammatory conditions other than PSO or PsA, including but not limited to rheumatoid arthritis, sarcoidosis, or systemic lupus erythematosus. Subjects with a diagnosis of Crohn's disease or ulcerative colitis are allowed as long as they have no active symptomatic disease at Screening or Baseline.
- 16. Subject has had major surgery (including joint surgery) within the 3 months prior to the Baseline Visit, or has planned major surgery within 6 months after entering the study.
- 17a. Subject has any systemic disease (ie, cardiovascular, neurological, renal, liver, metabolic, gastrointestinal, hematological, immunological, etc.) considered by the Investigator to be uncontrolled, unstable, or likely to progress to a clinically significant degree during the course of the study.
- 18. Subject has had myocardial infarction or stroke within the 6 months prior to the Screening Visit.
- 19. Subject has laboratory abnormalities at Screening, including any of the following:
  - a. ≥3.0x ULN of any of the following: ALT, AST, alkaline phosphatase (ALP); or >ULN total bilirubin (≥1.5xULN total bilirubin if known Gilbert's syndrome)
  - b. White blood cell (WBC) count  $< 3.00 \times 10^3 / \mu L$
  - c. Absolute neutrophil count <1.5x10<sup>3</sup>/µL
  - d. Lymphocyte count <500 cells/μL
  - e. Hemoglobin < 8.5g/dL
  - f. Any other laboratory abnormality, which, in the opinion of the Investigator, will prevent the subject from completing the study or will interfere with the interpretation of the study results

Individual screening tests for which the results are in error, borderline, or indeterminate for inclusion in the study can be repeated once for confirmation during the Screening Period. Upon retesting, subjects whose results remain outside this threshold should not be randomized.

- 20. Subject has any other condition, including medical or psychiatric, which, in the Investigator's judgment, would make the subject unsuitable for inclusion in the study.
- 21. Subject has had previous exposure to adalimumab.
- 22. Criterion deleted
- 23. Subject has experienced primary failure (no response within 12 weeks) to 1 or more IL-17 biologic response modifier (eg, brodalumab, ixekizumab, secukinumab) OR more than 1 biologic response modifier other than an IL-17.
- 24. Subject is taking PsA medications other than stable doses (ie, stable for at least 1 week prior to the Screening Visit) of nonsteroidal anti-inflammatory drugs (NSAIDs) or analgesics (see Section 7.8.1.2).

- 25. Subject has a history of chronic alcohol or drug abuse within 6 months prior to Screening as evaluated by the Investigator based on medical history, site interview, and/or results of the specified urine drug screen.
- 26. Presence of active suicidal ideation, or positive suicide behavior using the "Screening" version of the electronic Columbia Suicide Severity Rating Scale (eC-SSRS) and with either of the following criteria:
- History of a suicide attempt within the 5 years prior to the Screening Visit. Subjects with a history of a suicide attempt more than 5 years ago should be evaluated by a mental healthcare practitioner (HCP) before enrolling into the study.

  Suicidal ideation in the past are response.
  - response ("Yes") to either Question 4 or Question 5 of the "Screening" version of the eC-SSRS.
- 27a. Subject has presence of moderately severe major depression or severe major depression, indicated by a score of >15 using the screening PHO-9. Medication used to treat depression should be stable for 8 weeks prior to Baseline.
- 28. Subject is a member of Investigator site personnel directly affidiated with this study and/or their immediate families. Immediate family is defined as a spouse, parent, child, or sibling, whether biological or legally adopted.
- 29. Subject is a UCB employee or employee of third-party organizations involved in the study.
- 30. Subject is taking or has taken prohibited psoriasis medications without meeting the mandatory washout period relative to the Baseline Visit (Table 7–2).

### Withdrawal criteria 6.3

Subjects are free to withdraw from the study at any time, without prejudice to their continued care. Subjects who withdraw from the study should complete the PEOT Visit (see Section 8.4).

Subjects should be withdrawn from the study and will be encouraged to come back for the SFU visit 20 weeks after final dose of IMP if the subject withdraws his/her consent or the Sponsor or a regulatory agency requests withdrawal of the subject.

A subject should be withdrawn from IMP and will be asked to come back for the SFU visit 20 weeks after final dose of IMP if any of the following events occur:

- 1. Subject develops an illness that in the opinion of the Investigator would interfere with his/her continued participation if the risk of continuing IMP outweighs the potential benefit.
- 2. Subject develops erythrodermic, guttate, or pustular form of PSO.
- Criterion deleted
- 4. Subject is noncompliant with the study procedures or medications in the opinion of the Investigator.
- 5. Subject uses prohibited concomitant medications, with the exception of topicals, as defined in this protocol (Section 7.8.2), that may present a risk to the safety of the subject or the integrity of the study data, in the opinion of the Investigator and/or the Medical Monitor.

- 6. Subject has a clinical laboratory value meeting any of the following criteria:
  - a. Hepatotoxicity as described in Section 6.3.1

Absolute lymphocyte count <0.2x10³/μL

Subjects may remain in the study if the result is transient. A retest is required within 1 to 2 weeks at a scheduled or unscheduled visit. If the repeat absolute neutrophil count or absolute lymphocyte count is still below the allowable values, the subject must be repeat absolute neutrophil count or absolute lymphocyte may continue in the

- 7. The subject experiences a severe AE, an SAE, or a clinically significant change in a laboratory value that, in the opinion of the Investigator, merits the discontinuation of the IMP and appropriate measures being taken.
- 8. At Week 28 and all following visits, subjects on continuous treatment with the same IMP for at least 12 weeks with a persistent IGA score  $\geq 3$  over at least a 4-week period are defined as nonresponders and should discontinue IMP.
- 9. There is confirmation of a pregnancy during the study, as evidenced by a positive pregnancy test (see Section 12.1.4 for more information regarding pregnancies).
- 10. A subject considered as having either a suspected new LTB infection or who develops active TB or NTMB infection during the study (including but not limited to, conversion demonstrated by IGRA or other diagnostic means) must be immediately discontinued from IMP and a PEOT Visit must be scheduled as soon as possible, but not later than the next regular visit.

The subject must be permanently withdrawn if further examinations result in a diagnosis of active TB, or if the subject is diagnosed with latent TB infection (LTBI) with no initiation of prophylactic treatment, prematurely discontinues prophylactic treatment, or, in the opinion of the Investigator or Sponsor, is noncompliant with prophylactic TB therapy.

Confirmed active TB is an SAE and must be captured on an SAE Report Form and provided to the Sponsor in accordance with SAE reporting requirements. As with all SAEs, periodic follow-up reports should be completed as per protocol requirements until such time as the TB infection resolves.

Additional information on TB policies is provided in Section 12.3.1.

- 11. Subjects with newly diagnosed inflammatory bowel disease (IBD) or with IBD flares during the study must:
  - Be referred, as appropriate, to a health care professional treating IBD, such as a gastroenterologist
  - Discontinue IMP and be followed-up until resolution of active IBD symptoms

If IBD flares increase in severity or frequency during the study, the Investigator should use clinical judgement in deciding whether the subject should continue in the study and contact the Medical Monitor and UCB study physician to confirm the subject's suitability for continued participation in the study.

- 12. Subjects **must be referred** immediately to a mental health care professional and may be withdrawn from the study based upon the Investigator's judgment of benefit/risk for:
- Moderately severe major depression as indicated by a PHQ-9 score of 15 to 19 if this represents an increase of 3 points compared to last visit.

  jects must be referred immediately to a mental healthcare.
- 13. Subjects must be referred immediately to a mental healthcare professional and must be withdrawn in case of:
- Active suicidal ideation as indicated by a positive response ("Yes") to Question 5 of the "Since Last Visit" version of the eC-SSRS
- Any suicidal behavior since last visit.
- Severe major depression as indicated by a PHQ-9 score  $\geq 20$ .

The mental health consultation must be recorded in source documentation.

Investigators should attempt to obtain information on subjects in the case of withdrawal or discontinuation. For subjects considered as lost to follow-up, the Investigator should make an effort (at least 1 phone call and 1 written message to the subject), and document his/her effort (date and summary of the phone call and copy of the written message in the source documents), to complete the final evaluation. All results of these evaluations and observations, together with a narrative description of the reason(s) for removing the subject, must be recorded in the source documents. The electronic Case Report Form (eCRF) must document the primary reason for withdrawal or discontinuation.

Investigators should contact the Medical Monitor, whenever possible, to discuss the withdrawal of a subject in advance.

### Potential drug-induced liver injury IMP discontinuation criteria 6.3.1

Subjects with potential drug-induced liver injury (PDILI) must be assessed to determine if IMP must be discontinued. In addition, all concomitant medications and herbal supplements that are not medically necessary should also be discontinued.

The PDILI criteria below require immediate and permanent discontinuation of IMP for subjects with either of the following:

ALT or AST >8xULN

ALT or AST  $\ge 3xULN$  and coexisting total bilirubin  $\ge 2xULN$ 

The PDILI criterion below requires immediate discontinuation of IMP for:

Subjects with ALT or AST >3xULN who exhibit temporally associated symptoms of in a nondrug-related cause for the symptoms can be confirmed, these subjects may resume IMP administration after discussion with the responsible UCB physician, but only when the requirements for rechallenge with IMP as provided in Section 12.2.1.2.1 are followed.

PDILI criterion below allows for subjects to continue on IMP and the estigator. hepatitis or hypersensitivity. Hepatitis symptoms include fatigue, nausea, vomiting, right

The PDILI criterion below allows for subjects to continue on IMP at the discretion of the Investigator.

Subjects with ALT or AST  $\geq$ 5xULN and  $\leq$ 8xULN, total bilirubin  $\leq$ 2xULN, and no eosinophilia (ie, \le 5\%), with no fever, rash, or symptoms of hepatitis (eg, fatigue, nausea, vomiting, right upper quadrant pain, or tenderness).

Evaluation of PDILI must be initiated as described in Section 12.2.1 with repeat tests performed in 2 weeks. Upon re-test, if ALT or AST values have reduced to <5xULN, the subject can continue with the study. However, if ALT or AST remains >5xULN and <8xULN after re-test, IMP should be temporarily withheld and subject should undergo a</p> repeat test in 2 weeks. If ALT or AST values remain  $\geq 5$ xULN even after the second re-test, then the subject should be permanently withdrawn from the study and should be followed for possible drug-induced liver injury.

If subjects are unable to comply with the applicable monitoring schedule, IMP must be discontinued immediately.

Investigators should attempt to obtain information on subjects in the case of IMP discontinuation to complete the final evaluation. Subjects with PDILI should not be withdrawn from the study until investigation and monitoring are complete. All results of these evaluations and observations, as well as the reason(s) for IMP discontinuation and subject withdrawal (if applicable), must be recorded in the source documents. The eCRF must document the primary reason for IMP discontinuation.

### STUDY TREATMENT(S) 7

### **Description of investigational medicinal product(s)** 7.1

The IMPs used in this study are bimekizumab, adalimumab, and placebo.

Bimekizumab will be supplied in a 1mL prefilled syringe (PFS) at a concentration of for sc injection.

- Adalimumab is commercially available and will be supplied as a PFS for sc injection (at a concentration of 40mg/0.8mL or 40mg/0.4mL depending on regional availability) in a singleuse syringe.
- Placebo will be supplied as 0.9% sodium chloride aqueous solution (physiological saline, preservative-free) of pharmacopoeia (USP/Ph.Eur) quality in a 1mL PFS for sc injection.

Further details of the IMPs and their specifications are provided in the IMP Handling Manual.

### 7.2 Treatment(s) to be administered

Unblinded study staff will be responsible for preparation of the clinical study material, including recording the administration information on source documents, and administration of the IMP as sc injections. The unblinded personnel will not be involved in the study in any way other than assuring the medication is taken from the correct kit and administering the IMP to the subjects.

Suitable areas for sc injections are the lateral abdominal wall and upper outer thigh. During each dosing visit, each of the injections should be administered at a separate injection site. Injection sites should be rotated at each visit and injections should not be given into a PSO plaque or areas where the skin is tender, bruised, erythematous, or indurated. The injection should last approximately 10 to 15 seconds.

An IMP Handling Manual will be provided to each site containing instructions regarding drug preparation and dosing.

Eligible subjects will be randomized 1:1:1 to receive the following blinded study treatment regimens: bimekizumab 320mg Q4W throughout the study, bimekizumab 320mg Q4W until Week 16, or adalimumab.

Because of differences in the dosing schedule between bimekizumab and adalimumab and in order to maintain blinding, all subjects will receive 2 injections sc on Weeks 0 (Baseline), 4, 8, 12, 16, 20, and 24, and 1 injection sc in other weeks:

- Subjects randomized to receive bimekizumab 320mg Q4W throughout the study will receive 2 bimekizumab 160mg injections sc Q4W at Weeks 0 (Baseline), 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52. These subjects will receive 1 placebo injection at Weeks 1, 3, 5, 7, 9, 11, 13, 15, 17, 19, 21, and 23.
- Subjects randomized to receive bimekizumab 320mg Q4W/Q8W will receive 2 bimekizumab 160mg injections sc Q4W at Weeks 0 (Baseline), 4, 8, and 12. Subjects will then receive 2 bimekizumab 160mg injections sc Q8W at Weeks 16, 24, 32, 40, and 48. These subjects will receive 1 placebo injection at Weeks 1, 3, 5, 7, 9, 11, 13, 15, 17, 19, 21, and 23, and 2 placebo injections at Weeks 20, 28, 36, 44, and 52.
- Subjects randomized to receive adalimumab will receive 2 adalimumab 40mg injections sc at Week 0 (Baseline). At Weeks 1, 3, 5, 7, 9, 11, 13, 15, 17, 19, 21, and 23, they will receive 1 adalimumab 40mg injection sc. These subjects will receive 2 placebo injections at Weeks 4, 8, 12, 16, and 20. These subjects will then receive bimekizumab 320mg Q4W given as 2 bimekizumab 160mg injections sc Q4W at Weeks 24, 28, 32, 36, 40, 44, 48, and 52.

The dosing scheme is depicted in Table 7–1.



Table 7-1: **Dosing scheme** 

| Week O | | | ı | | | 1 | | 1 | 1 | 1 | 1 | | 1 | | 1 | | | 3); | 1 | 1 | 1 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| bimekizumab 320mg | Week<br>Dose Assignment | 0 | | 4 | | 8 | | 12 | | 16 | | 20 | | 24 | 28 | 32 | 36 | 40 | 44 | 48 | 52 |
| Q4W/Q8W adalimumab 40mg/bimekizumab 220mg Q4W/ | | •• | 0 | •• | 0 | •• | 0 | •• | 0 | •• | 0 | •• | 0 | •• | •• | RSION | •• | •• | •• | •• | •• |
| adalimumab 40mg/bimekizumab 220mg OAW | | •• | 0 | •• | 0 | •• | 0 | •• | 0 | •• | 0 | 00 | 0 | 472 | <b>6</b> | •• | 00 | •• | 00 | •• | 00 |
| Q4W=every 4 weeks; Q8W=every 8 weeks Notes: A bimekizumab 160mg injection is depicted by a black circle (•). A placebo injection is depicted by a white circle (o). An adalimumab 40mg injection is depicted by a black triangle (•). An adalimumab 40mg injection is depicted by a black circle (•). A placebo injection is depicted by a white circle (o). An adalimumab 40mg injection is depicted by a black triangle (•). | 40mg/bimekizumab<br>320mg Q4W | | | | | | | | | | | | ol sil | •• | | | | | | | |
| | be used to support any marketing authorization. | | | | | | | | | | | | | | | | | | | | |

#### 7.3 **Packaging**

or variations thereof Bimekizumab, adalimumab, and placebo will be packaged and labeled according to Good Manufacturing Practice (GMP) guidelines and applicable laws or regulations. They will be suitably packaged in such a way as to protect the product from deterioration during transport and storage. Further information regarding storage and transport conditions are provided in the IMP Handling Manual.

#### 7.4 Labeling

Bimekizumab, adalimumab, and placebo will be labeled in accordance with the current International Council for Harmonisation (ICH) guidelines on Good Clinical Practice (GCP) and GMP and will include any locally required statements. If necessary, labels will be translated into

Refer to the IMP Handling Manual for the storage conditions of the IMP.

The Investigator (or designee) is responsible for the safe and Investigational medicinal manual for the safe and Investigation for the s The Investigator (or designee) is responsible for the safe and proper storage of IMP at the site. Investigational medicinal product stored by the Investigator is to be kept in a secured area with limited access according to the storage conditions mentioned on the label.

Appropriate storage conditions must be ensured either by controlling the temperature (eg, room, refrigeration unit) or by completion of a temperature log in accordance with local requirements on a regular basis (eg, once a week), showing actual and minimum/maximum temperatures reached over the time interval.

In case an out-of-range temperature is noted, it must be immediately reported as per instructions contained in the IMP Handling Manual.

The IMP will be shipped to the study sites in temperature controlled containers. Out-of-range shipping or storage conditions must be brought to the attention of the Sponsor or designee, immediately. Authorization to use any out-of-range IMP must be documented and received prior to dispensing or administering the IMP at the study site.

### Drug accountability 7.6

A Drug Accountability Form will be used to record IMP dispensing and return information on a by subject basis and will serve as source documentation during the course of the study. Details of any IMP lost, damaged (eg, due to breakage or wastage), not used, partially used, disposed of at the study site, or returned to the Sponsor or designee must also be recorded on the appropriate forms. All supplies and pharmacy documentation must be made available throughout the study for UCB (or designee) to review.

In order to maintain the blind, all IMP documentation (eg, shipping receipts, drug accountability logs, Interactive Response Technology (IRT) randomization materials) must be maintained and accessed by unblinded, trained site personnel only. Designated, unblinded site personnel must be appropriately trained and licensed (per country guidelines) to administer injections.

Unblinded study staff will be delegated the responsibility to receive, inventory and destroy the used kits. The packaging identifies each kit by a unique number, but due to the commercial packaging of the comparator, the unblinded study staff will be responsible in order to maintain

the blind. Unblinded study staff will be responsible for preparation (breaking tamper proof sticker on kit, etc) of the clinical study material, including recording the administration information on source documents.

The Investigator may assign some of the Investigator's duties for drug accountability at the study site to an appropriate pharmacist/designee.

The Investigator must ensure that the IMP is used only in accordance with the protocol.

Periodically, and/or after completion of the clinical phase of the study of the stud destroyed at the site according to local laws, regulations, and UCB Standard Operating Procedures (SOPs) or returned to UCB (or designee). Investigational medicinal product intended for the study cannot be used for any other purpose than that described in this protocol.

### Procedures for monitoring subject compliance 7.7

During the Treatment Period of this study, the IMP will be administered in the clinic and compliance will be determined at the visit by study personnel. Drug accountability must be recorded on the Drug Accountability Form.

#### 7.8 Concomitant medication(s)/treatment(s)

Any treatment administered from the time of informed consent to the final study visit will be considered concomitant medication. This includes medications that were started before the study and are ongoing during the study.

#### Permitted concomitant treatments (medications and therapies) 7.8.1

#### Topical medications 7.8.1.1

Subjects may continue to use topical moisturizers or emollients, bath oils, or oatmeal bath preparations for skin conditions during the study, as needed. Over-the-counter shampoos for the treatment of PSO of the scalp are also permitted.

Mild and low potency topical steroids will be permitted for use limited to the face, axilla, and/or genitalia, as needed. These topical medications should not be used within approximately 24 hours prior to study visits requiring IGA and PASI measures.

#### Other medications 7.8.1.2

Subjects who are already receiving an established NSAID regimen for PsA or symptoms of arthritis and have been on a stable dose for at least 1 week prior to the Screening Visit may continue their use during the study. However, initiation of, or increase in dosage of NSAIDs during the study (especially in subjects with a history of gastrointestinal (GI) intolerance to NSAIDs or a history of GI ulceration) should not occur prior to Week 24 and should not happen within 2 weeks of the Week 56 Visit.

Subjects may take mild pain relievers (acetaminophen/paracetamol, mild opiates) as needed for arthritis pain but preferably not within 24 hours of the Baseline and Week 56 Visits.


Intra-articular steroid injections of any joint and hyaluronic acid injections are allowed after Week 24.

Subjects who are receiving an established regimen for depression should remain on stable dosing prior to Baseline and throughout the study.

## 7.8.2 Prohibited concomitant treatments (medications and therapies)

Table 7–2 presents the list of prohibited medications.

Table 7–2: Prohibited psoriasis medications

| Drug | Washout period relative to Baseline Visit |
|---|---|
| Topicals except for those permitted (Section 7.8.1.1) | 2 weeks |
| Systemic retinoids | 3 months |
| Systemic treatment (nonbiological): | 1 month |
| systemic immunosuppressant agents (eg, methotrexate, cyclosporine, azathioprine, thioguanine) | 3 months 1 month Any exposure to adalimumab 1 month for etanercept 3 months for infliximab (including biosimilar), |
| fumaric acid esters specifically used for the treatment of PSO | ot oplicati |
| systemic corticosteroids | Of Low |
| phototherapy | ijo' |
| Anti-TNFs: | XLC I |
| Anti-TNFs: adalimumab (including biosimilar) etanercept (including biosimilar) | Any exposure to adalimumab |
| etanercept (including biosimilar) | 1 month for etanercept |
| infliximab (including biosimilar), golimumab, certolizumab pegol | 3 months for infliximab (including biosimilar), golimumab, certolizumab pegol |
| Other biologics and other systemic therapies, eg: | |
| apremilast, tofacitinib | 2 weeks for apremilast and tofacitinib |
| alefacept, efalizumab, guselkumab | 3 months for alefacept, efalizumab, and guselkumab |
| tildrakizumab, risankizumab | 5 months for tildrakizumab and risankizumab |
| ustekinumab <sub>s</sub> Briakinumab | 6 months for ustekinumab and briakinumab |
| rituximab | 12 months for rituximab |
| Anti-IL-17 therapy: | 3 months |
| brodalumab | (bimekizumab is excluded per exclusion |
| ixekizumab | criteria) |
| secukinumab | |
| Any other antipsoriatic agent (systemic) under investigation (or approved after the protocol is approved) | 3 months or 5 half-lives, whichever is greater |

### Table 7-2: Prohibited psoriasis medications

| Drug | Washout period relative to Baseline Visit |
|---|---|
| Any other antipsoriatic agent (topical) under investigation | 1 month |

IL-17=interleukin 17; PSO=psoriasis; TNF=tumor necrosis factor

Subjects who take prohibited medications may be withdrawn from IMP but followed until the SFU Visit. The decision to withdraw a subject for taking prohibited medications should be made in consultation with the Medical Monitor.

### **7.8.2.1 Vaccines**

Administration of live (including attenuated) vaccines is not allowed during the conduct of the study and for 20 weeks after the final dose of the IMP (see Exclusion Criterion #10, Section 6.2). Administration of inactivated vaccines is allowed during the study at the discretion of the Investigator.

## 7.9 Blinding

Due to differences in presentation between the bimekizumab and adalimumab, special precautions will be taken to ensure study blinding and study sites will have blinded and unblinded personnel.

All Sponsor and Investigator site personnel involved in the study will be blinded to the randomized IMP assignment with the following exceptions:

- Unblinded study staff will be responsible for preparation (breaking tamper proof sticker on kit, etc) of the clinical trial material, including recording the administration information on source documents, and administration of the IMP as sc injections. The unblinded personnel will not be involved in the study in any way other than assuring the medication is taken from the correct kit and administering the drug to the subjects.
- Bioanalytical staff analyzing blood samples for bimekizumab and anti-bimekizumab antibody determination.

During the study, the Sponsor will provide blinded and unblinded site monitors for the purposes of verifying safety, efficacy, and drug administration and documentation records. Unblinded study site personnel need to be available in order to resolve queries. Study monitors and study site personnel blinded to treatment assignment will not discuss or have access to any drug-related information.

Study sites will be required to have a written blinding plan in place, signed by the Principal Investigator, which will detail the site's steps for ensuring that the double-blind nature of the study is maintained. Sites will be instructed to keep study subjects blind to the IMP as detailed in the site blinding plan.

Further details are provided in the study manual and site blinding plan.

ations thereof

### 7.9.1 Procedures for maintaining and breaking the treatment blind

### 7.9.1.1 Maintenance of IMP blind

All subject treatment details (bimekizumab or adalimumab) will be allocated and maintained by the IRT system.

### 7.9.1.2 Breaking the treatment blind in an emergency situation

The integrity of this clinical study must be maintained by observing the treatment blind. In the event of an emergency for which the appropriate treatment for a subject cannot be made without knowing the treatment assignment, it will be possible to determine to which treatment arm and dose the subject has been allocated by contacting the IRT. All sites will be provided with details of how to contact the system for code breaking at the start of the study. The Medical Monitor or equivalent should be consulted prior to unblinding, whenever possible.

The Clinical Project Manager (CPM) will be informed immediately via the IRT when a code is broken, but will remain blinded to specific treatment information. Any unblinding of the IMP performed by the Investigator must be recorded in the source documents and on the Study Termination eCRF page.

## 7.10 Randomization and numbering of subjects

An IRT will be used for assigning eligible subjects to a treatment regimen based on a predetermined production randomization and/or packaging schedule provided by UCB (or designee). The randomization schedule will be produced by the IRT vendor. The IRT will generate individual assignments for subject kits of IMP, as appropriate, according to the visit schedule. Subject treatment assignment will be stratified by region (North America, Western Europe, Central/Eastern Europe and Asia/Australia) and prior biologic exposure (yes/no). The IRT will generate individual assignments for subject kits of IMP, as appropriate, according to the visit schedule.

At Screening, each subject will be assigned a 5-digit number that serves as the subject identifier throughout the study. The subject number will be required in all communication between the Investigator or designee and the IRT regarding a particular subject.

At the Baseline Visit, a subject will be randomized into the study. The Investigator or designee will use the IRT for randomization. The IRT will automatically inform the Investigator or designee of the subject's identification number. The IRT will allocate kit numbers to the subject based on the subject number during the course of the study. The kits are blinded.

Subject numbers and kit numbers will be tracked via the IRT.

### 8 STUDY PROCEDURES BY VISIT

Table 5–1 (Schedule of study assessments) provides a general overview of study assessments. A list of procedures to be completed at each visit is described below.

From the Week 1 Visit to the Week 24 Visit, visit windows of ±3 days on either side of the scheduled dosing are permitted; however, the Investigator should try to keep the subjects on the original dosing schedule. From the Week 28 Visit to the Week 52 Visit, visit windows are ±7 days. Changes to the dosing schedule outside of the visit window must be discussed with the Medical Monitor.


- The dosing window is  $\pm 3$  days relative to the scheduled dosing visit through Week 24. The dosing window is  $\pm 7$  days relative to the scheduled dosing visit from Week 28 through the end of the study.

Screening Visit (2 to 5 weeks)

Prior to any study specific activities, subjects will be asked to read, sign, and date an ICF that has been approved by the Sponsor and an Institutional Review Board (IRB)/Independent Ethics.

Committee (IEC), and that complies with regulatory requirements. Subject adequate time to consider any information concerns or designee. As part of the information concerns. ask the Investigator any questions regarding potential risks and benefits of participation in the study.

Where local regulations permit, subjects will also be given the option to participate in the genomics, genetics, and proteomics substudy. Subjects agreeing to participate in the substudy will be required to complete a separate ICF. The ICF must be signed prior to collecting any samples for the substudy. The substudy will only be conducted where ethically accepted and authorized by the regulatory agencies. Refusal to participate in the substudy will not affect a subject's ability to participate in the main PS0008 study.

The following procedures or assessments will be performed at the Screening Visit:

- Obtain written informed consent
- Assessment of inclusion and exclusion criteria
- Urine drug screen
- Demographic data (age, gender, race, and ethnicity [according to local regulations])
- Psoriasis history including the date of onset and past treatments
- Significant past medical history including clinically relevant past or coexisting medical conditions and surgeries
- Physical examination including evaluation of signs and symptoms of active TB and risk for exposure to TB
- Vital signs (sitting systolic and diastolic blood pressure [BP], pulse rate, and body temperature) should be obtained prior to blood sampling
- Collect blood and urine samples for the following clinical laboratory tests:

Hematology and biochemistry

- Urinalysis
- Serum pregnancy test for women of childbearing potential
- Hepatitis B and Hepatitis C
- HIV

IGRA tuberculosis test; it is recommended that the QuantiFERON TB test be performed

Bimekizumab

- Record 12-lead ECG
- COPT application and any extensions of variations thereoff itation application and any extensions of variations of variations of variations and any extensions of variations of variatio Chest x-ray (not necessary if performed within 3 months prior to Screening Visit and report is available)
- TB questionnaire
- **PASI**
- **IGA**
- Percentage of BSA
- PHQ-9
- eC-SSRS
- Daily Patient Symptom Diary
- Concomitant medications
- Record AEs
- Confirm subject eligibility and contact the IRT

#### **Initial Treatment Period** 8.2

#### 8.2.1 **Baseline Visit**

The following procedures or assessments will be performed/recorded at the Baseline Visit prior to administration of the IMP:

- Re-assessment of inclusion and exclusion criteria
- Significant past medical history and concomitant diseases to ensure no significant changes since screening
- Physical examination including evaluation of signs and symptoms of active TB and risk for exposure to TB
- Height
- Body weight
- Vital signs (sitting systolic and diastolic BP, pulse rate, and body temperature) should be obtained prior to blood sampling
- Obtain blood and urine samples for the following analyses prior to dosing:

Hematology and biochemistry

- Urinalysis
- Urine pregnancy test
- Bimekizumab plasma concentrations
- Anti-bimekizumab antibodies

- Genomic, proteomic, metabolomics, and candidate biomarker analyses (participating subjects only)
- Genetic/epigenetic analyses (participating subjects only)
- TB questionnaire
- **PASI**
- **IGA**
- Percentage of BSA
- DLQI
- PHQ-9
- eC-SSRS
- **Daily Patient Symptoms Diary**
- scalp IGA
- mNAPSI
- pp-IGA
- EQ-5D-3L
- SF-36
- **PASE**
- **PGADA**
- WPAI-SHP V2.0
- Concomitant medications
- Record AEs
- Contact the IRT

After completion of the above-mentioned procedures, administration of bimekizumab or adalimumab will occur.

#### 8.2.2 Week 1 (±3 days)

The following procedures or assessments will be performed/recorded prior to administration of

- obtain blood samples for "

  Hemat" Vital signs (sitting systolic and diastolic BP, pulse rate, and body temperature) should be
  - Obtain blood samples for the following analyses prior to dosing:
    - Hematology and biochemistry
    - Bimekizumab plasma concentrations

eations

Party Property Copy of a policy in a policy i

- Genomic, proteomic, metabolomics, and candidate biomarker analyses (participating subjects only)
- PASI
- IGA
- Percentage of BSA
- DLOI
- eC-SSRS
- Daily Patient Symptom Diary
- Scalp IGA for subjects with scalp involvement at Baseline
- Concomitant medications
- Record AEs
- Contact the IRT

After completion of the above-mentioned procedures, administration of adalimumab or placebo will occur.

### 8.2.3 Week 3 (±3 days)

The following procedures or assessments will be performed/recorded prior to administration of the IMP:

- Vital signs (sitting systolic and diastolic BP, pulse rate, and body temperature) should be obtained prior to blood sampling
- Obtain blood samples for the following analyses prior to dosing:
  - Hematology and biochemistry
  - Bimekizumab plasma concentrations
- PASI
- IGA
- Percentage of BSA
- DLOI
- eC-SSRS
- Daily Patient Symptom Diary
- Scalp IGA for subjects with scalp involvement at Baseline
- Concomitant medications
- Record AEs
- Contact the IRT

After completion of the above-mentioned procedures, administration of adalimumab or placebo will occur.

Bimekizumab

## 8.2.4

The following procedures or assessments will be performed/recorded prior to administration of the IMP:

- eC-SSRS

  Daily Patient Symptom Diary

  Scalp IGA for subjects with nail involvement at Baseline
  nNAPSI for subjects with palmoplantar involvement
  -5D-3L

  A for subjects with PsA at P
  mitant medications
  AEs
  re IRT

- Contact the IRT

with comparing the second will occur.

8.2 F After completion of the above-mentioned procedures, administration of bimekizumab or placebo

### Week 5 and 7 (±3 days)

The following procedures or assessments will be performed/recorded prior to administration of the IMP:

- Vital signs (sitting systolic and diastolic BP, pulse rate, and body temperature) should be obtained prior to blood sampling
- eC-SSRS
- Daily Patient Symptom Diary
- Concomitant medications
- Record AEs
- Contact the IRT

After completion of the above-mentioned procedures, administration of adalimumab or placebo will occur.

### 8.2.6 Week 8 (±3 days)

The following procedures or assessments will be performed/recorded prior to administration of the IMP:

- Vital signs (sitting systolic and diastolic BP, pulse rate, and body temperature) should be obtained prior to blood sampling
- Obtain blood and urine samples for the following analyses prior to dosing:
  - Hematology and biochemistry
  - Urine pregnancy test
  - Bimekizumab plasma concentrations
  - Anti-bimekizumab antibodies
  - Genomic, proteomic, metabolomics, and candidate biomarker analyses (participating subjects only)
- PASI
- IGA
- Percentage of BSA
- DLOI
- PHQ-9
- eC-SSRS<sup>©</sup>
- Daily Patient Symptom Diary
- Scalp IGA for subjects with scalp involvement at Baseline
- mNAPSI for subjects with nail involvement at Baseline
- pp-IGA for subjects with palmoplantar involvement at Baseline
- EQ-5D-3L
- SF-36

- Concomitant medications
- Record AEs

- Week 9 and 11 (±3 days)

  The following procedures or assessments will be performed/recorded prior to administration of the IMP:

   Vital signs (sitting systolic and diastolic BP, pulse rate, and body obtained prior to blood sampling

   eC-SSRS
- eC-SSRS
- Daily Patient Symptom Diary
- Concomitant medications
- Record AEs
- Contact the IRT

After completion of the above-mentioned procedures, administration of adalimumab or placebo will occur.

8.2.8 Week 12 (±3 days)

The following procedures or assessments will be performed/recorded prior to administration of the IMP:

- Physical examination including evaluation of signs and symptoms of active TB and risk for exposure to TB
- Body weight
- Vital signs (sitting systolic and diastolic BP, pulse rate, and body temperature) should be obtained prior to blood sampling
- Obtain blood and urine samples for the following analyses prior to dosing:
  - Hematology and biochemistry
  - Urine pregnancy test
  - Bimekizumab plasma concentrations

Anti-bimekizumab antibodies

- Genomic, proteomic, metabolomics, and candidate biomarker analyses (participating subjects only)
- Record 12-lead ECG
- TB questionnaire

- **PASI**
- **IGA**

- ...daseline
  ...daseline
  ...das

with comparing the second will occur.

8.2 4

### Week 16 (±3 days)

The following procedures or assessments will be performed/recorded prior to administration of the IMP:

- Vital signs (sitting systolic and diastolic BP, pulse rate, and body temperature) should be obtained prior to blood sampling
- PASI
  GA
  'ercentage of BSA
  LQI
  HO-0 Daily Patient Symptom Diary
  Scalp IGA for subjects with scalp involvement at Baseline
  mNAPSI for subjects with nail involvement at Baseline
  p-IGA for subjects with palmoplantar involvement

  2-5D-3L
  -36
  ADA
  AI-SHP\*

- WPAI-SHP V2.0
- Concomitant medications
- Record AEs
- Contact the IRT

After completion of the above-mentioned procedures, the Maintenance Treatment Period will begin with administration of bimekizumab or placebo.

#### 8.3 **Dose-blind Maintenance Treatment Period**

#### 8.3.1 Week 17 and 19 (±3 days)

The following procedures or assessments will be performed/recorded prior to administration of the IMP:

- Vital signs (sitting systolic and diastolic BP, pulse rate, and body temperature) should be obtained prior to blood sampling
- eC-SSRS
- Daily Patient Symptom Diary
- Concomitant medications
- Record AEs
- Contact the IRT

After completion of the above-mentioned procedures, administration of adalimumab or placebo will occur.

### 8.3.2 Week 20 (±3 days)

The following procedures or assessments will be performed/recorded prior to administration of the IMP:

- Vital signs (sitting systolic and diastolic BP, pulse rate, and body temperature) should be obtained prior to blood sampling
- Obtain blood and urine samples for the following analyses prior to dosing:
  - Hematology and biochemistry
  - Urine pregnancy test
  - Bimekizumab plasma concentrations
  - Anti-bimekizumab antibodies
- PASI
- IGA
- Percentage of BSA
- DLQI
- PHQ-9
- eC-SSRS
- Daily Patient Symptom Diary
- Scalp IGA for subjects with scalp involvement at Baseline
- mNAPSI for subjects with nail involvement at Baseline
- pp-IGA for subjects with palmoplantar involvement at Baseline
- Concomitant medications
- Record AEs
- Contact the IRT

After completion of the above-mentioned procedures, administration of bimekizumab or placebo will occur.

## 8.3.3 Week 21 and 23 (±3 days)

The following procedures or assessments will be performed/recorded prior to administration of the IMP:

- Vital signs (sitting systolic and diastolic BP, pulse rate, and body temperature) should be obtained prior to blood sampling
- eC-SSRS
- Daily Patient Symptom Diary
- Concomitant medications
- Record AEs
- Contact the IRT

After completion of the above-mentioned procedures, administration of adalimumab or placebo will occur.

### 8.3.4 Week 24 (±3 days)

The following procedures or assessments will be performed recorded prior to administration of the IMP:

- Physical examination including evaluation of signs and symptoms of active TB and risk for exposure to TB
- Body weight
- Vital signs (sitting systolic and diastolic BP, pulse rate, and body temperature) should be obtained prior to blood sampling
- Obtain blood and urine samples for the following analyses prior to dosing:
  - Hematology and biochemistry
  - Urinalysis
  - Urine pregnancy test
  - Bimekizumab plasma concentrations
  - Anti-bimekizumab antibodies
- TB questionnaire
- Record 12-lead ECG
- PASI
- IGA
- Percentage of BSA
- DLQI

- PHQ-9
- eC-SSRS
- Daily Patient Symptom Diary
- Scalp IGA for subjects with scalp involvement at Baseline
- mNAPSI for subjects with nail involvement at Baseline
- pp-IGA for subjects with palmoplantar involvement at Baseline
- EQ-5D-3L
- SF-36
- Patient global assessment of PSO
- **PGADA**
- WPAI-SHP V2.0
- Concomitant medications
- Record AEs
- Contact the IRT

After completion of the above-mentioned procedures, administration of bimekizumab or placebo will occur.

8.3.5 Week 28 (±7 days)

The following procedures or assessments will be performed/recorded prior to administration of the IMP:

- Vital signs (sitting systolic and diastolic BP, pulse rate, and body temperature) should be obtained prior to blood sampling
- Obtain urine sample for the following analyses prior to dosing:
  - Hematology and biochemistry
  - Urine pregnancy test
- **PASI**
- **IGA**
- Percentage of BSA
- PHQ-9
- eC-SSRS
- Concomitant medications
- Record AEs
- Contact the IRT

After completion of the above-mentioned procedures, administration of bimekizumab or placebo will occur.

## 8.3.6

The following procedures or assessments will be performed/recorded prior to administration of the IMP:

- ...or to dosing:

  ...or to dosing:

  ...or to dos

After completion of the above-mentioned procedures, administration of bimekizumab or placebo will occur.

#### 8.3.7 Week 36 (±7 days)

The following procedures or assessments will be performed/recorded prior to administration of

- ne folle imp: Physical examination including evaluation of signs and symptoms of active TB and risk for exposure to TB
  - Body weight

- Vital signs (sitting systolic and diastolic BP, pulse rate, and body temperature) should be obtained prior to blood sampling

- ...omitant medications

   Record AEs

   Contact the IRT

  After completion of the above-mentioned procedures, administration of bimekizumab or placebo will occur.

  3.8 Week 40 (±7 days)

   following procedures or assessments will be performed/recorded prior to administration of bimekizumab or placebo will occur.

  Vital signs (sitting systolic and diastolic BP, pulse rate, and body btained prior to blood sampling vain blood and upine samples for the following anal-Hematology and biochemistry brinalysis inc pregnancy test

  - **J**ĞA
  - Percentage of BSA
  - **DLQI**
  - Scalp IGA for subjects with scalp involvement at Baseline
  - mNAPSI for subjects with nail involvement at Baseline

- pp-IGA for subjects with palmoplantar involvement at Baseline
- PHO-9
- eC-SSRS
- EQ-5D-3L
- SF-36
- Patient global assessment of PSO
- PGADA for subjects with PsA at Baseline
- WPAI-SHP V2.0
- Concomitant medications
- Record AEs
- Contact the IRT

After completion of the above-mentioned procedures, administration of bimekizumab or placebo will occur.

#### 8.3.9 Week 44 (±7 days)

The following procedures or assessments will be performed/recorded prior to administration of the IMP:

- Vital signs (sitting systolic and diastolic BP, pulse rate, and body temperature) should be obtained prior to blood sampling
- Obtain urine sample for the following analyses prior to dosing:
  - Urine pregnancy test
- **PASI**
- **IGA**
- Percentage of BSA
- PHQ-9
- eC-SSRS
- Concomitant medications
- Record AEs
- Contact the IRT

after comparing the second sec After completion of the above-mentioned procedures, administration of bimekizumab or placebo

### Week 48 (±7 days)

The following procedures or assessments will be performed/recorded prior to administration of the IMP:

- Physical examination including evaluation of signs and symptoms of active TB and risk for exposure to TB
- . ercentage of BSA
  DLQI
  Scalp IGA for subjects with scalp involvement at Baseline
  nNAPSI for subjects with nail involvement at Baseline
  2-IGA for subjects with palmoplantar involvement
  1Q-9
  SSRS
  nt global assessment of PSC
  DA for subjects with
  nitant medic

- Record AEs
- Contact the IRT

After completion of the above-mentioned procedures, administration of bimekizumab or placebo will occur.

#### 8.3.11 Week 52 (±7 days)

The following procedures or assessments will be performed/recorded prior to administration of the IMP:

Obtain informed consent for the open-label study

- Vital signs (sitting systolic and diastolic BP, pulse rate, and body temperature) should be obtained prior to blood sampling
- Obtain blood and urine samples for the following analyses prior to dosing:
  - Urine pregnancy test
  - IGRA tuberculosis test; it is recommended that the QuantiFERON TB test be performed
- **PASI**
- Percentage of BSA
- **IGA**
- PHQ-9
- eC-SSRS
- Concomitant medications
- Record AEs
- Contact the IRT

ion and any extensions or variations thereof. After completion of the above-mentioned procedures, administration of bimekizumab or placebo will occur.

8.3.12 Week 56 (±7 days)

The following procedures or assessments will be performed/recorded:

- Urine drug screen
- Physical examination including evaluation of signs and symptoms of active TB and risk for exposure to TB
- Body weight
- Vital signs (sitting systolic and diastolic BP, pulse rate, and body temperature) should be obtained prior to blood sampling
- Obtain blood and urine samples for the following analyses prior to dosing:
  - Hematology and biochemistry
  - Urinalysis
  - Urine pregnancy test
  - Bimekizumab plasma concentrations
    - Anti-bimekizumab antibodies
  - Genomic, proteomic, metabolomics, and candidate biomarker analyses (participating subjects only)
  - Genetic/epigenetic analyses (participating subjects only)
- Record 12-lead ECG

- TB questionnaire
- **PASI**
- **IGA**
- Percentage of BSA
- DLQI
- PHQ-9
- eC-SSRS
- Scalp IGA for subjects with scalp involvement at Baseline
- mNAPSI for subjects with nail involvement at Baseline
- pp-IGA for subjects with palmoplantar involvement at Baseline
- EQ-5D-3L
- SF-36
- Patient global assessment of PSO
- **PASE**
- PGADA for subjects with PsA at Baseline
- WPAI-SHP V2.0
- Concomitant medications
- Record AEs
- Contact the IRT

### Premature End of Treatment Visit 8.4

If a subject is withdrawn from the study:

- The subject will be withdrawn from IMP, will undergo the same assessments as the Week 56 visit (see Section 8.3.12), and will enter the SFU Period.
- The subject will be encouraged to return for the SFU Visit (20 weeks after the last received dose; see Section 8.5).

Treat

#### 8.5 Safety Follow-Up Visit (20 weeks after final dose ±7 days)

Anti-bimekizumab plasma concentrations

Anti-bimekizumab antibodies

TB questionnaire

PASI

GA

Percentage of BSA

C-SSRS

Oncomitant medications

ecord AEs

ontact the IRT

Unscheduled Visit

Investigator's disappoint to ITB

Vial signs (sitting systolic and diastolic blood pressure, pulse rate, and body temperature) antibulation of signs and symptoms of active TB and risk for exposure to TB

Vital signs (sitting systolic and diastolic blood pressure, pulse rate, and body temperature) antibulation should be obtained prior to blood sampling

Obtain blood and urine samples for the following analyses prior to dosing:

— Hematology and biochemistry

— Urinalysis

— Urine pregnancy test

— Bimekizumab plasma concentrations

— Anti-bimekizumab antibodies

TB questionnaire

PASI

GA

Vercentage of BSA

C-SSRS

Oncomitant medications

ecord AEs

ontact the IRT

Unscheduled Visit

Investigator's disappoints

Investigator's disappoints

Unscheduled Visit All subjects not continuing in the open-label study, including those withdrawn from study treatment, will have a SFU Visit 20 weeks after their final dose of IMP. The following procedures or assessments will be performed/recorded:

### 8.6

At the Investigator's discretion, an Unscheduled Visit may be completed at any time during the study but prior to the SFU Visit, if deemed necessary for the subject's safety and well-being.

If an Unscheduled Visit is conducted due to safety or efficacy reasons, an eC-SSRS assessment will be performed with the subject during the visit. If an Unscheduled Visit is conducted for reasons other than safety or efficacy concerns (eg. repeated collection of a laboratory specimen due to collection or analysis issues), an eC-SSRS will not be required at these visits.

At this visit, any assessment may be performed, as needed, depending on the reason for the visit.

## ASSESSMENT OF EFFICACY

The PASI, BSA, IGA, scalp IGA, mNAPSI, and pp-IGA should be performed by the Investigator, another delegated physician, or an appropriately qualified medical professional (based on local requirements) who has had documented training on how to perform these assessments correctly. The same assessor should evaluate the subject at each assessment.

## 9.1 Psoriasis Area and Severity Index

The PASI is the most commonly used and validated assessment for grading the severity of PSO in clinical studies (Feldman, 2004). The PASI quantifies the severity and extent of the disease and weighs these with the percentage of BSA involvement.

The percent area of involvement (BSA%) is estimated across 4 body areas; head, upper extremities, trunk, and lower extremities. Assessors will enter the degree of involvement for a given region on a scale of 0 to 6 (0=none; 1=1% to <10% affected, 2=10% to <30% affected, 3=30% to <50% affected, 4=50% to <70% affected, 5=70% to <90% affected, 6=90% to 100% affected) (Table 9–3).

The Investigator assesses the average redness, thickness, and scaliness of lesions in each body area (each on a 5-point scale); 0=none, 1=slight, 2=moderate, 3=marked, and 4=very marked.

The PASI score ranges from 0 to 72 with a higher score indicating increased disease severity.

Table 9-3: Body areas for calculation of percent BSA for PASI

| Body area | Details of area | BSA | Degree of involvement of body area |
|---|---|---|---|
| Head | Face, back of head | 10% | 0 to 6 |
| Upper extremities | Left, right, upper lower, flexor surface, extensor surface | 20% | 0 to 6 |
| Trunk | Front, back, groin | 30% | 0 to 6 |
| Lower extremities | Left, right, upper lower, flexor surface, extensor surface, including buttocks | 40% | 0 to 6 |
| Total | Mal | 100% | |

BSA=body surface area; PASI=Psoriasis Area and Severity Index

The PASI50, PASI75, PASI90, and PASI100 responses are based on at least 50%, 75%, 90%, and 100% improvement in the PASI score, respectively.

The total BSA affected by PSO will be entered as a percentage from 0 to 100.

The PASI will be completed at the visits specified in Table 5–1.

## 9.2 Investigator's Global Assessment

A static IGA for PSO will be used to assess disease severity in all subjects during the study. The IGA will be completed at the visits specified in Table 5–1.

The Investigator will assess the overall severity of PSO using the following 5-point scale presented in Table 9–4.

<sup>&</sup>lt;sup>a</sup> Where 0=none; 1=1% to <10% affected; 2=10% to <30% affected; 3=30% to <50% affected; 4=50% to <70% affected; 5=70% to <90% affected; 6=90% to 100% affected

### Table 9–4: Five-point IGA

| Score | <b>Short Descriptor</b> | Detailed Descriptor |
|---|---|---|
| 0 | Clear | No signs of PSO; post-inflammatory hyperpigmentation may be present |
| 1 | Almost clear | No thickening; normal to pink coloration; no to minimal focal scaling |
| 2 | Mild | Just detectable to mild thickening; pink to light red coloration; predominately fine scaling |
| 3 | Moderate | Clearly distinguishable to moderate thickening; dull to bright red, moderate scaling |
| 4 | Severe | Severe thickening with hard edges; bright to deep dark red coloration; severe/coarse scaling covering almost all or all lesions |

IGA=Investigator's Global Assessment; PSO=psoriasis

## 9.3 Dermatology Life Quality Index

The DLQI is a questionnaire designed for use in adult subjects with PSO. The DLQI is a skin disease-specific questionnaire aimed at the evaluation of how symptoms and treatment affect subjects' health related QOL. This instrument asks subjects about symptoms and feelings, daily activities, leisure, work and school, personal relationships and treatment. It has been shown to be valid and reproducible in subjects with PSO. The DLQI score ranges from 0 to 30 with higher scores indicating lower health related QOL. A 4-point change in the DLQI score (DLQI response) has been reported to be meaningful for the subject (within-subject minimal important difference); while a DLQI absolute score of 0 or 1 indicates no or small impact of the disease on health related QOL. Subjects will be asked to complete the DLQI as outlined in the Schedule of Study Assessments (Table 5–1).

# 9.4 Patient Health Questionnaire 9

The PHQ-9 is a multipurpose instrument for screening, diagnosing, monitoring, and measuring the severity of depression (Kroenke et al, 2001). The PHQ-9 scores for depression range from 0 to 27 with higher scores indicating worse state. A score of 5 to 9 is considered to be minimal symptoms of depression. A score of 10 to 14 is considered minor depression, dysthymia, or mild major depression. A score of 15 to 19 is considered to indicate moderately severe major depression, and a score ≥20 is considered to be severe major depression.

The PHQ-9 will be assessed at the visits specified in Table 5–1.

Refer to Section 6.3 for PHQ-9-related withdrawal criteria.

## 9.5 Scalp IGA

A static IGA for scalp PSO will be used to assess disease severity on the scalp.

All subjects will complete the scalp IGA at Baseline. Only subjects with scalp involvement at Baseline will complete the scalp IGA at the other visits specified in Table 5–1. Subjects with scalp involvement at Baseline are defined as those with a scalp IGA score >0 at Baseline.

Scalp lesions will be assessed in terms of clinical signs of redness, thickness, and scaliness using a 5-point scale (Table 9–5).

**UCB** 

| Score | <b>Short Descriptor</b> | Detailed Descriptor |
|---|---|---|
| 0 | Clear | Scalp has no signs of PSO; post-inflammatory hyperpigmentation may be present |
| 1 | Almost clear | Scalp has no thickening; normal to pink coloration; no to minimal focal scaling |
| 2 | Mild | Scalp has just detectable to mild thickening; pink to light red coloration; predominately fine scaling |
| 3 | Moderate | Scalp has clearly distinguishable to moderate thickening; dull to bright red, moderate scaling |
| 4 | Severe | Scalp has severe thickening with hard edges; bright to deep dark red coloration; severe/coarse scaling covering almost all or all lesions |

PSO=psoriasis; scalp IGA=scalp-specific Investigator's Global Assessment

#### 9.6 **mNAPSI**

Nail PSO will be evaluated using the mNAPSI. All affected nails will be scored (0 to 3) for onycholysis/oil drop dyschromia, nail plate crumbling, and pitting and will be scored (0 for "no" or 1 for "yes") for leukonychia, nail bed hyperkeratosis, splinter hemorrhages, and red spots in the lunula. The score for an individual nail ranges from 0 to 13 with higher scores indicative of more severe nail PSO. The total mNAPSI score is the sum of the scores for each individual nail. If a nail is unaffected, it will be recorded as such and will not contribute to the total mNAPSI score. Subjects with nail PSO at Baseline are defined as those with an mNAPSI score >0 at Baseline.

The mNAPSI will be assessed at the visits specified in Table 5–1.

#### 9.7 pp-IGA

A static IGA for palmoplantar PSO will be used to assess palmoplantar disease severity.

All subjects will complete the pp-IGA at Baseline. Only subjects with palmoplantar involvement at Baseline will complete the pp-IGA at the other visits specified in Table 5–1. Subjects with palmoplantar involvement at Baseline are defined as those with a pp-IGA score >0 at Baseline.

Palmoplantar disease will be assessed in terms of clinical signs of redness, thickness, and scaliness using a 5-point scale (Table 9–6).



#### Table 9–6: pp-IGA

| Score | <b>Short Descriptor</b> | Detailed Descriptor |
|---|---|---|
| 0 | Clear | Palmoplantar areas have no signs of PSO; post-inflammatory hyperpigmentation may be present |
| 1 | Almost clear | Palmoplantar areas have no thickening; normal to pink coloration; no to minimal focal scaling |
| 2 | Mild | Palmoplantar areas have just detectable to mild thickening; pink to light red coloration; predominately fine scaling |
| 3 | Moderate | Palmoplantar areas have clearly distinguishable to moderate thickening; dull to bright red and clearly distinguishable coloration; moderate scaling |
| 4 | Severe | Palmoplantar areas have severe thickening with hard edges; bright to deep dark red coloration; severe/coarse scaling covering almost all or all lesions; numerous fissures |

PSO=psoriasis; pp-IGA=palmoplantar-specific Investigator's Global Assessment

### Euro Quality of Life 5-Dimensions, 3-Level 9.8

The EQ-5D-3L health questionnaire provides a descriptive profile and a single index value for health status. The instrument is comprised of a 5-item health status measure and a VAS. The EQ-5D-3L VAS records the respondent's self-rated health status on a vertical 20cm scale, graduated from 0 to 100 (0=worst imaginable health status, 100=best imaginable health status).

The EQ-5D-3L will be assessed at the visits specified in Table 5–1.

### Short Form 36-Item Health Survey 9.9

The SF-36 (Version 2, standard recall) is a 36-item generic health related QOL instrument that uses a recall period of 4 weeks. Items are grouped into 8 domains as follows: Physical Functioning (10 items), Role Physical (4 items), Bodily Pain (2 items), General Health (5 items), Vitality (4 items), Social Functioning (2 items), Role Emotional (3 items), Mental Health (5 items), and 1 item for perceived stability or change in health (Health Transition) during the last year. The concepts represented by these domains contribute to physical, mental, and social aspects of health-related QOL. In addition to domain scores, the PCS and MCS scores are calculated from the 8 domains (excluding the Health Transition item). Component scores appreciate the impact of each domain on physical and mental health status (Maruish, 2011). Each of the 8 domain scores and the component summary scores range from 0 to 100, with a higher score indicating a better health status. The domains and the 2 component summary scores are standardized with a mean of 50 and a standard deviation (SD) of 10 in the general USA Functioning, 3; Role Emotional, 4; and Mental Health, 3.

The SF-36 will be completed: population. The minimally important differences (MIDs), in terms of T-score points at a group level, for SF-36 domains and component summaries are the following: PCS, 2; MCS, 3; Physical

### 9.10 Patient Global Assessment of psoriasis

The Patient Global Assessment of PSO is a PSO-specific item in which the patient responds to the multiple-choice question, "How severe are your psoriasis-related symptoms right now?" Possible responses to the question are "no symptoms," "mild symptoms," "moderate symptoms," "severe symptoms," or "very severe symptoms."

The Patient Global Assessment of PSO will be performed as part of the patient symptoms diary from Screening through the Initial Treatment Period.

During the double-blind Maintenance Treatment Period, this assessment will be completed at the visits specified in Table 5–1.

### 9.11 Patient Symptom Diary responses

UCB developed a new patient-reported outcome (PRO) measure that will be used to assess key symptoms relevant to patients with moderate to severe chronic plaque PSO. PS0010 used the draft PRO measure in selected countries to enable psychometric validation of the PRO. Site staff will train the participating subjects on the use of the electronic PRO (ePRO) diary at the Screening Visit, following which the device will be dispensed to the subject for home use until the Week 24 Visit. The ePRO diary will be administered on a daily basis from Screening to the Week 24 Visit.

The ePRO diary will also administer the patient global assessment of PSO as noted above appropriate anchor items at the end of every study week. The ePRO diary software will be programmed such that the subjects will be given a window of opportunity to complete the ePRO diary. The data collected on the ePRO diary will be uploaded to a central server database and will be 21 CFR Part 11 compliant. Appropriate GCP procedures (including subject/site training and testing) will be performed at the study sites.

# 9.12 sPASE questionnaire

The PASE questionnaire is a self-administered tool to screen for active PsA in patients with PSO (Husni et al, 2014). The questionnaire consists of 15 items that are divided into a 7-item symptoms subscale and an 8-item functions subscale. Standardized responses are based on 5 categories relating to agreement (strongly agree [5], agree [4], no idea [3], disagree [2], and strongly disagree [1]). The total maximum score is 75 points (symptom score: 35 points and function score: 40 points). Psoriatic Arthritis Screening and Evaluation questionnaire scores ≥47 points are indicative of active PsA.

If a subject with a PASE score  $\geq$ 47 points is referred to a rheumatologist, the referral will be recorded in the eCRF. Subjects with PsA, defined as a past medical history of PsA or PASE  $\geq$ 47, are required to receive the additional PsA assessments as noted in Section 9.13.

The PASE questionnaire will be completed at the visits in Table 5–1.

# 9.13 PGADA for the arthritis visual analog scale

The PGADA for the arthritis VAS will be used to provide an overall evaluation of arthritis disease symptoms. Subjects will respond to the question, "Considering all the ways your arthritis affects you, please mark a vertical line on the scale below to show how you are feeling today," using a VAS where 0 is "very good, no symptoms" and 100 is "very poor, severe symptoms."
All subjects will complete the PGADA at Baseline. Subjects with PsA at Baseline (defined as a past medical history of PsA or PASE  $\geq$ 47) will complete the PGADA at the visits specified in Table 5–1.

### 9.14 WPAI-SHP V2.0

The WPAI-SHP V2.0 is a patient-reported questionnaire that assesses subject's employment status, work absenteeism, work impairment while working (presenteeism), overall work, and daily activity impairment attributable to a specific health problem (WPAI-SHP) (Reilly et al, 1993). It has been used in several clinical studies of biologic therapy in subjects with plaque PSO (Kimball et al, 2012; Vender et al, 2012).

Five out of 6 items of the WPAI-SHP are regrouped into the 4 dimensions, with scores expressed as percentage, where higher numbers indicate greater impairment and less productivity, ie, worse outcomes, as described in the WPAI-SHP scoring rules.

The WPAI-SHP V2.0 will be assessed at the visits specified in Table 5–1.

# 10 ASSESSMENT OF PHARMACOKINETIC AND PHARMACOGENOMIC VARIABLE(S)

### 10.1 Pharmacokinetic variables

Blood samples for measurement of PK assessments (Section 4.3.3) will be collected at the time points specified in the schedule of study assessments (Table 5–1).

At dosing visits, blood samples will be drawn prior to dosing, and will be drawn at the same time of the sampling for clinical laboratory tests. The time and date of collection will be recorded in the eCRF.

Instructions pertaining to sample collection, processing, storage, labeling, and shipping are provided in the laboratory manual for this study. Detailed information on sample analysis will be provided in a bioanalytical report.

Pharmacokinetic samples from subjects receiving adalimumab will not be analyzed, but stored for potential future PK analysis and anti-drug antibody determination.

# 10.2 Pharmacogenomic variables

A separate ICF will be required for those subjects who agree to participate in the genomics, genetics, and proteomics substudy, and must be signed prior to collection of any samples for the substudy. The substudy will only be conducted where ethically accepted and authorized by the regulatory agencies. Refusal to participate in the substudy will not affect a subject's ability to participate in the main study.

These analyses will enable evaluation of biomarkers relative to disease biology and progression, drug treatment, and inflammatory and immune response processes. The nature and format of these tentative analyses will be determined at a later date.

For individuals consenting to the genomics, genetics, and proteomics substudy, blood samples will be drawn for exploratory genetic/epigenetic, genomic, proteomic, and metabolomics analysis and for candidate exploratory biomarker analyses. Candidate exploratory biomarker evaluations may include, but are not limited to, IL-17A/IL-17F pathway signaling and PSO

biology (eg, IL-17A, IL-17F, IL-23, IL-6, tumor necrosis factor, dendritic cell-specific transmembrane protein, and circulating osteoclast precursors).

Collection of these samples will occur at the time points specified in the schedule of study assessments (Table 5–1). At dosing visits, blood samples will be drawn prior to dosing, and will be drawn at the same time of the sampling for clinical laboratory tests. The time and date of collection will be recorded in the eCRF. The samples will be stored at -80°C at the central biorepository for up to 20 years.

Instructions pertaining to sample collection, processing, storage, labeling, and shipping are provided in the laboratory manual for this study. Detailed information on sample analysis will be provided in a bioanalytical report.

# 11 ASSESSMENT OF IMMUNOLOGICAL VARIABLE(S)

Blood samples for measurement of antibodies to bimekizumab will be collected at the visits specified in Table 5–1. The threshold for antibody positivity will be defined prior to analysis.

At dosing visits, blood samples will be drawn prior to dosing, and will be drawn at the same time of the sampling for clinical laboratory tests. The time and date of collection will be recorded in the eCRF.

Instructions pertaining to sample collection, processing, storage, labeling, and shipping are provided in the laboratory manual for this study. The presence of antibodies to bimekizumab will be determined using a validated bioanalytical method. Detailed information on sample analysis will be provided in a bioanalytical report.

# 12 ASSESSMENT OF SAFETY

## 12.1 Adverse events

### 12.1.1 Definitions

### 12.1.1.1 Adverse event

An AE is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.

In order to ensure complete safety data collection, all AEs occurring during the study (ie, after the signing of the ICF), including any pretreatment and posttreatment periods required by the protocol, must be reported in the eCRF even if no IMP was taken but specific study procedures were conducted. This includes all AEs not present prior to the initial visit and all AEs that recurred or worsened after the initial visit.

Signs or symptoms of the condition/disease for which the IMP is being studied should be recorded as AEs only if their nature changes considerably or their frequency or intensity increases in a clinically significant manner as compared to the clinical profile known to the Investigator from the subject's history or the Baseline Period.

#### 12.1.1.2 Serious adverse event

Once it is determined that a subject experienced an AE, the seriousness of the AE must be determined. An SAE must meet 1 or more of the following criteria:

- (Life-threatening does not include a reaction that might have caused death had it occurred in a more severe form.)

  Significant or persistent disability/incapacity

  Congenital anomaly/birth defect (including that occurring in a fetus)

  Important medical event that, based upon appropriate medical judgment maxical patient or subject and may require medical or surgical putcomes listed in the definition.

(Important medical events may include, but are not limited to, potential Hy's Law [see Section 12.1.1.3], allergic bronchospasm requiring intensive treatment in an emergency room or at home, blood dyscrasias that do not result in inpatient hospitalization, or the development of drug dependency or drug abuse.)

Initial inpatient hospitalization or prolongation of hospitalization

(A patient admitted to a hospital, even if he/she is released on the same day, meets the criteria for the initial inpatient hospitalization. An emergency room visit that results in admission to the hospital would also qualify for the initial inpatient hospitalization criteria. However, emergency room visits that do not result in admission to the hospital would not qualify for this criteria and, instead, should be evaluated for 1 of the other criteria in the definition of serious [eg, life-threatening adverse experience, important medical event].

Hospitalizations for reasons not associated with the occurrence of an AE [eg, preplanned surgery or elective surgery for a pre-existing condition that has not worsened or manifested in an unusual or uncharacteristic manner] do not qualify for reporting. For example, if a subject has a condition recorded on his/her medical history and later has a preplanned surgery for this condition, it is not appropriate to record the surgery or hospitalization as an SAE, since there is no AE upon which to assess the serious criteria. Please note that, if the pre-existing condition has worsened or manifested in an unusual or uncharacteristic manner, this would then qualify as an AE and, if necessary, the seriousness of the event would need to be determined.)

Confirmed active TB must be reported as an SAE. The Investigator is to complete and submit the TB Follow-Up Form provided.

### 12.1.1.2.1 **Anticipated serious adverse events**

The following Anticipated SAEs are anticipated to occur in the population studied in this protocol at some frequency that is independent of drug exposure.

This list does not change the Investigator's obligation to report all SAEs (including Anticipated SAEs) as detailed in Section 12.1.2.3.

Table 12.1: Anticipated serious adverse events for the population of subjects with moderate to severe chronic plaque psoriasis

| MedDRA® system order class | MedDRA preferred term |
|---|---|
| Skin and subcutaneous tissue disorders | Any psoriatic condition HLT |
| Musculoskeletal and connective tissue disorders | Psoriatic arthropathy |

HLT=High Level Term; MedDRA=Medical Dictionary for Regulatory Activities; SAE=serious adverse event Note: Exception: Listed events will not be regarded as anticipated SAEs if they are life threatening or if they result in the death of the study subject ionsor in the death of the study subject.

#### 12.1.1.3 Adverse events of special interest

An AE of special interest (AESI) is any AE that a regulatory authority has mandated be reported on an expedited basis, regardless of the seriousness, expectedness, or relatedness of the AE to the administration of a UCB product/compound.

Potential Hy's Law, defined as  $\ge 3xULN$  ALT or AST with coexisting  $\ge 2xULN$  total bilirubin in the absence of  $\geq 2xULN$  ALP, with no alternative explanation for the biochemical abnormality, must ALWAYS be reported to UCB as an AESI (ie, without waiting for any additional etiologic investigations to have been concluded). Follow-up information should then be reported if an alternative etiology is identified during investigation and monitoring of the subject.

### Other safety topics of interest 12.1.1.4

Pre-specified safety topics of interest for the study are: infections (serious, opportunistic, fungal, and TB), neutropenia, hypersensitivity, suicidal ideation and behavior, depression, major cardiovascular events, liver function test changes/enzyme elevations, malignancies, and inflammatory bowel diseases (with gastroenterology referral, as appropriate). This is based on findings from the IMP clinical program to date, potential risks generally associated with biologic immunomodulators, or findings from other medicines with a related mechanism of action. There are no specific AE reporting requirements for these topics, however special monitoring, additional data collection activities, and/or enhanced signal detection activities (within UCB) are in place.

### Procedures for reporting and recording adverse events 12.1.2

The subject will be given the opportunity to report AEs spontaneously. A general prompt will also be given at each study visit to detect AEs. For example:

"Did you notice anything unusual about your health (since your last visit)?"

In addition, the Investigator should review any self-assessment procedures (eg, diary cards) employed in the study.

### 12:1.2.1 **Description of adverse events**

When recording an AE, the Investigator should use the overall diagnosis or syndrome using standard medical terminology, rather than recording individual symptoms or signs. The eCRF and source documents should be consistent. Any discrepancies between the subject's own words on his/her own records (eg, diary card) and the corresponding medical terminology should be clarified in the source documentation.

When recording the severity of an AE in the eCRF (ie, mild, moderate, or severe), the Investigator may refer to the Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0 (http://ctep.cancer.gov/protocolDevelopment/electronic applications/ctc.htm) for Rule for repetition of an adverse event

An increase in the intensity of an AE should lead to the repetition of the AE being reported with:

The outcome date of the first AE that is not related to the natural course of the distance of the same as the start date of the repeated AE. and the

- The AE verbatim term being the same for the first and repeated AE, so that the repeated AE can be easily identified as the worsening of the first one

### 12.1.2.3 Additional procedures for reporting serious adverse events

If an SAE is reported, UCB must be informed within 24 hours of receipt of this information by the site (see contact information for SAE reporting listed in the Serious Adverse Event Reporting section at the front of the protocol). The Investigator must forward to UCB (or its representative) a duly completed "Investigator SAE Report Form for Development Drug" (SAE report form) provided by UCB, even if the data are incomplete, or if it is obvious that more data will be needed in order to draw any conclusions. Information recorded on this form will be entered into the global safety database.

An Investigator SAE Report Form will be provided to the Investigator. The Investigator SAE Report Form must be completed in English.

It is important for the Investigator, when completing the SAE Report Form, to include the assessment as to a causal relationship between the SAE and the IMP administration. This insight from the Investigator is very important for UCB to consider in assessing the safety of the IMP and in determining whether the SAE requires reporting to the regulatory authorities in an expedited manner.

Additional information (eg. autopsy or laboratory reports) received by the Investigator must be provided within 24 hours. All documents in the local language must be accompanied by a translation in English, or the relevant information included in the same document must be summarized in the Investigator SAE Report Form.

The Investigator is specifically requested to collect and report to UCB (or its representative) any SAEs (even if the Investigator is certain that they are in no way associated with the IMP), up to 30 days from the end of the study for each subject, and to also inform participating subjects of the need to inform the Investigator of any SAE within this period. Serious AEs that the Upon receipt of the SAE Report Form, UCB will perform an assessment of expectedness of the reported SAE. The assessment of the expectedness of the SAE is based on the ID

#### 12.1.3 Follow up of adverse events

An AE should be followed until it has resolved, has a stable sequelae, the Investigator determines that it is no longer clinically significant, or the subject is lost to follow up. This

n an AE is ongoing at the end of the study for a subject, follow up should be provided until resolution/stable level of sequelae is achieved, or until the Investigator no longer deems that it is clinically significant, or until the subject is lost to follow up. If no follow up is provided, the Investigator must provide a justification. The follow up will usually be after the subject has discontinued his/her INTE

Information on SAEs obtained after clinical database lock will be captured through the Patient Safety (PS) database without limitation of time.

#### 12.1.4 **Pregnancy**

If an Investigator is notified that a subject has become pregnant after the first intake of any IMP, the Investigator must immediately notify UCB's PS department by providing the completed Pregnancy Report and Outcome Form (for contact details see Serious Adverse Event reporting information at the beginning of this protocol). The subject should be withdrawn from the study as soon as pregnancy is known (by positive pregnancy test), and the following should be completed:

- The subject should return for an early discontinuation visit.
- The subject should immediately stop the intake of the IMP.
- A SFU Visit should be scheduled 20 weeks after the subject has discontinued her IMP.

The Investigator must inform the subject of information currently known about potential risks and about available treatment alternatives.

The pregnancy will be documented on the Pregnancy Report and Outcome Form provided to the Investigator. The progression of the pregnancy and the eventual birth (if applicable) must be followed up using the Pregnancy Report and Outcome Form in which the Investigator has to report on the health of the mother and of the child. Every reasonable attempt should be made to follow the health of the child for 30 days after birth for any significant medical issues. In certain circumstances, UCB may request that follow up is continued for a period longer than 30 days. If the subject is lost to follow up and/or refuses to give information, written documentation of attempts to contact the subject needs to be provided by the Investigator and filed at the site. UCB's PS department is the primary contact for any questions related to the data collection for the pregnancy, eventual birth, and follow up.

In cases where the partner of a male subject enrolled in a clinical study becomes pregnant, the Partner Pregnancy Consent form that has been approved by the responsible IRB/IEC and should be available in the Investigator site file. In case of questions about 41. Investigator may contact the UCB/contract research organization (CRO) contract monitor for the study. The Investigator will complete the Pregnancy Report and Outcome form and send it to UCB's PS department (for contact details see Serious Adverse Event reporting information at the

beginning of this protocol) only after the partner has agreed that additional information can be captured and has provided the signed Partner Pregnancy Consent form. UCB's PS department is also the primary contact for any questions related to the data collection for the partner pregnancy, eventual birth, and follow-up.

A pregnancy becomes an SAE in the following circumstances: miscarriage, elective abortion when medically indicated (e.g. when pregnancy is endangering life or health of woman or when fetus will be born with severe abnormalities), unintended pregnancy after hormonal contraceptive failure (if the hormonal contraceptive was correctly used), ectopic pregnancy, fetal demise, or any congenital anomaly/birth defect of the baby. Those SAEs must be additionally reported using the Investigator SAE Report Form.

Should a subject become pregnant while participating in the study the cultivation option to enroll in a separate of

Should a subject become pregnant while participating in the study, the subject may be offered the option to enroll in a separate observational pregnancy follow-up study sponsored by UCB and conducted independently from study PS0008. If the study is available locally, the PS0008 Investigator will be provided with locally approved information about the observational pregnancy follow-up study to inform the subject at the time the pregnancy is reported. Participation in this separate study will be voluntary and will not impact the therapeutic management of the subject nor interfere with termination and follow-up procedures as described in protocol PS0008.

# 12.1.5 Suspected transmission of an infectious agent via a medicinal product

For the purposes of reporting, any suspected transmission of an infectious agent via a medicinal product should be considered as an SAE; such cases must be reported immediately, recorded in the AE module of the eCRF, and followed as any other SAE. Any organism, virus, or infectious particle (eg, prion protein transmitting transmissible spongiform encephalopathy), pathogenic or nonpathogenic, is considered an infectious agent.

### 12.1.6 Overdose of investigational medicinal product

Excessive dosing (beyond that prescribed in the protocol and including overdose) should be recorded in the eCRF. Any SAE or nonserious AE associated with excessive dosing must be followed as any other SAE or nonserious AE. These events are only considered AEs or SAEs if there are associated clinical signs and symptoms or if the act of taking the excess medicine itself is an AE or SAE (eg, suicide attempt).

# 12.1.7 Safety signal detection

Selected data from this study will be reviewed periodically to detect as early as possible any safety concern(s) related to the IMP so that Investigators, clinical study subjects, regulatory authorities, and IRBs/IECs will be informed appropriately and as early as possible.

In addition, an independent Data Monitoring Committee (DMC) will periodically review and monitor safety data from this study and advise UCB. Details are provided in the DMC Charter.

Cardiovascular and Neuropsychiatric Adjudication Committees will also periodically review and monitor safety data from this study and advise UCB. Details are provided in the Adjudication Committee Charters.

The Study Physician or medically qualified designee/equivalent will conduct an ongoing review of SAEs and perform ongoing SAE reconciliations in collaboration with the PS representative.

Laboratory measurements

Clinical laboratory assessments consist of serum chemistry, hematology, urinalysis, and urine drug screen. A centralized laboratory will be used to supply all laboratory test supplies and analyze all blood and urine samples for hematology, biochemistry, and urine to rule out hepatitis B, hepatitis C and the partition of the property of the partition of performed at Screening in addition to those measurements listed in Table 12–2.

Specific details regarding the handling and processing of serum chemistry, hematology, and urinalysis samples are provided in the study laboratory manuals.

The following laboratory parameters will be measured:

Table 12–2: Laboratory measurements

| Hematology | Chemistry | <b>U</b> rinalysis dipstick <sup>a</sup> |
|---|---|---|
| Basophils | Calcium | pH |
| Eosinophils | Chloride Chloride | Albumin (protein) |
| Lymphocytes | Magnesium | Glucose |
| Monocytes | Potassium | Blood |
| Neutrophils | Sodium | Leukocyte esterase |
| Hematocrit | Glucose | Nitrite |
| Hemoglobin | BUN | Urine dipstick for pregnancy testing <sup>b</sup> |
| MCH SUP | Creatinine | Urine drug screen <sup>c</sup> |
| MCHC | ALP | |
| MCV | AST | |
| Platelet count | ALT | |
| RBC count | GGT | |
| WBC count | Total bilirubin | |
| | Serum pregnancy testing <sup>a</sup> | C DIDITI |

ALP=alkaline phosphatase; ALT=alanine aminotransferase; AST=aspartate aminotransferase; BUN=blood urea nitrogen; GGT=gamma-glutamyltransferase; MCH=mean corpuscular hemoglobin; MCHC=mean corpuscular hemoglobin concentration; MCV=mean corpuscular volume; PEOT=Premature End of Treatment; RBC=red blood cell; SFU=Safety Follow-Up; WBC=white blood cell


Evaluation of PDILI

The PDILI IMP discontinuation criteria for this study are provided in Section 6.3.1, with the accompanying required follow-up investigation and monitoring detailed below. All PDILI eventmust be reported as an AE and reported to the study site and Sponsor with reported as an AESI (see Section 6.3.1). Section 12.1.1.2).

Evaluation of PDILI consists of the diagnostic testing and continued monitoring included in Table 12–3 (specific tests dependent on laboratory results and corresponding symptoms) and consultation with a local hepatologist (if applicable; discussed in Section 12.2.1.1). The local hepatologist is the expert usually consulted by the treating physician for assessment and management of potential hepatic disease. This would usually be a hepatologist, but may be a gastroenterologist. Additional investigation and monitoring may be required and adapted based on the diagnosis after the cause of the liver injury/abnormality is confirmed (details in Section 12.2.1.4).

The results of all monitoring, including laboratory testing and other testing, should be made available to the study site and Sponsor.

All initial tests resulting in abnormal hepatic laboratory values need to be repeated, but appropriate medical action must not be delayed waiting for the repeat result.

If tests are done locally for more rapid results, a concurrent sample should also be sent to the central laboratory whenever possible. Medical care decisions are to be made initially using the most rapidly available results and a conservative approach must be taken if the results from the 2 laboratory tests are significantly different. Data from the local and central laboratory are to be recorded on the applicable eCRF pages.

When IMP is discontinued, all concomitant medications and herbal supplements that are not medically necessary should also be discontinued. In these cases, the Investigator should also consider dose reduction for medically necessary concomitant medication and consider changing any medically required concomitant medication known to be hepatotoxic to a suitable alternative

When MP is stopped due to PDILI (as described in Section 6.3.1), IMP must be permanently discontinued unless a subsequent alternative diagnosis fully explains the hepatic findings. If a subsequent alternative diagnosis fully explains the hepatic findings, and the requirements provided in Section 12.2.1.2.1 are met, rechallenge with IMP may be appropriate.

Table 12–3 summarizes the approach to investigate PDILI.

Table 12–3: Required investigations and follow-up for PDILI

| UCB Clinical Study Protocol Table 12–3: Required investigation | | | Bimekizumab s and follow-up for PDILI | | | 96 Apr 20:<br>PS000 |
|---|---|---|---|---|---|---|
| Laborat | ory value | | Immediate | | Follow up | |
| ALT or<br>AST | Total<br>bilirubin | Symptoms of hepatitis of hypersensitivity | Consultation requirements | Actions | Testing Relations | Evaluation |
| ≥3xULN | ≥2xULN <sup>b</sup> | NA | Hepatology consult | Immediate, | Essential: Must have | Monitoring of liver |
| ≥3xULN | NA | Yes | Medical Monitor must<br>be notified within<br>24 hours (eg, by<br>laboratory alert) and<br>subject discussed with<br>Medical Monitor<br>ASAP. | permanent IMP discontinuation. | repeat liver<br>chemistry values<br>and additional<br>testing completed<br>ASAP (see<br>Section 12.2.1.3);<br>recommended to | chemistry values at least<br>twice per week until<br>values normalize,<br>stabilize, or return to<br>within baseline values. <sup>d</sup> |
| ≥8xULN | NA | NA | Need for hepatology consult to be discussed (required if ALT or AST ≥8xULN). Medical Monitor must be notified within 24 hours (eg, by laboratory alert) and subject discussed with Medical Monitor ASAP | Immediate, permanent IMP discontinuation. | occur at the site with HCP. | |

Table 12–3: Required investigations and follow-up for PDILI

| UCB<br>Clinical Study<br>Table 12- | | ed investigation | Bim<br>s and follow-up for | ekizumab<br>PDILI | | 96 Apr 2018<br>PS0008 |
|---|---|---|---|---|---|---|
| Laborat | ory value | | Immediate | | Follow up | |
| ALT or<br>AST | Total<br>bilirubin | Symptoms of hepatitis of hypersensitivity | Consultation requirements | Actions | Testing Lensions | Evaluation |
| ≥5xULN<br>(and ≥2x<br>baseline)<br>and<br><8xULN | <2xULN | No No | Discussion with Medical Monitor required. Consider need for hepatology consult if there is no evidence of resolution (see Follow up requirements).c | Further investigation — immediate IMP discontinuation not required (see Section 12.2.1.2). IMP discontinuation required if any of the following occur: Subject cannot comply with monitoring schedule. Liver chemistry values continue to increase. Liver chemistry values remain ≥5xULN (and ≥2x baseline) after 4 weeks of monitoring without evidence of resolution. | Essential: Every attempt must be made to have repeat liver chemistry values and additional testing completed within 48 hours at the site with HCP (see Section 12.2.1.3). | Monitoring of liver chemistry values at least twice per week for 2 weeks.d • Immediate IMP discontinuation required if liver chemistry values continue to increase. After 2 weeks of monitoring liver chemistry values: • ALT or AST remains ≥5xULN <8xULN, IMP should be temporarily withheld and subject should undergo repeat test in 2 weeks. Continue IMP if ALT or AST values <5xULN; continue to monitor at least twice per week until values normalize, stabilize, |

### Table 12-3: Required investigations and follow-up for PDILI

| Laboratory value | | | Immediate | | Fo | llow up |
|---|---|---|---|---|---|---|
| ALT or<br>AST | Total<br>bilirubin | Symptoms of hepatitis of hypersensitivity | Consultation requirements | Actions | Testing | Evaluation |
| | | | | | and any of | or return to within baseline values. |
| | | | | ED COPY application | , alle | If ALT or AST remains ≥5xULN after second re-test, immediate, permanent IMP discontinuation required. |
| | | | RELING OF | Litho | | Continue to monitor until values normalize, stabilize, or return to within baseline values. <sup>d</sup> |

ALP=alkaline phosphatase; ALT=alanine aminotransferase; ASAP=as soon as possible; AST=aspartate aminotransferase; HCP=healthcare practitioner; IMP=investigational medicinal product; NA=not applicable; PDILI=potential drug-induced liver injury; ULN=upper limit of normal

<sup>&</sup>lt;sup>a</sup> Hepatitis symptoms include fatigue, nausea, vomiting, and right upper quadrant pain or tenderness; hypersensitivity symptoms include eosinophilia (>5%), rash, and fever (without clear alternative cause).

<sup>&</sup>lt;sup>b</sup> If the subject also has ≥2xULN ALP, the possibility of an indication of biliary obstruction should be discussed with the Medical Monitor.

<sup>&</sup>lt;sup>c</sup> Details provided in Section 12.2.1.1. The local hepatologist is the expert usually consulted by the treating physician for assessment and management of potential hepatic disease. This would usually be a hepatologist, but may be a gastroenterologist.

<sup>&</sup>lt;sup>d</sup> Unless an alternative monitoring schedule is agreed by the Investigator and UCB responsible physician. Determination of stabilization is at the discretion of the Investigator in consultation with the hepatologist (as applicable) and UCB responsible physician, as needed.

#### 12.2.1.1 Consultation with Medical Monitor and local hepatologist

Potential drug-induced liver injury events require notification of the Medical Monitor within sions or variations thereof 24 hours (eg, by laboratory alert), and the subject must be discussed with the Medical Monitor as soon as possible. If required, the subject must also be discussed with the local hepatologist. The local hepatologist is the expert usually consulted by the treating physician for assessment and management of potential hepatic disease. This would usually be a hepatologist, but may be a gastroenterologist. If determined necessary, this discussion should be followed by a full hepatology assessment (see Section 12.2.1.3) and SAE report (if applicable).

#### 12.2.1.2 Immediate action: determination of IMP discontinuation

All PDILI events require immediate action, testing, and monitoring.

The immediate action is dependent on the laboratory values and symptoms of hepatitis or hypersensitivity and ranges from continuation of IMP (followed by immediate investigation) to immediate and permanent discontinuation (see Section 6.3.1 and Table 12–3 for details).

When IMP is discontinued, all concomitant medications and herbal supplements that are not medically necessary should also be discontinued. The Investigator should also consider dose reduction for medically necessary concomitant medication and consider changing any medically required concomitant medication known to be hepatotoxic to a suitable alternative.

#### 12.2.1.2.1 IMP restart/rechallenge

Rechallenge with IMP can occur only if ALL of the following requirements are met:

- The results of additional testing and monitoring described in Section 12.2.1.3 and Section 12.2.1.4 confirm a nondrug-related cause for the abnormal hepatic laboratory parameters and any associated symptoms (ie, a subsequent alternative diagnosis fully explains the hepatic findings).
- The subject has shown clear therapeutic benefit from the IMP.
- Subject's ALT or AST elevations do not exceed  $\geq 5xULN$ .
- Subject's total bilirubin is <2xULN.
- Subject has no signs or symptoms of hypersensitivity or hepatitis.
- The rechallenge is approved by the UCB responsible physician, DMC, and a hepatologist. The hepatologist must be external to UCB but may be a member of the DMC. It is recommended that the hepatologist be a local hepatology expert or the hepatologist treating the subject.
- Subject agrees to the Investigator-recommended monitoring plan.

### 12,2,1.3 Testing: identification/exclusion of alternative etiology

The measurements and additional information required for the assessment of PDILI events when there is a reasonable possibility that they may have been caused by the IMP are detailed in Table 12–4 (laboratory measurements) and Table 12–5 (additional information). Results of the laboratory measurements and information collected are to be submitted to the Sponsor on the corresponding eCRF. If the medical history of the subject indicates a requirement for other

assessments not included below, these additional assessments should be completed and submitted, as applicable.

All blood samples should be stored, if possible. If tests are done locally for more rapid results, a concurrent sample must also be sent to the central laboratory.

The following measurements are to be assessed:

Table 12–4: PDILI laboratory measurements

| Virology-related | Hepatitis A IgM antibody |
|---|---|
| | HBsAg |
| | Hepatitis E IgM antibody |
| | HBcAb-IgM |
| | Hepatitis C RNA |
| | Cytomegalovirus IgM antibody |
| | Epstein-Barr viral capsid antigen IgM antibody (if unavailable, obtain heterophile antibody or monospot testing) |
| Immunology | Anti-nuclear antibody (qualitative and quantitative) |
| | Anti-smooth muscle antibody (qualitative and quantitative) |
| | Type 1 anti-liver kidney microsomal antibodies (qualitative and quantitative) |
| Hematology | Eosinophil count |
| Urinalysis | Urine drug screen |
| Chemistry | Amylase |
| | Sodium, potassium, chloride, glucose, BUN, creatinine |
| | Total bilirubin, ALP, AST, ALT, GGT, total cholesterol, albumin |
| | If total bilirubin ≥1.5xULN, obtain fractionated bilirubin to obtain % direct bilirubin |
| ,10 | Serum CPK and LDH to evaluate possible muscle injury causing transaminase elevation |
| Additional | Prothrombin time/INR <sup>b</sup> |
| , pe | Serum pregnancy test <sup>c</sup> |
| anno | PK |
| ATD a'fil' 1' 1 1 . | A I T-glaning amingtransferage: A ST-generate amingtransferage: PI IN-blood uran |

ALP=alkaline phosphatase; ALT=alanine aminotransferase; AST=aspartate aminotransferase; BUN=blood urea nitrogen; CPK=creatine phosphokinase; GGT=gamma glutamyl transferase; HBcAb-IgM=hepatitis B core antibody-IgM; HBsAg=hepatitis B surface antigen; IgM=immunoglobulin M; INR=international normalized ratio; LDH=lactate dehydrogenase; PDILI=potential drug-induced liver injury; PK=pharmacokinetic; RNA=ribonucleic acid; ULN=upper limit of normal

### Table 12–4: PDILI laboratory measurements

- <sup>a</sup> Tests in addition to the specified analytes may be performed based on the Investigator's medical judgment and subject history.
- ions or variations thereof <sup>b</sup> Measured only for subjects with ALT >8xULN, elevations in total bilirubin, and symptoms of hepatitis or hypersensitivity. Hepatitis symptoms include fatigue, nausea, vomiting, and right upper quadrant pain or tenderness; hypersensitivity symptoms include eosinophilia (>5%), rash, and fever (without clear alternative
- <sup>c</sup> For women of childbearing potential.

The following additional information is to be collected:

### Table 12–5: PDILI information to be collected

### New or updated information

Concomitant prescription and over-the-counter medications (eg. acetaminophen, herbal remedies, vitamins); dosages and dates should be included.

Pertinent medical history, including the following:

- History of liver disease (eg, autoimmune hepatitis, nonalcoholic steatohepatitis or other "fatty liver disease")
- Adverse reactions to drugs
- Allergies
- Relevant family history or inheritable disorders (eg.) Gilbert's syndrome, alpha-1 antitrypsin deficiency)
- Recent travel

Progression of malignancy involving the liver (Note: Metastatic disease to the liver, by itself, should not be used as an explanation for significant AST and/or ALT elevations.)

The appearance or worsening of clinical symptoms of hepatitis or hypersensitivity (eg., fatigue, nausea, vomiting, right upper quadrant pain or tenderness, decreased appetite, abdominal pain, jaundice, fever, or rash)

Recent clinically significant hypotension or hypoxemia with compromised cardiopulmonary function

Alcohol and illicit drug use

Results of liver imaging or liver biopsy, if done

Results of any specialist or hepatology consult, if done

Any postmortem/pathology reports

ALT=alanine aminotransferase; AST=aspartate aminotransferase; PDILI=potential drug-induced liver injury

Table 12–3. Monitoring should continue until liver chemistry values normalize, stabilize, or return to Baseline. Determination of stabilization is at the discretion of the Investigation with the hepatologist (as applied 1). consultation with the hepatologist (as applicable) and UCB responsible physician, as needed.

### 12.3 Other safety measurements

#### 12.3.1 Assessment and management of TB and TB risk factors

At Screening, all subjects will have an IGRA test (QuantiFERON TB test is recommended), a chest x-ray (unless already performed within 3 months of Screening) and examination for signs and symptoms of TB. In addition, each subject will complete a TB questionnaire directed at potential exposure and symptoms of TB.

For the purposes of this study, TB definition.

- a. Known TB infection:
  - Active TB infection or clinical signs and symptoms suspicious for TB (pulmonary or extra-pulmonary).
  - History of active TB infection involving any organ system or findings in other organ systems consistent with TB infection, unless adequately treated and proven to be fully recovered upon consult with a TB specialist.
  - Any evidence by radiography or other imaging modalities consistent with previously active TB infection that is not reported in the subject's medical history.
- b. High risk of acquiring TB infection:
  - Known close exposure to another person with active TB infection within the 3 months prior to Screening.
  - Time spent in a healthcare delivery setting or institution where individuals infected with TB are housed and where the risk of transmission of infection is high.
- c. Latent TB infection (unless appropriate prophylaxis is initiated at least 8 weeks prior to IMP dosing and continued to completion of prophylaxis):
  - The absence of signs, symptoms, or physical findings suggestive of TB infection with a positive IGRA test (or 2 indeterminate IGRA test results) and a chest x-ray (or other imaging) without evidence of TB infection. If the result of the IGRA test is indeterminate, the particular IGRA test previously performed may be repeated once; if positive or indeterminate on retest, the subject may not be randomized to IMP without further evaluation by a TB specialist and discussion with the Study Physician, if LTB infection is identified. The retest must be done during the protocol-defined Screening window.

Note: If available, respiratory or other specimens must also be smear and culture negative for TB (CDC diagnosis of LTB infection) http://www.cdc.gov/TB/topic /testing/default.htm).

- d. NTMB infection is defined as a clinical infection caused by mycobacterial species other than those belonging to the Mycobacterium tuberculosis complex.
- Tuberculosis test conversion:

The december taken to support any management and produce the support of the suppo

Figure 12-1: Schematic diagram of TB test results and study eligibility



IGRA=interferon-gamma release assay; TB=tuberculosis

<sup>&</sup>lt;sup>a</sup> IGRA retest must be done during the protocol-defined Screening window

<sup>&</sup>lt;sup>b</sup> Subjects with LTBI may enter the study only after they have completed at least 8 weeks of appropriate prophylactic therapy and thereafter, will continue and complete the entire regimen.

### 12.3.1.1 Tuberculosis assessment by IGRA

During conduct of the study, the TB assessment by IGRA (QuantiFERON TB test is recommended) will be performed as described in Table 5–1 for all subjects. The test results will be reported as positive, negative, or indeterminate. Positive and indeterminate TB test results must be reported as an AE and appropriately updated once the final diagnosis is known (e.g. active TB, latent TB, or false positive TB test). UCB also recommends that a TB specialist be consulted where TB (latent or active) is suspected or if there are doubts regarding test results. If latent or active TB is identified, subject must undergo appropriate study-specified withdrawal procedures. The retest during Screening must be done during the protocol-defined Screening window.

### 12.3.1.2 Chest x-ray for tuberculosis

A plain posteroanterior chest x-ray must be performed in the Screening Period unless one has been performed within 3 months prior to the Screening Visit. The chest x-ray (or, if done, Computed Axial Tomography [CAT] of the Chest) must be clear of signs of TB infection (previous or current) before first IMP administration. All chest imaging (particularly x-rays) should be available for review by the Investigator before randomization of the subject. The chest x-ray reading should be repeated if the TB test was confirmed positive. If the second read of the pretreatment chest x-ray is confirmed to be clear, the subject may be included in the study 8 weeks after the start of the TB prophylactic treatment. If the pretreatment chest x-ray is not available for a re-read, it should be repeated after notification to the radiologist that this subject is IGRA positive, and confirmed to be clear for signs of TB.

The chest imaging must be negative for any old or recent TB infection as determined by a qualified radiologist and/or pulmonary physician. Any new clinically significant findings post Baseline on chest x-ray must be documented in the source documents and the eCRF as an AE.

### 12.3.1.3 Tuberculosis questionnaire

The questionnaire "Evaluation of signs and symptoms of tuberculosis" should be used as a source document. The questionnaire will be completed as described in Table 5–1. The questionnaire will assist with the identification of subjects who may require therapy for TB. A subject who answers "Yes" to the question "Has the subject been in close contact with an individual with active TB, or an individual who has recently been treated for TB?" at Screening is excluded. A "Yes" response to any of the other questions within the questionnaire at Screening should trigger further careful assessment to determine if subject has LTB or active TB (see Exclusion Criterion #12 Section 6.2). A "Yes" response to any of the questions during the study should trigger further assessments to determine if the subject has either LTB or active TB infection.

### 12.3.1.4 Tuberculosis management

During the study, subjects who develop evidence of LTB infection or active TB must immediately stop further administration of IMP and will be referred to an appropriate TB specialist (pulmonologist or infectious disease specialist) for further evaluation. Evidence of LTB infection is defined as subject's IGRA test converts to positive or indeterminate (and confirmed indeterminate on repeat), or the subject's questionnaire or history and physical indicates that TB infection or exposure may have occurred. Evidence of active TB includes, in addition to the aforementioned tests, signs and symptoms of organ involvement. In either situation, the subject should be carefully assessed by a TB specialist for active TB. Subjects diagnosed with active TB should be withdrawn from the study and receive appropriate TB or prophylaxis therapy.

If a TB specialist excludes an active TB infection the subject can proceed with the MP no earlier than 4 weeks after the start of an appropriate prophylactic therapy.

Any presumptive diagnosis or diagnosis of a TB infection is a reportable event. Confirmed active TB must be reported as an SAE. The Investigator is to complete and submit the TB Follow-Up Form provided.

The subject should be transferred to the care of his/her physician and managed according to the best available standard of care. Subjects identified as having converted to active TB during the study must be withdrawn and scheduled to return for the PEOT Visit as soon as possible but no later than the next scheduled study visit and complete all PEOT Visit assessments.

The subject should be encouraged to complete a SFUV isit (20 weeks after the final dose of IMP).

If infection with NTMB is identified during the study, the same procedure as for active TB acquired during the study must be followed

# 12.3.2 Pregnancy testing

Pregnancy testing will consist of serum testing at the Screening Visit. The pregnancy test will be urine at all other visits.

The Screening Visit serum pregnancy testing results must be negative and received and reviewed prior to randomization. A negative urine pregnancy test result should be obtained immediately prior to each administration of IMP at the visits specified in Table 5–1. Pregnancy tests should be administered to all female subjects of childbearing potential, regardless of their use of birth control.

# 12.3.3 Vital signs

Vital signs will be collected at every visit and will include systolic and diastolic BP, pulse rate, and body temperature (oral, axillary, or otic). Subjects should be sitting for 5 minutes before and during vital signs assessments.

Vital signs are to be measured prior to blood sampling, and prior to dosing, where applicable.

# 12.3.4 12-lead electrocardiograms

Twelve-lead standard ECGs will be recorded at the visits specified in Table 5–1, and read by a central ECG reader.

Full details of ECG recording will be provided in the ECG Manual.

#### 12.3.5 Physical examination

Wextensions of variations thereof. A physical examination will be performed at the visits specified in Table 5–1. The physical examination will include general appearance; ear, nose, and throat; eyes, hair, and skin; respiratory; CV; GI; musculoskeletal; hepatic; neurological (including limb reflexes); and mental status. All physical examinations will also include evaluation of signs and symptoms of active TB and risk for exposure to TB. Findings considered clinically significant changes since the physical examination at the Screening Visit will be recorded as AEs.

#### 12.3.6 Height and body weight

Height will be measured at Baseline only.

Body weight will be measured at the visits specified in Table 5–1.

#### 12.3.7 Assessment of suicidal ideation and behavior

Suicidal ideation and behavior will be assessed by using the eC-SSRS; the questionnaire will be self-administered by the subject and assessed by trained study personnel. This scale will be used to assess suicidal ideation and behavior that may occur during the study. The visits at which the eC-SSRS assessments will be performed are specified in the schedule of study assessments (Table 5–1).

The eC-SSRS is a standardized and validated instrument developed for the assessment of the severity and frequency of suicidal ideation and behavior (Posner et al, 2011; Mundt et al, 2010). Subjects respond to standardized clinical questions that are presented in a uniform fashion. The eC-SSRS defines 5 subtypes of suicidal ideation and behavior in addition to self-injurious behavior with no suicidal intent. The eC SSRS takes approximately 3 to 10 minutes to complete.

Refer to Section 6.3 for eC-SSRS-related withdrawal criteria.

#### 12.4 Other study measurements

### **Demographic information** 12.4.1

Demographic information will be collected in all subjects and include age, gender, race, and ethnicity. Information on demographics will be collected according to local rules and regulations. Demographic information will be recorded in the eCRF.

### Medical History 12.4.2

A complete medical history will be collected as part of the Screening assessment and include all clinically relevant past or coexisting medical conditions and surgeries. Findings will be recorded in the eCRF.

### 12.4.3 **Psoriasis History**

and past treatments for PSO.

12.4.4

Data A detailed history of each subject's PSO history will be collected and include the date of onset

### **Data Monitoring and Adjudication Committees**

The DMC membership includes experienced clinicians and a statistician, all of whom have expertise in clinical trials. Cardiovascular and Neuropsychiatric Adjudication Committees will

 also periodically review data from this trial. Both Data Monitoring and Adjudication Committee members may not participate in the study as principal or co-Investigators, or as study subject care physicians. The duration of membership for the committees will be inclusive of planned analyses for PS0008. Detailed role, scope, responsibilities, and complete procedures, as well as the identity of members, are described in the separate committee charters.

### 13 STUDY MANAGEMENT AND ADMINISTRATION

### 13.1 Adherence to protocol

The Investigator should not deviate from the protocol. However, the Investigator should take any measure necessary in deviation from or not defined by the protocol in order to protect clinical study subjects from any immediate hazard to their health and safety. In this case, this action should be taken immediately, without prior notification of the regulatory authority, IRB/IEC, or Sponsor.

After implementation of such measure, the Investigator must notify the CPM of the Sponsor within 24 hours and follow any local regulatory requirements.

# 13.2 Monitoring

UCB (or designee) will monitor the study to meet the Sponsor's monitoring SOPs, ICH-GCP guideline, and applicable regulatory requirements, and to ensure that study initiation, conduct, and closure are adequate. Monitoring of the study may be delegated by UCB to a CRO or a contract monitor.

The Investigator and his/her staff are expected to cooperate with UCB (or designee) and to be available during the monitoring visits to answer questions sufficiently and to provide any missing information. The Investigator(s)/institution(s) will permit direct access to source data/documents for study-related monitoring, audits, IRB/IEC review, and regulatory inspection(s).

The Investigator will allow UCB (or designee) to periodically review all CRFs and corresponding source documents (eg, hospital and laboratory records for each subject). Monitoring visits will provide UCB (or designee) with the opportunity to evaluate the progress of the study, verify the accuracy and completeness of CRFs, ensure that all protocol requirements, applicable authorities regulations, and Investigator's obligations are being fulfilled, and resolve any inconsistencies in the study records.

### 13.2.1 Definition of source data

All source documents must be accurate, clear, unambiguous, permanent, and capable of being audited. Source documentation should be made using some permanent form of recording (ink, typing, printing, optical disc). They should not be obscured by correction fluid or have temporary attachments (such as removable self-stick notes). Photocopies and/or print-outs of e-CRFs are not considered acceptable source documents.

Source documents are original records in which raw data are first recorded. These may include hospital/clinic/general practitioner records, charts, diaries, x-rays, laboratory results, printouts, pharmacy records, care records, ECG or other printouts, completed scales, or QOL questionnaires, for example. Source documents should be kept in a secure, limited access area.


Source documents that are computer-generated and stored electronically must be printed for review by the monitor (eg, ECG reports). Once printed, these copies should be signed and dated by the Investigator and become a permanent part of the subject's source documents. The Investigator will facilitate the process for enabling the monitor to compare the content of the printout and the data stored in the computer to ensure all data are consistent.

Electronic data records, such as Holter monitor records or electroencephalogram records, must be saved and stored as instructed by UCB (or designee).

Patient-reported outcome measures (eg, DLQI, EQ-5D-3L, SF-36, Patient Global Assessment of PSO, and PGADA) and ePRO diary data will be entered electronically by the subject.

The ePRO diary data will be entered into an electronic diary by the subject. The data collection and database management system will be supplied by a vendor and will be compliant with the US Food and Drug Administration (FDA) Part 11. The data collected on the ePRO diary will be uploaded to a central server database and will be sent electronically to UCB (or a designated CRO).

### 13.2.2 Source data verification

Source data verification ensures accuracy and credibility of the data obtained. During monitoring visits, reported data are reviewed with regard to being accurate, complete, and verifiable from source documents (eg, subject files, recordings from automated instruments, tracings [ECG], x-ray films, laboratory notes). All data reported on the eCRF should be supported by source documents, unless otherwise specified in Section 13.2.1.

### 13.3 Data handling

# 13.3.1 Case Report Form completion

The Investigator is responsible for prompt reporting of accurate, complete, and legible data in the eCRFs and in all required reports.

Any change or correction to the eCRF after saving must be accompanied by a reason for the change.

Corrections made after the Investigator's review and approval (by means of a password/electronic signature) will be reapproved by the Investigator.

The Investigator should maintain a list of personnel authorized to enter data into the eCRF.

Detailed instructions will be provided in the eCRF Completion Guidelines.

# 13.3.2 Database entry and reconciliation

Case Report forms/external electronic data will be entered/loaded into a validated electronic database using a clinical data management system (CDMS). Computerized data cleaning checks will be used in addition to manual review to check for discrepancies and to ensure consistency of the data. This study is performed using Electronic Data Capture: the data are entered into the eCRFs once and are subsequently verified.

An electronic audit trail system will be maintained within the CDMS to track all data changes in the database once the data have been saved initially into the system or electronically loaded. Regular backups of the electronic data will be performed.

### 13.3.3 Subject Screening and Enrollment log/Subject Identification Code list

The subject's screening and enrollment will be recorded in the Subject Screening and Enrollment

UCB reserves the right to temporarily suspend or prematurely discontinue this study either at a single site, multiple sites, or at all sites at any time for reasons including, but not himted to, safety or ethical issues, inaccurate or incomplete data recording, noncompliance, or unsatisfactory enrollment with respect to quality or quantity.

If the study is prematurely terminated or suspended. LICE nvestigators/institutions and the regulators reason(s) for the termination of the study is prematurely terminated or suspended. LICE nvestigators/institutions and the regulators regularement(s) The remination of the study is prematurely terminated or suspended. LICE nvestigators/institutions are respectively. termination or suspension by the Sponsor or by the Investigator/institution, as specified by the applicable regulatory requirement(s). In addition, arrangements will be made for the return of all unused IMP and other material in accordance with UCB procedures for the study.

### Archiving and data retention 13.5

The Investigator will maintain adequate records for the study, including CRFs, medical records, laboratory results, Informed Consent documents, drug dispensing and disposition records, safety reports, information regarding participants who discontinued, and other pertinent data.

All essential documents are to be retained by the Investigator until at least 2 years after the last approval of a marketing application in an ICH region and until there are no pending or contemplated marketing applications in an ICH region, or at least 2 years have elapsed since the formal discontinuation of clinical development of the IMP. These documents should be retained for a longer period, however, if required by the applicable regulatory requirement(s) or by an agreement with UCB (Committee for Proprietary Medicinal Products [CPMP]/ICH/135/95, 2002 [Section 4.9.5]). The Investigator will contact UCB for authorization prior to the destruction of any study records or in the event of accidental loss or destruction of any study records. The Investigator will also notify UCB should he/she relocate or move the study-related files to a location other than that specified in the Sponsor's trial master file.

### 13.6 **Audit and inspection**

The Investigator will permit study-related audits mandated by UCB, after reasonable notice, and inspections by domestic or foreign regulatory authorities.

The main purposes of an audit or inspection are to confirm that the rights and well-being of the subjects enrolled have been protected, that enrolled subjects (ie, signing consent and undergoing study procedures) are appropriate for the study, and that all data relevant for the evaluation of the

IMP have been processed and reported in compliance with the planned arrangements, the protocol, investigational site, and IRB/IEC SOPs, ICH-GCP, and applicable regulatory requirements.

Valiations the reof The Investigator will provide direct access to all study documents, source records, and source data. If an inspection by a regulatory authority is announced, the Investigator will immediately inform UCB (or designee).

#### 13.7 **Good Clinical Practice**

Noncompliance with the protocol, ICH-GCP, or local regulatory requirements by the Investigator, institution, institution staff, or designees of the Sponsor will lead to prompt action by UCB to secure compliance. Continued noncompliance may result in the termination of the site's involvement in the study.

#### 14 **STATISTICS**

A description of statistical methods follows and will be described in more detail in SAP.

#### 14.1 **Definition of analysis sets**

The Enrolled Set (ES) will consist of all subjects who have given informed consent.

The Randomized Set (RS) will consist of all randomized subjects.

The Safety Set (SS) will consist of all subjects that received at least 1 dose of the IMP.

The Bimekizumab Set (BKZ Set) will consist of all subjects who have received at least 1 dose of bimekizumab in this study.

The Full Analysis Set (FAS) will consist of all randomized subjects that receive at least 1 dose of the IMP and have a valid measurement for each of the co-primary efficacy variables at Baseline.

The Per-Protocol Set (PPS) will consist of all subjects in the RS who had no important protocol deviations affecting the primary efficacy variable. Important protocol deviations will be predefined and subjects with important protocol deviations will be evaluated during ongoing data cleaning meetings prior to unblinding of the data.

The Pharmacokinetics Per-Protocol Set (PK-PPS) consists of all randomized subjects who received at least 1 dose of the IMP and provided at least 1 quantifiable plasma concentration postdose without important protocol deviations that would affect the concentration.

#### 14.2 General statistical considerations

Summary statistics will consist of frequency tables for categorical variables. For continuous variables, summary statistics will consist of the number of available observations, arithmetic mean, SD, median, minimum, and maximum unless stated otherwise.

The statistical analysis of the co-primary efficacy variables and selected secondary efficacy variables will account for multiplicity and control the familywise Type I error rate at a 2-sided alpha level of 0.05 by using a fixed sequence testing procedure.

The hypotheses (H<sub>1</sub>, H<sub>2</sub>, H<sub>3</sub>, H<sub>4</sub>, H<sub>5</sub>, H<sub>6</sub>, H<sub>7</sub>, H<sub>8</sub>, H<sub>9</sub>, H<sub>10</sub>, H<sub>11</sub> and H<sub>12</sub>) comparing bimekizumab vs. adalimumab will be tested at a 2-sided alpha level of 0.05.

The first 2 hypotheses (H<sub>1</sub> and H<sub>2</sub>) will test whether bimekizumab is noninferior to adalimumab for the co-primary efficacy variables, PASI90 response at Week 16 and IGA response at Week 16. This evaluation of noninferiority will be tested at a 1-sided alpha level of 0.025 and will be based on a 1-sided 97.5% CI and a noninferiority margin of 10%. If noninferiority is achieved, the alpha will be passed to the next test in the sequence, allowing the testing procedure to proceed. The co-primary efficacy variables of PASI90 response at Week 16 and IGA response at Week 16 will then be evaluated for superiority relative to adalimumab at a 2-sided alpha level of 0.05, and testing will proceed only if superiority is achieved for both endpoints.

The hypotheses associated with the subsequent secondary efficacy endpoints are based on testing for superiority relative to adalimumab. See Figure 14-1 for details on this procedure.

Figure 14-1: Sequence of testing



Note: Calculations for H<sub>1</sub>-H<sub>9</sub> are based on the combined Bimekizumab arms with the sample size of 300. \* in H<sub>10</sub>-H<sub>12</sub> indicated calculations are based on the Bimekizumab Q4W/Q4W arm only with sample size of 150.

BKZ=bimekizumab; H=hypothesis; IGA=Investigator's Global Assessment; PASI=Psoriasis Area Severity Index; Q4W=every 4 weeks

### 14.3.1 Analysis of the primary efficacy variable

The co-primary efficacy variables for this study will be PASI90 response and IGA response at Week 16, and the corresponding analyses will be based on the RS. A subject will be classified as a PASI90 responder if the PASI score at Week 16 has improved at least 90% from Baseline, and an IGA responder will be any subject with a score of 0 or 1 (Clear or Almost Clear) with at least a 2-category improvement from Baseline in the IGA score. The primary analysis will be based on a stratified Cochran-Mantel-Haenszel (CMH) test where region and prior biologic exposure (yes/no) will be used as stratification variables. For the assessment of noninferiority, a noninferiority margin of 10% will be used and evaluated based on the confidence interval for the stratified Cochran Mantel-Haenszel risk difference between bimekizumab and adalimumab. A non-inferiority margin of 10% has been selected as this is considered to be a clinically relevant difference that could influence the choice of interventions used to treat chronic plaque PSO. Therefore, a difference within the 10% non-inferiority margin would suggest a similar impact on efficacy between the treatments. The evaluation of superiority will use pairwise treatment comparisons based on the CMH test using the p-value for the general association.

Nonresponder imputation (NRI) will be used to account for missing data in the primary analysis. Specifically, any subject who withdraws from study treatment prior to Week 16 or who has missing data for the primary efficacy variable at the Week 16 time point will be considered a nonresponder. Based on previous studies of biologics in subjects with moderate to severe chronic plaque PSO, it is expected that the number of subjects who discontinue prior to Week 16 will be low. For the small percentage of subjects for whom primary endpoint data are unavailable at Week 16, this lack of data is suggestive of an ineffective study treatment, thereby supporting the imputation of nonresponse. Therefore, NRI is considered an appropriate method for handling missing data since achieving the clinical response and making it through 16 weeks of study treatment are both critical components of the primary outcome.

# 14.3.1.1 Sensitivity analyses

The primary efficacy analysis described in Section 14.3 will be repeated based on the FAS and the PPS.

As a sensitivity analysis to the primary analysis method, logistic regression based on the RS will be used. The odds ratio of the responder rates at Week 16 will be estimated and tested between treatment groups using a logistic regression model with factors of treatment group, region, and prior biologic exposure (yes/no). The odds ratio, associated CI, and p-value based on the Wald test will be presented. If the logistic regression model is unable to converge, then prior biologic exposure may be dropped from the model to facilitate convergence. If the model is still unable to converge, then region may be removed from the model as well. As with the primary analysis, missing data will be handled using NRI.

The center-by-treatment interaction will be tested by replacing region with center in the logistic regression model described above and adding a center-by-treatment interaction term. In the model, center will be based on the original centers prior to pooling. However, if the model is unable to converge due to a low number of subjects at a given center, a pooling algorithm will be applied in order to allow the model to converge.


In order to obtain reasonable estimates of variability at a given center, a minimum of 15 subjects will be considered acceptable for a center to be included in the model without pooling. Given the 1:1:1 randomization allocation scheme, this should provide a minimum of about 5 subjects in the Centers with fewer than 15 subjects will be ordered from largest to smallest with pooling proceeding in the following manner:

Two or more centers will be combined until the cumulative and the fashion for the combined of the combined until the cumulative and the fashion for the combined until the cumulative and the combined until the bimekizumab Q4W arm, 5 subjects in the bimekizumab Q4W/Q8W arm, and 5 subjects in the adalimumab arm. Centers with fewer than 15 subjects will be eligible for pooling.

The following center pooling algorithm will be used for each geographic region:

- - each time at least 15 subjects has been reached in the previous pool.
  - If this iterative process reaches the end of the ordered list of centers where the final pooled center has fewer than 15 subjects, then the subjects from the centers in that pool will be combined with the pooled center formed in the previous iteration.

This procedure is only to be performed within a geographic region – there will be no pooling of centers across regions.

If the center-by-treatment interaction is not found to be significant ( $\alpha$ =0.10), then no further analyses will be performed. On the other hand, if the interaction is significant, further analyses will be conducted to determine which center or centers may be the source of the interaction. This will be done by running the logistic regression model (including the interaction term) where each center will be systematically removed from the model. The impact of a given center will be based on the change in the interaction p-value when that center is removed. The center or centers that appear to be driving the significant interaction effect will then be removed from the model to verify that conclusions remain the same with or without the influential center(s).

Additional sensitivity analyses to evaluate varying assumptions related to the handling of missing data will also be performed and are described in greater detail in Section 14.7.

### Other efficacy analyses 14.3.2

### Analysis of the secondary efficacy variables 14.3.2.1

### 14.3.2.1.1

The secondary efficacy variables for time points during the Initial Treatment Period will be analyzed for all subjects in the RS.

For comparisons with adalimumab at Week 16, the 2 bimekizumab arms will be pooled.

For binary secondary efficacy variables, the stratified CMH test as specified for the primary analysis will be implemented to test for superiority of bimekizumab to adalimumab. As in the primary analysis, NRI will be used to account for missing data.

Sensitivity analyses for the handling of missing data will be performed for the secondary efficacy variables that are part of the fixed sequence testing procedures. These analyses are described in Section 14.7.

#### 14.3.2.1.2 **Maintenance Treatment Period**

The secondary efficacy variables in the Maintenance Treatment Period include PASI90, PASI100, and IGA at Week 24 and Week 56.

In order to differentiate between subjects remaining on Q4W dosing from those switching to O8W dosing at Week 16, the treatment comparisons at Week 24 for PASI100, PASI90 and IGA will be performed in 2 different ways using the following randomized treatment arms:

- 1. Bimekizumab Q4W and bimekizumab Q4W/Q8W combined vs adalimumab (testing H<sub>7</sub>, H<sub>8</sub>, and H<sub>9</sub>)
- 2. Bimekizumab Q4W only vs adalimumab (testing  $H_{10}$ ,  $H_{11}$ , and  $H_{12}$ )

Since all subjects on adalimumab will be switched to bimekizumab at Week 24, the assessment of PASI90 and IGA at Week 56 will be for bimekizumab at the Q4W and Q8W dosing intervals. These summaries will include descriptive statistics by bimekizumab dose regimens at Week 24 and Week 56 based on the RS. Subjects with missing data at Week 56 or who discontinue study treatment prior to Week 56 will be imputed via NRI.

### Analysis of the other efficacy variables 14.3.2.2

The other efficacy variables will be analyzed for all subjects in the RS.

Binary (responder) variables will be summarized using frequency tables by treatment group for each visit.

Continuous variables will be summarized using descriptive statistics by treatment group for each visit.

Time to PASI50/75/90/100 response during the Initial Treatment Period will be estimated and presented using the Kaplan-Meier product-limit method for each treatment. Time to a given response will be defined as the length in days from the first dose of IMP until the first date when the response is achieved. Subjects who discontinue IMP prior to achieving a response will be censored at the date of IMP discontinuation. Subjects who reach the Week 24 Visit without achieving the given PASI response will be censored at the date of the Week 24 Visit. The median time to response, including the 2-sided 95% CI, will be calculated for each treatment. Between group differences will be analyzed with the log-rank statistic.

All other efficacy variables will be summarized based on imputed data (NRI and multiple imputation for binary and continuous variables, respectively, unless otherwise specified in the SAP) In some cases, variables may also be summarized based on observed case data (ie, subjects with missing data or who have prematurely discontinued IMP are treated as missing). There may be cases where the multiple imputation model fails to converge. In such situations, the last observation carried forward (LOCF) approach will instead be used to impute the missing data. If LOCF is used instead of multiple imputation for this reason, this will be clearly specified in the corresponding table summary. Should there be no missing data for a study variable, then only observed case data will be presented. Note that for LOCF imputation, any missing data or

data collected following discontinuation of IMP will be imputed with the most recent previous value. See Section 14.7 for further details.

age, gender, disease duration, region, weight, body mass systemic therapy of any kind, Baseline disease severity, and antibody positivity. These summaries will be based on imputed data (NRI) and will include descriptive statistics only 14.5 Planned safety and other analyses

Safety variables will be analyzed for 11 safety during the Months.

RS.

Adverse events will be coded according to the Medical Dictionary for Regulatory Activities (MedDRA®). Adverse events will be summarized descriptively by treatment group, primary system organ class, High Level Term (HLT), and preferred term. Additional tables will summarize AEs by intensity and relationship to IMP, AEs leading to withdrawal from the study, SAEs, and deaths. Specific safety topics of interest will be summarized and will be described in greater detail in the SAP.

For subjects who switch treatment, AEs will be allocated to the treatment the subject was on the day the event occurred. If the event occurs on the day of the switch, it will be attributed to the initial treatment, unless the event has a HLT of "Injection Site Reactions", in which case it will be attributed to the new treatment. Because the safety of switching from adalimumab to bimekizumab treatment is of particular interest, additional summaries to evaluate this will be specified in the SAP.

Laboratory values (including markedly abnormal labs), urinary values, vital signs, and extent of exposure will be presented descriptively by treatment group. Definitions for markedly abnormal laboratory values will be provided in the SAP.

### 14.5.2 Pharmacokinetic analyses

Pharmacokinetic variables will be analyzed for all subjects in the PK-PPS. Bimekizumab plasma concentrations will be summarized for each treatment at each scheduled visit.

### Immunogenicity analyses 14.5.3

will be used. Anti-bimekizumab antibodies (including positivity) summarized by treatment at each scheduled visit at which samples are collected.

14.6 Handling of protocol deviations

Important protocol 1 Anti-bimekizumab antibodies will be assessed using a tiered approach: screening, confirmatory, and titer assays will be used. Anti-bimekizumab antibodies (including positivity) will be

Important protocol deviations are deviations from the protocol which potentially could have a meaningful impact on study conduct, or on the primary efficacy, key safety, or PK outcomes for an individual subject. The criteria for identifying important protocol deviations will be defined

within the appropriate protocol-specific document at study start. Important protocol deviations will be reviewed as part of the ongoing data cleaning process and all important deviations will be identified and documented prior to unblinding to confirm exclusion from analysis sets.

as nonrespond.

as nonresponders for the primary analysis. The following sensitivity analyses for the co-primary efficacy variables will be performed:

- 1. Missing data will be addressed by using multiple imputation (Markov-Chain Monte Carlo [MCMC] method for intermittent missing data, followed by monotone regression for monotone missing data) to evaluate the effect of the method for handling missing data on the analysis. The actual PASI/IGA scores will be imputed and then dichotomized to obtain the response status. The treatment differences for each imputed data set will subsequently be evaluated using the stratified CMH test as used in the primary analysis. The results from each of the imputed data sets will be combined for overall inference using Rubin's rules, which account for the uncertainty associated with the imputed values (Rubin, 1987). This will be done using SAS PROC MIANALYZE. This procedure assumes a missing at random (MAR) pattern of missingness and corresponds to an estimand of the difference in outcome improvement if all subjects tolerated or adhered to treatment (Mallinckrodt et al, 2012). This is an estimand of efficacy to evaluate the de jure hypothesis.
- 2. Deviations from the MAR pattern assumed above will be evaluated. A sensitivity analysis will be performed in which, as with the above analysis, intermittent missing data will be imputed using multiple imputation (MI) based on the MCMC method. However, the remaining monotone missing data will be assumed to follow a missing not at random pattern. These data will be imputed using reference-based imputation. Typically, reference-based imputation uses an imputation model based on data from the placebo group, thereby assuming that monotone missing data follow a trajectory similar to the placebo group (Mallinckrodt et al, 2012). Since there is no placebo group in this study, and because it is assumed that bimekizumab is more efficacious than adalimumab, the adalimumab arm will be used as the reference arm. As specified in the previous procedure, actual PASI/IGA scores will be imputed and then dichotomized to get the response status. The treatment differences for each imputed data set will subsequently be evaluated using the stratified CMH test as used in the primary analysis. The estimand in this procedure is the difference in outcome improvement in all randomized subjects at the planned endpoint of the study attributable to the initially randomized medication (Mallinckrodt et al, 2012). This is an estimand of effectiveness to evaluate the de facto hypothesis.
- 3. A final sensitivity analysis will be based on observed data at Week 16. Subjects with missing data or who have prematurely discontinued study treatment will be treated as missing. The same CMH test as in the primary efficacy analysis will be used.

**UCB** 

Further details on the MI procedures will be provided in the SAP.

Missing data for binary secondary variables during the Initial Treatment Period will be imputed

For other continuous efficacy variables, MI will be used to impute missing data when possible. If the imputation model cannot converge, LOCF will be used. The MI procedure will be similarly sensitivity analysis #1 described above with the following differences: 10.11 will use the change from Baseline (instead of act. 12.12) be necessary; 2) instead = 6. and simple means and standard errors will be calculated using Rubin's rules (via SAS PROC MIANALYZE). For calculation of other descriptive statistics such as the median, min and max, Rubin's rules do not apply. Multiple imputation estimates will be computed by simply averaging the estimates from the multiple repetitions of the imputation algorithm.

### 14.8 Planned interim analysis and data monitoring

After the final Week 56 visit, an interim analysis will be performed and a corresponding interim CSR may be written. A final analysis and updated final CSR will be prepared once all data (through the SFU visit) have been collected.

### Determination of sample size 14.9

A total of 450 subjects will be randomly assigned in a 1:1:1 ratio to the following treatment groups:

- Bimekizumab 320mg Q4W throughout the study (150 subjects)
- Bimekizumab 320mg Q4W/Q8W (ie, bimekizumab 320mg Q4W until Week 16, then bimekizumab 320mg Q8W from Week 16 through Week 52 (150 subjects)
- Adalimumab 80mg administered as an initial dose, followed by 40mg Q2W starting 1 week after the initial dose (ie. adalimumab will be administered according to the labeling recommendations) until Week 24, then bimekizumab 320mg Q4W from Week 24 to Week 52 (150 subjects)

When comparing bimekizumab to adalimumab, the assumed responder rates for PASI90 and IGA at Week 16 for the bimekizumab group are 75% and 85%, respectively. These estimates are based on the results of the Phase 2b PS0010 study. The PASI90 responder rates at Week 16 for adalimumab from the VOYAGE-1 and VOYAGE-2 studies were 50% and 47%, respectively (Blauvelt et al, 2017; Reich et al, 2017). Additionally, the IGA responder rates at Week 16 for adalimumab in VOYAGE-1 and VOYAGE-2 were 66% and 68%, respectively. For the purposes of these sample size calculations at Week 16, we assume a PASI90 responder rate and IGA responder rate for adalimumab of 50% and 68%, respectively.

The testing procedure described in Section 14.3 indicates that the first test will be to demonstrate noninferiority to adalimumab for the co-primary variables of PASI90 and IGA at Week 16. If non-inferiority for both tests is demonstrated, then superiority to adalimumab will be tested.

Because the superiority evaluation is the more stringent test, sample size calculations are based on the testing of superiority to adalimumab for PASI90 and IGA at Week 16. Given these assumptions and a sample size of 150 subjects in the adalimumab arm and 300 subjects in the Note that the non-inferiority testing procedure will be based on a 1-sided significance level of 0.025 and a non-inferiority margin of 10%. The power to demonstrate non-inferiority to adalimumab using the other assumptions described above is >99% for both procedure.

ETHICS AND BECAUSE PASI and IGA response tend to be highly correlated, the same power for achieving superiority on both co-primary endpoints is not calculated here.

Note that the non-inferiority testing procedure will be based on a 1-sided significance level of 0.025 and a non-inferiority margin of 10%. The power to demonstrate non-inferiority to adalimumab using the other assumptions described above is >99% for both procedure.

# ETHICS AND REGULATORY REQUIREMENTS

#### 15.1 Informed consent

Subject's informed consent must be obtained and documented in accordance with local regulations, ICH-GCP requirements, and the ethical principles that have their origin in the principles of the Declaration of Helsinki.

Prior to obtaining informed consent, information should be given in a language and at a level of complexity understandable to the subject in both oral and written form by the Investigator (or designee). Each subject will have the opportunity to discuss the study and its alternatives with the Investigator.

Prior to participation in the study, the ICF should be signed and personally dated by the subject and by the person who conducted the informed consent discussion (Investigator or designee). The subject must receive a copy of the signed and dated ICF. As part of the consent process, each subject must consent to direct access to his/her medical records for study-related monitoring, auditing, IRB/IEC review, and regulatory inspection.

If the ICF is amended during the study, the Investigator (or the Sponsor, if applicable) must follow all applicable regulatory requirements pertaining to the approval of the amended ICF by the IRB/IEC and use of the amended form.

All studies conducted at centers in the United States must include the use of a Health Insurance Portability and Accountability Act Authorization Form.

The subject may withdraw his/her consent to participate in the study at any time. A subject is considered as enrolled in the study when he/she has signed the ICF. An eCRF must not be started, nor may any study-specific procedure be performed for a given subject, without having obtained his/her written consent to participate in the study.

### 15.2 Subject identification cards

Upon signing the Informed Consent and Assent Form (as applicable), the subject will be provided with a subject identification card in the language of the subject. The Investigator will fill in the subject identifying information and medical emergency contact information. The Investigator will instruct the subject to keep the card with him/her at all times.

### 15.3 **Institutional Review Boards and Independent Ethics Committees**

Ine Investigator/UCB will ensure that an appropriately constituted IRB/IEC that complies with the requirements of the current ICH-GCP version or applicable country-specific regulations will be responsible for the initial and continuing review and approval of the clinical study. Prior to initiation of the study, the Investigator/UCB will forward copies of the Investigator's curriculum vitae (if applicable) subject-related documents. subject-related documents to be used for the study to the IRB/IEC for its review and approval.

Before initiating a study, the Investigator will have written and dated full approval from the responsible IRB/IEC for the protocol.

The Investigator will also promptly report to the IRB/IEC all changes in the study, all unanticipated problems involving risks to human subjects or others, and any protocol deviations, to eliminate immediate hazards to subjects.

The Investigator will not make any changes in the study or study conduct without IRB/IEC approval, except where necessary to eliminate apparent immediate hazards to the subjects. For minor changes to a previously approved protocol during the period covered by the original approval, it may be possible for the Investigator to obtain an expedited review by the IRB/IEC as allowed.

As part of the IRB/IEC requirements for continuing review of approved studies, the Investigator will be responsible for submitting periodic progress reports to the IRB/IEC (based on IRB/IEC requirements), at intervals appropriate to the degree of subject risk involved, but no less than once per year. The Investigator should provide a final report to the IRB/IEC following study completion.

UCB (or its representative) will communicate safety information to the appropriate regulatory authorities and all active Investigators in accordance with applicable regulatory requirements. The appropriate IRB/IEC will also be informed by the Investigator or the Sponsor, as specified by the applicable regulatory requirements in each concerned country. Where applicable, Investigators are to provide the Sponsor (or its representative) with evidence of such IRB/IEC notification.

### Subject privacy 15.4

UCB staff (or designee) will affirm and uphold the subject's confidentiality. Throughout this study, all data forwarded to UCB (or designee) will be identified only by the subject number assigned at Screening.

The Investigator agrees that representatives of UCB, its designee, representatives of the relevant IRB/IEC, or representatives of regulatory authorities will be allowed to review that portion of the subject's primary medical records that directly concerns this study (including, but not limited to, laboratory test result reports, ECG reports, admission/discharge summaries for hospital

admissions occurring during a subject's study participation, and autopsy reports for deaths occurring during the study).

Significant changes to the protocol will only be made as an amendment to the protocol and must be approved by UCB, the IRB/IEC, and the regulatory authorities (if required), prior to being implemented.

16 FINANCE, INSUPARIO

Insurance coverage will be handled according to local requirements.

Finance, insurance, and publication rights are addressed in the Investigator and/or CRO agreements, as applicable.

#### 17 REFERENCES

Augustin M, Glaeske G, Radtke MA, Christophers E, Reich K, Schäfer I. Epidemiology and comorbidity of psoriasis in children. Br J Dermatol. 2010:162:633-6.

Blauvelt A, Tyring SK, Papp KA, Griffiths CEM, et al. Efficacy and safety of guselkumab, an anti-interleukin-23 monoclonal antibody, compared with adalimumab for the continuous treatment of patients with moderate to severe psoriasis: Results from the phase III, doubleblinded, placebo- and active comparator-controlled VOYAGE 1 trial. J Am Acad Dermatol 2017; 76:405-17.

Christophers E, Barker JN, Griffiths CE, Daudén E, Milligan G, Molta C, et al. The risk of psoriatic arthritis remains constant following initial diagnosis of psoriasis among patients seen in European dermatology clinics. J Eur Acad Dermatol Venereol. 2010;24:548-54.

Common Terminology Criteria for Adverse Events (CTCAE), Version 4.0. National Institutes of Health, National Cancer Institute, Division of Cancer Treatment and Diagnosis. http://ctep.cancer.gov/protocolDevelopment/electronic applications/ctc.htm. Updated 03 Mar 2016.

CPMP/ICH/135/95 Note for guidance on Good Clinical Practice (EMEA) Jul 2002.

Dowlatshahi EA, Wakkee M, Arends LR, Nijsten T. The prevalence and odds of depressive symptoms and clinical depression in psoriasis patients: a systematic review and meta-analysis. J Invest Dermatol. 2014;134:1542-51.

Feldman SR. A quantitative definition of severe psoriasis for use in clinical trials. J Dermatolog

Food and Drug Administration. Guidance for Industry. Drug-induced liver injury: premarketing clinical evaluation. US Dept of Health and Human Services. Contact Contac Research, Center for Biologics Evaluation and Research, 07/2009.

Gelfand JM, Neimann AL, Shin DB, Wang X, Margolis DJ, Troxel AB. Risk of myocardial infarction in patients with psoriasis. JAMA. 2006;296:1735-41.

Gisondi P, Tessari G, Conti A, Piaserico S, Schianchi S, Peserico A, et al. Prevalence of metabolic syndrome in patients with psoriasis: a hospital-based case-control study. Br J Dermatol. 2007;157:68-73.

Gottlieb AB. Psoriasis: Emerging therapeutic strategies. Nat Rev Drug Discov. 2005;4:19-34.

Husni ME, Qureshi AA, Keonig AS, Pedersen R, Robertson D. Utility of the PASE questionnaire, psoriatic arthritis (PsA) prevalenece and PsA improvement with anti-TNF therapy: results from the PRISTINE trial. J Dermatolog Treat. 2014;25(1):90-5.

Icen M, Crowson CS, McEvoy MT, Dann FJ, Gabriel SE, Maradit Kremers H. Trends in incidence of adult-onset psoriasis over three decades: a population-based study. J Am Acad Dermatol. 2009;60:394-401.

Kimball AB, Yu AP, Signorovitch J, Xie, J, Tsaneva M, Gupta SR, et al. The effects of adalimumab treatment and psoriasis severity on self-reported work productivity and activity impairment for patients with moderate to severe psoriasis. J Am Acad Dermatol. 2012;66(2):e67-e75.

Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001;16:606–13.

Krueger G, Ellis CN. Psoriasis—recent advances in understanding its pathogenesis and treatment. J Am Acad Dermatol. 2005;53(1 Suppl 1):S94-100.

Krueger G, Koo J, Lebwohl M, Menter A, Stern RS, Rolstad T. The impact of psoriasis on quality of Life. Results of a 1998 National Psoriasis Foundation patient-membership survey. Arch Dermatol. 2001;137:280-4.

Kurd SK, Smith N, VanVoorhees A, Troxel AB, Badmaev V, Seykora JT, et al. Oral curcumin in the treatment of moderate to severe psoriasis vulgaris: a prospective clinical trial. J Am Acad Dermatol. 2008;58:625-31.

Kurd SK, Gelfand JM. The prevalence of previously diagnosed and undiagnosed psoriasis in US adults: results from NHANES 2003-2004. J Am Acad Dermatol. 2009;60:218-24.

Langley RG, Krueger GG, Griffiths CEM. Psoriasis: epidemiology, clinical features, and quality of life. Ann Rheum Dis. 2005;64(Suppl II):ii18–ii23.

Mallinckrodt CH, Lin Q, Lipkovich I, Molenberghs G. A structured approach to choosing estimands and estimators in longitudinal clinical trials. Pharm Stat. 2012;11:456-61.

Maruish, M. E. (Ed.). User's manual for the SF-36v2 Health Survey (3rd ed.). Lincoln, RI: QualityMetric Incorporated. 2011.

Mukhtar R, Choi J, Koo JY. Quality of life issues in psoriasis. Dermatol Clin. 2004;22:389-95.

Mundt JC, Greist JH, Gelenberg AJ, Katzelnick DJ, Jefferson JW, Modell JG. Feasibility and Validation of a Computer-Automated Columbia-Suicide severity Rating Scale Using Interactive Voice Response Technology. J Psychiatr Res. 2010;44(16):1224-8.

Ortonne JP. Redefining clinical response in psoriasis: targeting the pathological basis of disease. J Drugs Dermatol. 2004;3:13-20.
Parisi R, Symmons DP, Griffiths CE, Ashcroft DM, Identification and Management of Psoriasis and Associated ComorbidiTy (IMPACT) project team. Global epidemiology of psoriasis: A systematic review of incidence and prevalence. J Invest Dermatol. 2013;133:377-385.

Rachakonda TD, Schupp CW, Armstrong AW. Psoriasis prevalence among adults in the United States. J Am Acad Dermatol. 2014;70:512-6.

Raychaudhuri SP, Gross J. A comparative study of pediatric psoriasis. Pediatric Dermatology. 202

Reich K, Armstrong AW, Foley P, et al. Efficacy and safety of guselkumab, an anti-interleukin-23 monoclonal antibody, compared with adalimumab for the treatment of patients with moderate to severe psoriasis with randomized withdrawal and retreatment: Results from the phase III. double-blind, placebo- and active comparator-controlled VOYAGE 2 trial PAm Acad Dermatol 2017; 76:418-31.

Reilly MC, Zbronzek AS, Dukes EM. The Validity and Reproducibility of a Work Productivity and Activity Impairment Instrument. PharmacoEconomics. 1993 4(5):353-365.

Rubin D.B. 1987. Multiple Imputation for Nonresponse in Surveys. New York: John Wiley and Sons.

Valizadeh A, Khosravi A, Zadeh LJ, Parizad EG, Role of IL-25 in Immunity. J Clin Diagn Res. 2015;9(4):OE01-OE04.

Vender R, Lynde C, Ho V, Chau D, Poulin-Costello M. Work Productivity and Healthcare Resource Utilization Outcomes for Patients on Etanercept for Moderate-to-Severe Plaque Psoriasis: Results from a 1-Year, Multicentre, Open-Lable, Single-Arm Study in a Clinical Setting. Appl Health Econ Health Policy. 2012:10(5):343-53.

Yeung H, Takeshita J, Mehta NN, Kimmel SE, Ogdie A, Margolis DJ, et al. Psoriasis severity Ajo.

Ajo.

This document cannot be used to supply the supply of the sup and the prevalence of major medical comorbidity: a population-based study. JAMA Dermatol.

## 18 APPENDICES

#### 18.1 Protocol Amendment 1

#### Rationale for the amendment

The purpose of this amendment was the following:

- Remove re-randomization at Week 24. Subjects in the bimekizumab groups will be allocated to bimekizumab 320mg Q4W throughout the study or bimekizumab 320mg Q4W through Week 16 and bimekizumab 320mg Q8W thereafter
- Remove change in dose based on PASI90 response
- Update the study design so subjects in the bimekizumab Q4W/Q8W arm switch at Week 16 instead of Week 24
- Add a new other efficacy variable (absolute and percent change from Baseline in the product of IGA and BSA [IGAxBSA])
- Add assessment of the Patient Symptom Diary (daily) to the Screening and Week 16 Visits
- Clarify the dosing window
- Add percentage of BSA as an assessments at all visits
- Clarify that PGADA will be performed on all subjects at Baseline
- Remove the criterion that excluded subjects exposed to more than 3 biologic response modifiers (including no more than 1 IL-17)
- Clarify that subjects who experienced primary failure (no response within 12 weeks) to 1 or more IL-17 biologic response modifiers or more than 1 biologic response modifiers other than an IL-17 should be excluded from the study
- Remove the withdrawal criterion that subjects who do not achieve a PASI50 response by Week 28 or later be withdrawn from the study
- Corrected discrepancies between Section 8 Study procedures by visit and Table 5-1 Schedule of study assessments
- Clarify that the same assessor should evaluate the subject at each efficacy assessment
- Clarify in footnote c of Table 12-2 Laboratory measurements the visits in which the urine drug screen will be performed
- Update the assessment and management of TB and TB risk factors
- Update the sequence testing and analysis of secondary efficacy variables

In addition, minor spelling, editorial, and formatting changes were made, and the List of abbreviations was updated.

#### **Modifications and changes**

**Specific changes** 

Change #1

Title page

A PHASE 3, MULTICENTER, RANDOMIZED, DOUBLE-BLIND STUDY WITH A 24-WEEK ACTIVE-CONTROLLED INITIAL TREATMENT PERIOD FOLLOWED BY A 32-4 WEEK, DOSE-BLIND MAINTENANCE TREATMENT PERIOD TO EVALUATE THE EFFICACY AND SAFETY OF BIMEKIZUMAB IN ADULT SUBJECTS WITH MODERATE TO SEVERE CHRONIC PLAQUE PSORIASIS

## Has been changed to:

A PHASE 3, MULTICENTER, RANDOMIZED, DOUBLE-BLIND STUDY WITH AN-24-**WEEK** ACTIVE-CONTROLLED INITIAL TREATMENT PERIOD FOLLOWED BY A 32 WEEK, DOSE-BLIND MAINTENANCE TREATMENT PERIODITO EVALUATE THE EFFICACY AND SAFETY OF BIMEKIZUMAB IN ADULT SUBJECTS WITH MODERATE TO SEVERE CHRONIC PLAQUE PSORIASIS

# Change #2

# **Section 1 Summary**

Approximately 540 subjects will be screened in order to have a total of 400 subjects randomized in the study. For each subject, the study will last a maximum of 76 weeks and will consist of 4 periods, a Screening Period (2 to 4 weeks), a double-blind, active comparator-controlled Initial Treatment Period (24 weeks), a dose-blind Maintenance Treatment Period (32 weeks), and a Safety Follow-Up (SFU) Period (20 weeks after the last dose of the investigational medicinal product [IMP]). After completion of the 32-week Maintenance Treatment Period, eligible subjects will be allowed to enroll in an open-label study.

During the Treatment Period, eligible subjects will be randomized 1:1 to receive the following blinded IMP regimens subcutaneously (sc):

Double-blind Initial Treatment Period:

- Bimekizumab 320mg administered Q4W (200 subjects)
- Adalimumab 80mg administered as an initial dose, followed by 40mg every 2 weeks (Q2W) starting P week after the initial dose (ie, adalimumab will be administered according to the labeling recommendations) (200 subjects)

• Subjects in the bimekizumab 320mg OAW response at Week 24 Subjects in the bimekizumab 320mg Q4W treatment arm who do not achieve a PASI90 response at Week 24 will continue to receive bimekizumab 320mg Q4W.

- Subjects in the bimekizumab 320mg Q4W treatment arm who achieve a PASI90 response at Week 24 will be re-randomized 1:1 to receive bimekizumab 320mg Q4W or bimekizumab 320mg Q8W.

Subjects who do not have a PASI50 response at Week 36 or later will be withdrawn from the study.

At Week 56, all subjects enrolling in the open-label study will under assessments before receiving their first open-label study will in the open-label SFU Period.

## Has been changed to:

Approximately 600540 subjects will be screened in order to have a total of 450400 subjects randomized in the study. For each subject, the study will last a maximum of 76 weeks and will consist of 4 periods, a Screening Period (2 to 4 weeks), a double-blind, active comparatorcontrolled Initial Treatment Period (1624 weeks), a dose-blind Maintenance Treatment Period (4032-weeks), and a Safety Follow-Up (SFU) Period (20 weeks after the last dose of the investigational medicinal product [IMP]). After completion of the 4032-week Maintenance Treatment Period, eligible subjects will be allowed to enroll in an open-label study.

During the Treatment Period, eEligible subjects will be randomized 1:1:1 to receive the following blinded IMP regimens subcutaneously (sc):

#### **Double blind Initial Treatment Period**?

- Bimekizumab 320mg Q4W administered Q4Wthroughout the study (150200 subjects)
- Bimekizumab 320mg Q4W/Q8W (ie, bimekizumab 320mg will be administered through Week 12, then bimekizumab 320mg Q8W from Week 16 through Week 52 (150 subjects)
- Adalimumab 80mg administered as an initial dose, followed by 40mg every 2 weeks (O2W) starting 1 week after the initial dose (ie, adalimumab will be administered according to the labeling recommendations) until Week 24, then bimekizumab Q4W from Week 24 to Week 52 (150200 subjects)

#### **Dose blind Maintenance Treatment Period:**

From Week 24 onwards, subjects will be treated as follows:

Subjects in the bimekizumab 320mg Q4W treatment arm who do not achieve a PASI90 response at Week 24 will continue to receive bimekizumab 320mg Q4W.

- Subjects in the bimekizumab 320mg Q4W treatment arm who achieve a PASI90
  response at Week 24 will be re-randomized 1:1 to receive bimekizumab 320mg Q4W or
  bimekizumab 320mg Q8W.
- Subjects in the adalimumab treatment arm will receive bimekizumab 320mg Q4W.

Bimekizumab will be administered in the clinic at Baseline and Q4W or Q8W thereafter, through Week 52. An initial dose of the active comparator, adalimumab 80mg, will be administered at Baseline followed by adalimumab 40mg Q2W from Week 1 through Week 23.

Subjects who do not have a PASI50 response at Week 36 or later will be withdrawn from the study.

#### Change #3

#### Section 2.1.2 Current treatments for psoriasis

Brodalumab has been approved in the US for the treatment of moderate to severe plaque psoriasis in adult patients who are candidates for systemic therapy or phototherapy and have failed to respond or have lost response to other systemic therapies. Brodalumab is a human monoclonal IgG2 antibody that selectively binds to human IL-17RA and inhibits its interactions with cytokines IL-17A, IL-17F, IL-17C, IL-17A/F heterodimer and IL-25. Blocking IL 17RA inhibits IL-17 cytokine-induced responses including the release of pro-inflammatory cytokines and chemokines. Brodalumab has a black box warning regarding suicidal ideation and behavior.

## Has been changed to:

Brodalumab has been approved in the US for the treatment of moderate to severe plaque psoriasis in adult patients who are candidates for systemic therapy or phototherapy and have failed to respond or have lost response to other systemic therapies. In the EU, brodalumab is indicated for the treatment of moderate to severe plaque PSO in adult patients who are candidates for systemic therapy. Brodalumab is a human monoclonal IgG2 antibody that selectively binds to human IL-17RA and inhibits its interactions with cytokines IL-17A, IL-17F, IL-17C, IL-17A/F heterodimer and IL-25. Blocking IL 17RA inhibits IL-17 cytokine-induced responses including the release of pro-inflammatory cytokines and chemokines. Brodalumab has a black box warning regarding spicidal ideation and behavior.

#### Change #4

# Section 2,2.1.1 Completed studies

Four clinical studies of bimekizumab have been completed: UP0008 in 39 subjects with mild to moderate plaque PSO, RA0124 in 30 healthy volunteers, PA0007 in 53 subjects with PsA, and UP0031 in 12 healthy volunteers. Three studies (RA0123, PS0010, and PS0016) are ongoing in subjects with moderate to severe rheumatoid arthritis (RA0123) and in subjects with moderate to severe PSO (PS0010 and PS0016).

Four clinical studies of bimekizumab have been completed: UP0008 in 39 subjects with mild to moderate plaque PSO, RA0124 in 30 healthy volunteers, PA0007 in 53 subjects with PsA, and UP0031 in 12 healthy volunteers. Three studies (RA0123, PS0010, and PS0016) are ongoing in subjects with moderate to severe rheumatoid arthritis (RA0123) and in subjects with moderate to severe PSO (PS0010 and PS0016).

#### Change #5

#### Section 2.2.1.2 Ongoing studies

Five additional studies of bimekizumab in the treatment of PSO are ongoing.

#### Has been changed to:

Four additional studies of bimekizumab in the treatment of PSO and 1 study in healthy volunteers are ongoing. Five additional studies of bimekizumab in the treatment of PSO are ongoing.

## Change #6

#### **Section 4.3.1 Other efficacy variables**

Change from Baseline variables evaluated during the Initial Treatment Period, are relative to the Baseline (first dose) Visit. For subjects who switch treatment at the Week 24 Visit, change from Baseline variables during the Maintenance Treatment Period may be evaluated relative to both the Baseline (first dose) Visit and the Week 24 Visit

## Has been changed to:

Change from Baseline variables evaluated during the Initial Treatment Period, are relative to the Baseline (first dose) Visit. In addition, Ffor subjects who started with adalimumab and switch treatment at the Week 24 Visit, change from Baseline variables during the Maintenance Treatment Period may be evaluated relative to both the Baseline (first dose) Visit and the Week 24 Visit.

#### Change #7

#### Section 4.3.1 Other efficacy variables

The following bullet has been added:

• Absolute and percent change from Baseline in the product of IGA and BSA (IGAxBSA)

#### Change #8

# Section 5.1 Study description

PS0008 is a Phase 3, multicenter study consisting of a 24-week, randomized, double-blind, parallel-group, active-comparator-controlled Initial Treatment Period followed by a 32-week, Maintenance Treatment Period to evaluate the efficacy and safety of bimekizumab in adult subjects with moderate to severe chronic plaque PSO. To be eligible to participate in this study, subjects must be adults with a diagnosis of moderate to severe PSO (Baseline PASI ≥12 and BSA affected by PSO ≥10% and IGA score ≥3 [on a 5-point scale]) who are candidates for systemic PSO therapy and/or phototherapy and/or photochemotherapy. Up to 30% of subjects

may have been previously exposed to a biologic therapy (see Exclusion Criteria #22 and #23, Section 6.2).

#### Has been changed to:

PS0008 is a Phase 3, multicenter study consisting of a **1624**-week, randomized, double-blind, parallel-group, active-comparator-controlled Initial Treatment Period followed by a **4032**-week, Maintenance Treatment Period to evaluate the efficacy and safety of bimekizumab in adult subjects with moderate to severe chronic plaque PSO. To be eligible to participate in this study, subjects must be adults with a diagnosis of moderate to severe PSO (Baseline PASI ≥12 and BSA affected by PSO ≥10% and IGA score ≥3 [on a 5-point scale]) who are candidates for systemic PSO therapy and/or phototherapy and/or photochemotherapy. **Adalimumab will be administered per the local label.** Up to 30% of subjects may have been previously exposed to a biologic therapy (see Exclusion Criterion #22-and #23, Section 6.2).

#### Change #9

#### **Section 5.2** Study periods

This study will include 4 periods, a Screening Period (2 to 4 weeks), an Initial Treatment Period (24 weeks), a Maintenance Treatment Period (32 weeks), and a SFU Period (20 weeks after the last dose of IMP). After completion of the Maintenance Treatment Period, eligible subjects will be allowed to enroll in an open-label study. Subjects enrolling into the open-label study will not have the PS0008 SFU Visit.

#### Has been changed to:

This study will include 4 periods, a Screening Period (2 to 4 weeks), an Initial Treatment Period (1624 weeks), a Maintenance Treatment Period (4032 weeks), and a SFU Period (20 weeks after the last dose of IMP). After completion of the Maintenance Treatment Period, eligible subjects will be allowed to enroll in an open-label study. Subjects enrolling into the open-label study will not have the PS0008 SFU Visit.

#### Change #10

# Section 5.2.2 Double-blind Initial Treatment Period

During the active-controlled 24-week Initial Treatment Period, approximately 400 subjects will be randomized 1:1 to receive the following blinded IMP regimens:

- Bimekizumab 320mg administered sc Q4W (200 subjects)
- Adalimumab 80mg administered as an initial dose, followed by 40mg every Q2W starting
  1 week after the initial dose (ie, adalimumab will be administered according to the labeling
  recommendations) (200 subjects)

During the active-controlled 1624-week Initial Treatment Period, approximately 450400 subjects will be randomized 1:1:1 to receive the following blinded IMP regimens:

- Bimekizumab 320mg administered se Q4W throughout the study (150200 subjects)
- Bimekizumab 320mg administered Q4W until Week 16 (150 subjects)
- Sions of variations thereof Adalimumab 80mg administered as an initial dose, followed by 40mg every Q2W starting 1 week after the initial dose (ie, adalimumab will be administered according to the labeling recommendations) until Week 24 (150200 subjects)

#### Change #11

#### **Section 5.2.3 Dose-blind Maintenance Treatment Period**

After the 24-week Initial Treatment Period, subjects will enter the 32-week Maintenance Treatment Period. Treatment during the Maintenance Treatment Period will start at Week 24 and subjects will return to the clinic O4W through Week 56. The IMP will be administered in the clinic by sc injection at the time points specified in the schedule of study assessments (Table 5-1). Treatment during the Maintenance Treatment Period will be based on initial treatment and response to treatment at Week 24, per the following rules:

- Subjects in the bimekizumab 320mg Q4W treatment arm who do not achieve a PASI90 response at Week 24 will continue to receive bimekizumab 320mg Q4W.
- Subjects in the bimekizumab 320mg Q4W treatment arm who achieve a PASI90 response at Week 24 will be re-randomized 1:1 to receive bimekizumab 320mg Q4W or bimekizumab 320mg Q8W.
- Subjects in the adalimumab treatment arm will receive bimekizumab 320mg Q4W.

Subjects may receive placebo injections at certain visits in order to blind the IMP (see Section 7.2).

If a subject does not achieve a PASI50 response at Week 36 or later, the subject will be withdrawn from the study at the time point when the PASI50 response is not achieved.

#### Has been changed to:

After the 1624-week Initial Treatment Period, subjects will enter the 4032-week Maintenance Treatment Period. Treatment during the Maintenance Treatment Period will start at Week 1624 and subjects will return to the clinic Q4W or Q8W through Week 56. The IMP will be administered in the clinic by sc injection at the time points specified in the schedule of study assessments (Table 5-1). Treatment during the Maintenance Treatment Period will be based on initial treatment and response to treatment at Week 24, per the following rules:

- Subjects in the bimekizumab 320mg Q4W treatment arm who do not achieve a PASI90
- Treatment Period 24, per the following ru 320mg Q4W treatment arm who do not achie response at Week 24 will continue to receive bimekizumab 320mg Q4W.

  Subjects in the bimekizumab 320mg Q4W treatment arm response at Week 24 will be re random bimekizumab 320mg. Subjects in the bimekizumab 320mg Q4W treatment arm who achieve a PASI90 response at Week 24 will be re randomized 1:1 to receive bimekizumab 320mg Q4W or bimekizumab 320mg Q8W. Subjects in the bimekizumab 320mg Q4W/Q8W treatment arm will receive bimekizumab Q8W from Week 16 through Week 52.

Subjects in the adalimumab treatment arm will bimekizumab 320mg Q4W from Week 24 to Week 52.

Subjects may receive placebo injections at certain visits in order to blind the IMP (see Section 7.2).

Jany extensions or variations thereof. If a subject does not achieve a PASI50 response at Week 36 or later, the subject will be withdrawn from the study at the time point when the PASI50 response is not achieved.

#### Change #12

#### Section 5.3 Study duration per subject

For each subject, the study will last a maximum of up to 76 weeks, as follows:

- Screening Period: 2 to 4 weeks
- Double-blind, active-controlled Initial Treatment Period: 24 weeks
- Maintenance Treatment Period: 32 weeks
- Safety Follow-Up Period: a SFU Visit is planned 20 weeks after the last dose of IMP (for subjects not enrolling in the open-label study)

After the 32-week Maintenance Treatment Period, subjects will be allowed to enroll in an openlabel study, in which case subjects will undergo the Week 56 study assessments before receiving their first open-label IMP dose. The SFU Visit will not be required for subjects who enroll in the open-label study.

# Has been changed to:

For each subject, the study will last a maximum of up to 76 weeks, as follows:

- Screening Period: 2 to 4 weeks
- Double-blind, active-controlled Initial Treatment Period: 1624 weeks
- Maintenance Treatment Period: 4032 weeks
- Safety Follow-Up Period a SFU Visit is planned 20 weeks after the last dose of IMP (for subjects not enrolling in the open-label study)

After the 4032-week Maintenance Treatment Period, subjects will be allowed to enroll in an open-label study, in which case subjects will undergo the Week 56 study assessments before receiving their first open-label IMP dose. The SFU Visit will not be required for subjects who enroll in the open-label study.

# Change #13

#### Section 5.4 Planned number of subjects and site(s)

Approximately 540 subjects will be screened in order to have 400 subjects randomized in the study. There will be approximately 200 subjects per treatment arm. The planned number of study sites is approximately 100. Every eligible subject who signs an ICF will be expected to be randomized.

The deciment dance to support any interest of the contract of


96 Apr 2018 PS0008

 Table 5-1:
 Schedule of study assessments

| Visit <sup>a</sup> /<br>Week | Screening | | | | | Doub | ole-blin<br>(wee | | al Trea<br>er first | | Period | | | | | Do | | .00. | intena<br>Period | d | | nent | W56PEO | SFUb |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Protocol activity | | Baseline (first dose) | 1 | 3 | 4 | 5, 7 | 8 | 9,<br>11 | 12 | 13,<br>15 | 16 | 17,<br>19 | 20 | 21,<br>23 | 242 | 28 | 32 | 36 | 40 | 44 | 48 | 52 | 56 | |
| Informed consent <sup>c</sup> | X | | | | | | | | | | | | | 101: | )· | | | | | | | X <sup>d</sup> | | |
| Inclusion/exclusion | X | X | | | | | | | | | | | | 0 | | | | | | | | | | |
| Urine drug screen | X | | | | | | | | | | | 7 | 166 | | | | | | | | | | X | |
| Demographic data | X | | | | | | | | | | 0 | .00 | O`` | | | | | | | | | | | |
| Psoriasis history | X | | | | | | | | | 1 | :1 | | | | | | | | | | | | | |
| Significant past<br>medical history and<br>concomitant<br>diseases | X | Xe | | | | | | < | 2EDR | | COLL | | | | | | | | | | | | | |
| Physical examination <sup>f,g</sup> | X | | | | | | | ~3 | X | | X | | | | X | | | X | | | X | | X | X |
| Height | | X | | | | | _ < | 4 | | | | | | | | | | | | | | | | |
| Body weight | | X | | | | | N.O | | | | X | | | | X | | | X | | | X | | X | |
| Vital signs <sup>h</sup> | X | X | X | X | X | XQ | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Hematology and biochemistry | X | X | X | X | XX | 5 | X | | X | | X | | X | | X | | X | | X | | X | | X | X |
| Urinalysis | X | X | | 1 | 5 | | | | | | X | | | | X | | X | | X | | X | | X | X |
| ECG | X | | . * | 100 | | | | | | | X | | | | X | | | X | | | X | | X | |
| Pregnancy testing <sup>i</sup> | X | X | MINO | | X | | X | | X | | X | | X | | X | X | X | X | X | X | X | X | X | X |

PS0008

Table 5-1: Schedule of study assessments

| Visit <sup>a</sup> /<br>Week | Screening | | | | | Doub | | | al Trea | tment l<br>dose) | Period | | | | | Dos | | nd Ma | intena<br>Period | i | | ent | W56PEO | SFUb |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Protocol activity | | Baseline<br>(first dose) | 1 | 3 | 4 | 5, 7 | 8 | 9,<br>11 | 12 | 13,<br>15 | 16 | 17,<br>19 | 20 | 21,<br>23 | 24 | 28 | 32 | 36 | 40 | 44 | 48 | 52 | 56 | |
| Hepatitis B and C testing <sup>j</sup> | X | | | | | | | | | | | | | dilon | | | | | | | | | | |
| HIV testing <sup>k</sup> | X | | | | | | | | | | | 7 | Oblie | | | | | | | | | | | |
| Chest x-ray <sup>l</sup> | X | | | | | | | | | | (ي | | ).< | | | | | | | | | | | |
| IGRA Tuberculosis test | X | | | | | | | | | | 177 | | | | | | | | | | | X | | |
| Tuberculosis questionnaire | X | X | | | | | | | 10° | ani | X | | | | X | | | X | | X | | X | X | X |
| Blood sample for<br>bimekizumab<br>plasma<br>concentrations <sup>m</sup> | | X | X | X | X | | X | .03 | X iii | 0 | X | | X | | X | | | X | | | X | | X | X |
| Blood sample for anti-bimekizumab antibodies <sup>m</sup> | | X | | | X | | X | A) | X | | X | | X | | X | | | X | | | X | | X | X |
| Blood sample<br>genomic,<br>proteomic, and<br>metabolomics, and<br>candidate<br>biomarker<br>analyses <sup>c,m</sup> | | X | X | , ve 1 | Sedic | SUP | X | | X | | X | | | | | | | | | | | | X | |
| analyses <sup>c,m</sup> Confidential | | eric | anno | | | | | | Pe | age 120 | ) of 19 | 0 | | | | | | | | | | | | |



 Table 5-1:
 Schedule of study assessments

| Table 5-1: | Sch | edu | le of | stud | y ass | sessr | ment | S | | | | | | | | | | | \ر | ailail | | | Apr 20<br>PS00 | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit <sup>a</sup> /<br>Week | Screening | | | | | Doub | | | al Treat | tment I<br>dose) | Period | | | | | Dos | | 00 | intena<br>Perioc<br>ofter fi | l | | ent | W56PEO<br>T | SFIT |
| Protocol activity | | Baseline<br>(first dose) | 1 | 3 | 4 | 5, 7 | 8 | 9,<br>11 | 12 | 13,<br>15 | 16 | 17,<br>19 | 20 | 21, 23 | 242 | 28 | 32 | 36 | 40 | 44 | 48 | 52 | 56 | |
| Blood sample<br>genetic/epigenetic<br>analyses <sup>c,m</sup> | | X | | | | | | | | | | 4 | 1110 | dion | <i>r</i> | | | | | | | | X | |
| PASI | X | X | X | X | X | | X | | X | | X | 27 | X, | | X | X | X | X | X | X | X | X | X | X |
| IGA | X | X | X | X | X | | X | | X | | X | ijor | X | | X | X | X | X | X | X | X | X | X | X |
| DLQI | | X | X | X | X | | X | | X | | XV | 0- | | | X | | X | | X | | X | | X | |
| PHQ-9 | X | X | | | X | | X | | X | | X | | X | | X | X | X | X | X | X | X | X | X | |
| eC-SSRS | X | X | X | X | X | X | X | X < | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Patient Symptom<br>Diary (daily) | | X | X | X | X | X | X | X | X | X | X | X | X | X | | | | | | | | | | |
| scalp IGA | | X | X <sup>n</sup> | X <sup>n</sup> | Xn | | Xn | 74. | X <sup>n</sup> | | X <sup>n</sup> | | | | X <sup>n</sup> | | X <sup>n</sup> | | Xn | | Xn | | X <sup>n</sup> | |
| mNAPSI | | X | | | Xº | | XoO | | Xº | | Xº | | | | Xº | | Xº | | Xº | | Xº | | Xº | |
| pp-IGA | | X | Xp | Xp | Xp | 191 | Xp | | Xp | | X <sup>p</sup> | | | | X <sup>p</sup> | | X <sup>p</sup> | | Xp | | Xp | | Xp | |
| EQ-5D-3L | | X | | | X | S | X | | X | | X | | | | X | | | | X | | | | X | |
| SF-36 | | X | | | X | | X | | X | | X | | | | X | | | | X | | | | X | |
| Patient global assessment of psoriasis <sup>q</sup> | | | Č | be | | | | | | | | | | | X | | X | | X | | X | | X | |
| PASE Confidential | | X | SILIVE | | | | | | | | | | | | | | | | | | | | X | |

# 96 Apr 2018 PS0008

Table 5-1: Schedule of study assessments

| Visit <sup>a</sup> /<br>Week | Screening | | | | | Douk | | d Initia<br>eks afte | | tment l<br>dose) | Period | | | | | Do | 4 | .00 | intena<br>Period<br>ofter fi | d | | nent | W56PEO<br>T | $\mathbf{SFU^b}$ |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Protocol activity | | Baseline<br>(first dose) | 1 | 3 | 4 | 5, 7 | 8 | 9,<br>11 | 12 | 13,<br>15 | 16 | 17,<br>19 | 20 | 21, 23 | 242 | 28 | 32 | 36 | 40 | 44 | 48 | 52 | 56 | |
| PGADA <sup>r</sup> | | X | | | X | | X | | X | | X | | | HOI | X | | X | | X | | X | | X | |
| WPAI-SHP V2.0 | | X | | | | | | | | | X | 1 | dic | 0 | X | | | | X | | | | X | |
| Concomitant medication | X | X | X | X | X | X | X | X | X | X | XO | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Adverse events | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| IRT <sup>s,t</sup> | X | X | X | X | X | X | X | X | X | X, | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Bimekizumab,<br>adalimumab, or<br>placebo<br>administration <sup>s,t</sup> | | X | X | X | X | X | X | x | X<br>X<br>X | X SIL | X | X | X | X | X <sup>u</sup> | X | X | X | X | X | X | X | | |

CV=cardiovascular; DLQI=Dermatology Life Quality Index; ECG=electrocardiogram; eCRF=electronic Case Report Form; eC-SSRS=electronic Columbia Suicide Severity Rating Scale; EQ-5D-3L=Euro-Quality of Life 5-Dimensions 3 Levels; GI=gastrointestinal HIV=human immunodeficiency virus; ICF=Informed Consent Form; IGA=Investigator's Global Assessment; IGRA=interferon-gamma release assay; IMP=investigational medicinal product; IRT=interactive response technology; PASE=Psoriatic Arthritis Screening and Evaluation; PASI=psoriasis area severity index; PEOT=Premature End of Treatment Visit; PGADA=Patient Global Assessment of Disease Activity; PHQ-9=Patient Health Questionnaire-9; PsA=psoriatic arthritis; SF-36=Short Form 36-item Health Survey; SFU=Safety Follow-Up; scalp IGA=scalp-specific Investigator's Global Assessment; TB=tuberculosis; VAS=visual analog scale; WPAI-SHP=Work Productivity and Activity Impairment Questionnaire-specific health problem

- <sup>a</sup> Visit windows of ±3 days from the first dose at all visits except SFU. The SFU Visit window is -3 and +7 days from last dose.
- <sup>b</sup> The SFU Visit will occur 20 weeks after the last dose.
- <sup>c</sup> A separate ICF will be required for subjects who decide to participate in the genomics, genetics, and proteomics substudy. The ICF must be signed prior to collecting any samples for the substudy. The samples will be stored at -80°C at the central biorepository for up to 20 years.
- <sup>d</sup> A separate ICF is required to be completed for the open-label study.
- <sup>e</sup> Ensure no significant changes in medical history.
- f Includes evaluation of signs and symptoms of active TB and risk for exposure to TB.
- <sup>g</sup> The physical examination will include examination of the following systems: eyes, hair, and skin; respiratory; CV; and GI.
- h Vital signs (blood pressures, pulse rate, and temperature) are to be measured prior to blood sampling, and prior to dosing, where applicable.


# Table 5-1: Schedule of study assessments

| Visit <sup>a</sup> /<br>Week | Screening | | | | | Doub | | d Initia | | tment l<br>dose) | Period | | | | | Dose-bl | | Perio | d | | ent | WS6PEO<br>T | $SFU^b$ |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Protocol activity | | Baseline<br>(first dose) | 1 | 3 | 4 | 5, 7 | 8 | 9,<br>11 | 12 | 13,<br>15 | 16 | 17,<br>19 | 20 | 21, 23 | 240 | 28 32 | 36 | 40 | 44 | 48 | 52 | 56 | |

Pregnancy testing will consist of serum testing at the Screening. The pregnancy test will be urine at all other visits.

Subjects who have evidence of or test positive for hepatitis B by any of the following criteria: 1) positive for hepatitis B surface antigen (HBsAg+); 2) positive for anti-hepatitis B core antibody (HBcAb+) are excluded. A positive test for HCV is defined as 1) positive for hepatitis C antibody (anti-HCV Ab), and 2) positive via a confirmatory test for HCV (for example, HCV polymerase chain reaction) are also excluded. Subjects will also be tested for anti-hepatitis B surface antibody.

<sup>k</sup> The HIV test results will not be recorded in the eCRF.

<sup>1</sup> Screening chest x-ray must occur within 3 months prior to Screening Visit.

<sup>m</sup> All blood samples taken prior to dosing.

<sup>n</sup> The scalp IGA will only be assessed for those subjects with scalp involvement (scalp IGA score >0) at Baseline.

<sup>o</sup> The mNAPSI will be assessed only in subjects with nail involvement (mNAPSI score >0) at Baseline.

<sup>p</sup> The pp-IGA will only be assessed in subjects with palmoplantar involvement (pp-IGA score >0) at Baseline.

<sup>q</sup> The Patient Global Assessment of psoriasis will be performed as part of the patient symptoms diary on a weekly basis from baseline through the initial treatment period with a +3 day completion window. During the maintenance period this assessment will be completed at each clinic visit specified with a ±3 day completion window.

<sup>r</sup> The PGADA is assessed only for subjects with PsA at Baseline (defined as a past medical history of PsA or PASE ≥47).

<sup>s</sup> IMP administration is based on randomization.

<sup>t</sup> For bimekizumab, the minimum time between doses should be no less than 24 days and no more than 32 days.

<sup>u</sup> At Week 24 subjects will be re-allocated based on original treatment and response to treatment and will receive their first Maintenance Treatment Period dose.

06 Apr 2018 PS0008 Bimekizumab

Table 5-1: Schedule of study assessments

| Visit <sup>a</sup> /<br>Week | Screening | | | Douk | ole-blin<br>(wee | d Initia | | | Period | | | | ] | Dose-bli | | intena<br>ks aft | | | | eriod | | | W56/PEOT | SFU |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Protocol activity | | Baseline<br>(first dose) | 1 | 3 | 4 | 5, 7 | 8 | 9,<br>11 | 12 | 13,<br>15 | 16 | 17,<br>19 | 20 | 21, 23 | 24 7 | 28 | 32 | 36 | 40 | 44 | 48 | 52 | 56 | S |
| Informed consent <sup>c</sup> | X | | | | | | | | | | | | | dion | | | | | | | | X <sup>d</sup> | | |
| Inclusion/exclusion | X | X | | | | | | | | | | -1 | die | 30 | | | | | | | | | | |
| Urine drug screen | X | | | | | | | | | | -0 | 8 | 96, | | | | | | | | | | X | |
| Demographic data | X | | | | | | | | | _< | | XiO! | | | | | | | | | | | | |
| Psoriasis history | X | | | | | | | | | CV. | oiil | | | | | | | | | | | | | |
| Significant past<br>medical history<br>and concomitant<br>diseases | X | Xe | | | | | | 4 | 2 ED | O DU | | | | | | | | | | | | | | |
| Physical examination <sup>f,g</sup> | X | | | | | | | 74 | X | | X | | | | X | | | X | | | X | | X | X |
| Height | | X | | | | | X | | | | | | | | | | | | | | | | | |
| Body weight | | X | | | | 5. | 20 | | | | X | | | | X | | | X | | | X | | X | |
| Vital signs <sup>h</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Hematology and biochemistry | X | X | X | X | XO. | | X | | X | | X | | X | | X | | X | | X | | X | | X | X |
| Urinalysis | X | X | | 'Se' | ) | | | | | | X | | | | X | | X | | X | | X | | X | X |
| ECG | X | | 20,00 | | | | | | | | X | | | | X | | | X | | | X | | X | |
| Pregnancy testing <sup>i</sup> | X | X | Sall | | X | | X | | X | | X | | X | | X | X | X | X | X | X | X | X | X | X |
| Confidential | CUIT | ent | | | | | | | P | age 12 | 4 of 19 | 90 | | | | | | | | | | | | |

Table 5-1: Schedule of study assessments

| UCB<br>Clinical Study Pro | toco | 1 | | | | | | | ] | Bimeki | zumab | ) | | | | | | | | | S | | Apr 20<br>PS00 | 018<br>008 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Table 5-1: Sivisit <sup>a</sup> / Week | Screening | | le of | Stud<br>Doub | ole-blin | d Initia | | tment l | Period | | | | 1 | Dose-bli | | aintena<br>eks aft | | reatu | ent P | eriod | | | W56/PEOT | SFUb |
| Protocol activity | | Baseline<br>(first dose) | 1 | 3 | 4 | 5, 7 | 8 | 9,<br>11 | 12 | 13,<br>15 | 16 | 17,<br>19 | 20 | 21, 23 | 24 | 28 | 32 | 36 | 40 | 44 | 48 | 52 | 56 | IS |
| Hepatitis B and C testing <sup>j</sup> | X | | | | | | | | | | | | | ation | | | | | | | | | | |
| HIV testing <sup>k</sup> | X | | | | | | | | | | < | 7 | 20 by | | | | | | | | | | | |
| Chest x-ray <sup>l</sup> | X | | | | | | | | | | CO | 70: | 0. | | | | | | | | | | | |
| IGRA Tuberculosis<br>test | X | | | | | | | | | | Dill | dil | | | | | | | | | | X | | |
| Tuberculosis<br>questionnaire | X | X | | | | | | | CO | an'i | X | | | | X | | | X | | X | | X | X | X |
| Blood sample for<br>bimekizumab<br>plasma<br>concentrations <sup>m</sup> | | X | X | X | X | | X | , 10 | Xeil | (9) | X | | X | | X | | | X | | | X | | X | X |
| Blood sample for<br>anti-bimekizumab<br>antibodies <sup>m</sup> | | X | | | X | 4 | X | 12 | X | | X | | X | | X | | | X | | | X | | X | X |
| Blood sample<br>genomic,<br>proteomic, and<br>metabolomics, and<br>candidate<br>biomarker<br>analyses <sup>c,m</sup> | | X | X | 100 | sedi | SUR | X | | X | | X | | | | | | | | | | | | X | |



Table 5-1: Schedule of study assessments

| Visit <sup>a</sup> /<br>Week | Screening | | | Doub | | d Initia | | | Period | | | | I | Dose-blii | | intena<br>ks afte | | | lent P | | | | Apr 20<br>PS00 | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Protocol activity | | Baseline<br>(first dose) | 1 | 3 | 4 | 5, 7 | 8 | 9,<br>11 | 12 | 13,<br>15 | 16 | 17,<br>19 | 20 | 21,<br>23 | 24 7 | 28 | 32 | 36 | 40 | 44 | 48 | 52 | 56 | SFIIb |
| Blood sample<br>genetic/epigenetic<br>analyses <sup>c,m</sup> | | X | | | | | | | | | | 1 | dic | ation | | | | | | | | | X | |
| PASI | X | X | X | X | X | | X | | X | | X | 5 | X | | X | X | X | X | X | X | X | X | X | X |
| IGA | X | X | X | X | X | | X | | X | .< | X, | ijor | X | | X | X | X | X | X | X | X | X | X | X |
| Percentage of<br>BSA | X | X | X | X | X | | X | | X | S, | N/I | | X | | X | X | X | X | X | X | X | X | X | X |
| DLQI | | X | X | X | X | | X | | X | 300 | X | | X | | X | | X | | X | | X | | X | |
| PHQ-9 | X | X | | | X | | X | | X | 9 | X | | X | | X | X | X | X | X | X | X | X | X | |
| eC-SSRS | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Patient Symptom<br>Diary (daily) | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | | | | | | | | | |
| scalp IGA | | X | X <sup>n</sup> | Xn | Xn | .4 | Xn | | X <sup>n</sup> | | Xn | | X <sup>n</sup> | | Xn | | X <sup>n</sup> | | Xn | | Xn | | X <sup>n</sup> | |
| mNAPSI | | X | | | Xº | SUP | Xº | | Xº | | Xº | | Xº | | Xº | | Xº | | Xº | | Xº | | Xº | |
| pp-IGA | | X | X <sup>p</sup> | Хp | X <sup>p</sup> X | Ď. | Xp | | Xp | | Xp | | Xp | | Xp | | Xp | | Xp | | Xp | | Xp | |
| EQ-5D-3L | | X | | , i | | | X | | X | | X | | | | X | | | | X | | | | X | |
| SF-36 Confidential | | X | | 100 | X | | X | | X | | X | | | | X | | | | X | | | | X | |

Apr 2018 PS0008

Table 5-1: Schedule of study assessments

| Visit <sup>a</sup> /<br>Week | Screening | | | Doul | | d Initia | | | Period | | | | I | Dose-bli | | nintena<br>eks aft | | . ( ). | | eriod | | | W56/PEOT | SFUb |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Protocol activity | | Baseline<br>(first dose) | 1 | 3 | 4 | 5, 7 | 8 | 9,<br>11 | 12 | 13,<br>15 | 16 | 17,<br>19 | 20 | 21, 23 | 24 | 28 | 32 | 36 | 40 | 44 | 48 | 52 | 56 | S |
| Patient global<br>assessment of<br>psoriasis <sup>q</sup> | | | | | | | | | | | | _1 | 0/1/ | ation. | X | | X | | X | | X | | X | |
| PASE | | X | | | | | | | | | -C | | 964 | | | | | | | | | | X | |
| PGADA <sup>r</sup> | | X | | | X | | | | X | _< | X | ijo | | | X | | X | | X | | X | | X | |
| WPAI-SHP V2.0 | | X | | | | | | | | C | Xil | | | | X | | | | X | | | | X | |
| Concomitant medication | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Adverse events | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| IRT <sup>s,ŧ</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Bimekizumab,<br>adalimumab, or<br>placebo<br>administration <sup>s,†</sup> | | X | X | X | X | X | X | X | X | X | X | X | X | X | Xu | X | X | X | X | X | X | X | | |

BSA=body surface area; CV=cardiovascular; DLQI=Dermatology Life Quality Index; ECG=electrocardiogram; eCRF=electronic Case Report Form; eC-SSRS=electronic Columbia Suicide Severity Rating Scale; EQ-5D-3L=Euro-Quality of Life 5-Dimensions 3 Levels; GI=gastrointestinal HIV=human immunodeficiency virus; ICF=Informed Consent Form; IGA=Investigator's Global Assessment; IGRA=interferon-gamma release assay; IMP=investigational medicinal product; IRT=interactive response technology; PASE=Psoriatic Arthritis Screening and Evaluation; PASI=psoriasis area severity index; PEOT=Premature End of Treatment Visit; PGADA=Patient Global Assessment of Disease Activity; PHQ-9=Patient Health Questionnaire-9; PsA=psoriatic arthritis; SF-36=Short Form 36-item Health Survey; SFU=Safety Follow-Up; scalp IGA=scalp-specific Investigator's Global Assessment; TB=tuberculosis; VAS=visual analog scale; WPAI-SHP=Work Productivity and Activity Impairment Questionnaire-specific health problem a Visit windows of ±3 days from the first dose at all visits except SFU. The SFU Visit window is -3 and +7 days from last dose.

<sup>&</sup>lt;sup>b</sup> The SFU Visit will occur 20 weeks after the last dose for subjects who do not enroll in the open-label study.

- <sup>c</sup> A separate ICF will be required for subjects who decide to participate in the genomics, genetics, and proteomics substudy. The ICF must be signed prior to collecting any samples for the substudy. The samples will be stored at -80°C at the central biorepository for up to 20 years.
- <sup>d</sup> A separate ICF is required to be completed for the open-label study.
- <sup>e</sup> Ensure no significant changes in medical history.
- <sup>f</sup> Includes evaluation of signs and symptoms of active TB and risk for exposure to TB.
- g The physical examination will include examination of the following systems: eyes, hair, and skin; respiratory; CV; and GI.
- h Vital signs (blood pressures, pulse rate, and temperature) are to be measured prior to blood sampling, and prior to dosing, where applicable.
- <sup>1</sup> Pregnancy testing will consist of serum testing at the Screening. The pregnancy test will be urine at all other visits.
- Subjects who have evidence of or test positive for hepatitis B by any of the following criteria: 1) positive for hepatitis B surface antigen (HBsAg+); 2) positive for anti-hepatitis B core antibody (HBcAb+) are excluded. A positive test for HCV is defined as: 1) positive for hepatitis C antibody (anti-HCV Ab), and 2) positive via a confirmatory test for HCV (for example, HCV polymerase chain reaction) are also excluded. Subjects will also be tested for anti-hepatitis B surface antibody.
- <sup>k</sup> The HIV test results will not be recorded in the eCRF.
- <sup>1</sup> Screening chest x-ray must occur within 3 months prior to Screening Visit.
- <sup>m</sup> All blood samples taken prior to dosing.
- <sup>n</sup> The scalp IGA will only be assessed for those subjects with scalp involvement (scalp IGA score 0) at Baseline.
- o The mNAPSI will be assessed only in subjects with nail involvement (mNAPSI score >0) at Baseline.
- <sup>p</sup> The pp-IGA will only be assessed in subjects with palmoplantar involvement (pp-IGA score >0) at Baseline.
- <sup>q</sup> The Patient Global Assessment of psoriasis will be performed as part of the patient symptoms diary on a weekly basis from **baselineScreening** through the Initial Treatment Period with a +3 day completion window. During the **Maintenance Treatment Period** this assessment will be completed at each clinic visit specified with a ±3 day completion window.
- The PGADA is assessed for all subjects at Baseline. At all subsequent visits, the PGADA is only for subjects with PsA at Baseline (defined as a past medical history of PsA or PASE ≥47).
- <sup>s</sup> IMP administration is based on randomization.
- <sup>‡</sup> For bimekizumab, the minimum time between doses should be no less than 24 days and no more than 32 days.
- \*At Week 24 subjects will be re-allocated based on original treatment and response to treatment and will receive their first Maintenance Treatment

  Period


#### Change #15

Figure 5-1: Schematic diagram of PS0008



PASI=Psoriasis Area and Severity Index; Q4W=every 4 weeks; Q8W=every 8 weeks; SFU=Safety Follow-Up

Note: If a subject does not achieve a PASI50 response at Week 36 or later, the subject will be withdrawn from the study at the time point when the PASI50 response is not achieved.

Note: Refer to Section 5.2.2 for treatments during the Initial Treatment Period and to Section 5.2.3 for treatments during the Maintenance Treatment Period.

Figure 5-1: Schematic diagram of PS0008



Note: If a subject does not achieve a PASI50 response at Week 36 or later, the subject will be withdrawn from the study at the time point when the PASI50 response is not achieved.

Note: Refer to Section 5.2.2 for treatments during the Initial Treatment Period and to Section 5.2.3 for treatments during the Maintenance Treatment Period.

#### Change #16

#### Section 5.8.1 Study design

A randomized, active-controlled study design has been selected to demonstrate efficacy and safety of bimkizumab for regulatory approval. The study population will include adults with moderate to severe chronic plaque PSO and allow subjects who have received previous biologic treatment as well as those who are biologic treatment naïve. The primary efficacy outcome measures (based on PASI and IGA) and other efficacy assessments included in this study are consistent with those used for other PSO studies and are considered appropriate for establishing efficacy of bimekizumab. An initial treatment period of 24 weeks will be used to demonstrate the efficacy of bimekizumab compared with adalimumab. The study duration extends beyond the initial treatment period (to 56 weeks) to allow for collection of long-term safety and efficacy data.

At Week 24, subjects on adalimumab treatment are re-allocated to treatment with bimekizumab 320mg Q4W. This allows for a controlled evaluation of the safety and efficacy of switching from a product with one mechanism of action to another, which is known to occur in clinical practice due to either loss of response or access. In a recent PSO study in which subjects were switched from adalimumab to a treatment with a different mechanism of action there was no evidence of an increased safety risk following the switch (Reich et al, 2017)

#### Has been changed to:

A randomized, active-controlled study design has been selected to demonstrate efficacy and safety of bimkizumab for regulatory approval. The study population will include adults with moderate to severe chronic plaque PSO and allow subjects who have received previous biologic treatment as well as those who are biologic treatment naïve. The primary efficacy outcome measures (based on PASI and IGA) and other efficacy assessments included in this study are consistent with those used for other PSO studies and are considered appropriate for establishing efficacy of bimekizumab. An initial treatment period of 1624 weeks will be used to demonstrate the efficacy of bimekizumab compared with adalimumab. The study duration extends beyond the initial treatment period (to 56 weeks) to allow for collection of long-term safety and efficacy data.

At Week 24, subjects on adalimumab treatment are re-allocated to treatment with bimekizumab 320mg Q4W. This allows for a controlled evaluation of the safety and efficacy of switching from a product with one mechanism of action to another, which is known to occur in clinical practice due to either loss of response or access. In a recent PSO study in which subjects were switched from adalimumab to a treatment with a different mechanism of action, there was no evidence of an increased safety risk following the switch without washout (Reich et al, 2017).

## Change #17

#### Section 5.8.1 Study design

#### The following paragraph has been deleted:

If subjects do not respond after a switch in treatment or if they lose response over time, the mandatory withdrawal criterion for subjects who do not achieve a PASI50 response at Week 36 or later will ensure that subjects do not continue to receive prolonged exposure to study

 treatment that is providing a sub-optimal response, regardless of their initial randomized treatment.

#### Change #18

#### Section 6.2 **Exclusion criterion #22**

#### The following criterion has been deleted.

sions or variations thereof 1. Subject has been exposed to more than 3 biological response modifiers (including no more than 1 IL-17).

#### Change #19

#### Section 6.2 **Exclusion criterion #23**

2. Subject has experienced one primary failure to an IL-17 biological response modifier (no response within 12 weeks).

#### Has been changed to:

3. Subject has experienced one primary failure to an IL-17 biological response modifier (no response within 12 weeks) to 1 or more IL-17 biologic response modifier (eg, brodalumab, ixekizumab, secukinumab) OR more than 1 biologic response modifier other than an IL-17.

#### Change #20

#### Section 6.2 **Exclusion criterion #27**

27. Subject has presence of severe depression, indicated by a score ≥15 using the screening PHQ-9. Medication used to treat depression should be stable for 4 weeks prior to baseline.

Has been changed to:

27. Subject has presence of severe depression, indicated by a score ≥of 15 to 19 using the screening PHQ 9. Medication used to treat depression should be stable for 4 weeks prior to Baseline.

#### Change #21

# Section 6.3 Withdrawal criterion #2

2. Moderately severe depression as indicated by a PHQ-9 score ≥15 if this represents an increase of 3 points compared to last visit.

#### Has been changed to:

2. Moderately severe depression as indicated by a PHQ-9 score  $\geq$  of 15 to 19 if this represents an increase of 3 points compared to last visit.

#### Change #22

#### Section 6.3 Withdrawal criterion #3

#### The following criterion has been deleted:

Subject does not achieve a PASI50 response at Week 26 or later.

Change #23

#### Section 7.2 Treatment(s) to be administered

Bimekizumab

- Subjects randomized to receive adalimumab will receive 2 adalimumab 40mg injections sc at Week 0 (Baseline). At Weeks 1, 3, 5, 7, 9, 11, 13, 15, 17, 19, 21, and 23 they will receive 1 adalimumab 40mg injection sc. These subjects will receive 2 placebo injections at Weeks 4, 8, 12, 16, and 20.

#### Maintenance Treatment Period dosing

Investigational medicinal product treatment during the Maintenance Treatment Period will be based on initial treatment and response to treatment at Week 24 as described in Section 5.2.3.

- Subjects who receive bimekizumab 320mg Q4W will receive 2 bimekizumab 160mg injections sc Q4W at Weeks 24, 28, 32, 36, 40, 44, 48, and 52. Note: Subjects initially randomized to adalimumab who switch to bimekizumab 320mg Q4W at Week 24 will receive their first bimekizumab 320mg dose at Week 24.
- Subjects who receive bimekizumab 320mg Q8W will receive 2 bimekizumab 160mg injections sc Q8W at Weeks 24, 32, 40, and 48. These subjects will receive 2 placebo injections at Weeks 28, 36, 44, and 52.

This document cannot be used to support The dosing scheme is depicted in Table 7-1.

**Table 7-1: Dosing Scheme** 

| | | | | | In | itial T | reatme | nt | | | | | | | | Main | <del>o`</del><br>tenanc | ee | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Week Dose Assignment | 0 | 1, | 4 | 5,<br>7 | 8 | 9,<br>11 | 12 | 13,<br>15 | 16 | 17,<br>19 | 20 | 21,<br>23 | 24 | 28 | 32 | <b>36</b> | 40 | 44 | 48 | 52 |
| bimekizumab 320mg<br>Q4W/Q4W | •• | 0 | •• | 0 | •• | 0 | •• | 0 | •• | 0 | •• | 0 | •• | ete | •• | •• | •• | •• | •• | •• |
| bimekizumab 320mg<br>Q4W/Q8W | •• | 0 | •• | 0 | •• | 0 | •• | 0 | •• | 0 | •• | ٥ | 36 | 00 | •• | 00 | •• | 00 | •• | 00 |
| adalimumab 40mg | <b>A A</b> | <b>A</b> | 00 | <b>A</b> | 00 | <b>A</b> | 00 | <b>A</b> | 00 | <b>A</b> | 00 | -17A | •• | •• | •• | •• | •• | •• | •• | •• |

NR=nonresponder; Q4W=every 4 weeks; Q8W=every 8 weeks
Notes: A bimekizumab 160mg injection is depicted by a black circle (•). A placebo injection is depicted by a white circle (o). An adalimumab 40mg injection is

#### **Double blind Initial Treatment Period dosing**

During the Initial Treatment Period, Eligible subjects will be randomized 1:1:1 to receive the following blinded study treatment regimens: bimekizumab 320mg Q4W throughout the study, bimekizumab 320mg Q4W through Week 16, or adalimumab.

Because of differences in the dosing schedule between bimekizumab and adalimumab and in order to maintain blinding, all subjects will receive 2 injections sc on Weeks 0 (Baseline), 4, 8, 12, 16, and 20, and 24 and 1 injection sc in other weeks based on the following dosing scheme:

- Subjects randomized to receive bimekizumab 320mg Q4W **throughout the study** will receive 2 bimekizumab 160mg injections sc Q4W at Weeks 0 (Baseline), 4, 8, 12, 16, and 20, 24, 28, 32, 36, 40, 44, 48, and 52. These subjects will receive 1 placebo injection at Weeks 1, 3, 5, 7, 9, 11, 13, 15, 17, 19, 21, and 23.
- Subjects randomized to receive bimekizumab 320mg Q4W/Q8W will receive 2 bimekizumab 160mg injections sc Q4W at Weeks 0 (Baseline), 4, 8, and 12. Subjects will then receive 2 bimekizumab 160mg injections sc Q8W at Weeks 16, 24, 32, 40, and 48. These subjects will receive 1 placebo injection at Weeks 1, 3, 5, 7, 9, 11, 13, 15, 17, 19, 21, and 23, and 2 placebo injections at Weeks 20, 28, 36, 44, and 52.
- Subjects randomized to receive adalimumab will receive 2 adalimumab 40mg injections sc at Week 0 (Baseline). At Weeks 1, 3, 5, 7, 9, 11, 13, 15, 17, 19, 21, and 23, they will receive 1 adalimumab 40mg injection sc. These subjects will receive 2 placebo injections at Weeks 4, 8, 12, 16, and 20. These subjects will then receive bimekizumab 320mg Q4W given as 2 bimekizumab 160mg injections sc Q4W at Weeks 24, 28, 32, 36, 40, 44, 48, and 52.

#### **Maintenance Treatment Period dosing**

Investigational medicinal product treatment during the Maintenance Treatment Period will be based on initial treatment and response to treatment at Week 24 as described in Section 5.2.3.

- Subjects who receive bimekizumab 320mg Q4W will receive 2 bimekizumab 160mg injections sc Q4W at Weeks 24, 28, 32, 36, 40, 44, 48, and 52. Note: Subjects initially randomized to adalimumab who switch to bimekizumab 320mg Q4W at Week 24 will receive their first bimekizumab 320mg dose at Week 24.
- Subjects who receive bimekizumab 320mg Q8W will receive 2 bimekizumab 160mg injections se Q8W at Weeks 24, 32, 40, and 48. These subjects will receive 2 placebo injections at Weeks 28, 36, 44, and 52.

The dosing scheme is depicted in Table 7-1.

**Table 7-1: Dosing Scheme** 

| UCB<br>Clinical Study Protocol Table 7-1: Dosi | na Sa | chem | | | | | E | Bimekiz | umab | | | | | | | | i dil | us ill | 06 Apr<br>Ps | 2018<br>\$0008 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Week | 0 | 1 | 4 | Initia | al Treat | tment<br>9, | 12 | 13, | 16 | 17, | 20 | 21, | Ma<br>24 | inten<br>28 | ance T | reatm | 3/10 | 44 | 48 | 52 |
| Dose Assignment | U | 3 | 4 | 7 | 0 | 11 | 12 | 15, | 10 | 19 | 20 | 23 | 24 | 20 | Sion | 5 30 | 40 | 44 | 40 | 32 |
| bimekizumab 320mg<br>Q4W/Q4W | •• | 0 | •• | 0 | •• | 0 | •• | 0 | •• | 0 | •• | 0 | •• | ete | •• | •• | •• | •• | •• | •• |
| bimekizumab 320mg<br>Q4W/Q8W | •• | 0 | •• | 0 | •• | 0 | •• | 0 | •• | 0 | 00 | · | 86 | 00 | •• | 00 | •• | 00 | •• | 00 |
| adalimumab 40mg | <b>A A</b> | <b>A</b> | 00 | <b>A</b> | 00 | <b>A</b> | 00 | <b>A</b> | 00 | <b>A</b> | 00 | 11/201 | •• | •• | •• | •• | •• | •• | •• | •• |

NR=nonresponder; Q4W=every 4 weeks; Q8W=every 8 weeks

Notes: A bimekizumab 160mg injection is depicted by a black circle (•). A placebo injection is depicted by a white circle (o). An adalimumab 40mg injection is


### Change #24

#### Section 7.8.1 Permitted concomitant treatments (medications and therapies)

## The following was deleted:

The following concomitant medications are permitted during the study.

#### Change #25

## Table 7-2 Prohibited psoriasis medications

| Other biologics and other systemic therapies: | 2501 |
|---|---|
| apremilast, tofacitinib | 2 weeks for apremilast and tofacitinib |
| alefacept, efalizumab, guselkimab | 3 months for alefacept, efalizumab, and guselkimab |
| ustekinumab, briakinumab | 6 months for ustekinumab and briakinumab |
| rituximab | 12 months for rituximab |
| Anti-IL-17 therapy | 3 months |
| | (bimekizumab is excluded per exclusion criteria) |
| | criteria |

#### Has been changed to:

| Other biologics and other systemic therapies: | |
|---|---|
| apremilast, tofacitinib | 2 weeks for apremilast and tofacitinib |
| alefacept, efalizumab, guselkumab | 3 months for alefacept, efalizumab, and guselkumab |
| ustekinumab, briakinumab | 6 months for ustekinumab and briakinumab |
| rituximab | 12 months for rituximab |
| Anti-IL-17 therapy: | 3 months |
| brodalumab | (bimekizumab is excluded per exclusion |
| ixekizumab | criteria) |
| secukinumab | |

#### Change #26

# Section 7.10 Randomization and numbering of subjects

An IRT will be used for assigning eligible subjects to a treatment regimen based on a predetermined production randomization and/or packaging schedule provided by UCB (or designee). The randomization schedule will be produced by the IRT vendor. The IRT will generate individual assignments for subject kits of IMP, as appropriate, according to the visit schedule. Subject treatment assignment will be stratified by region and prior biologic exposure (yes/no). The IRT will generate individual assignments for subject kits of IMP, as appropriate, according to the visit schedule. Efforts should be made to limit the enrollment of subjects with prior biologic exposure to approximately 30% of the total study population.

An IRT will be used for assigning eligible subjects to a treatment regimen based on a predetermined production randomization and/or packaging schedule provided by UCB (or isions of variations thereof. designee). The randomization schedule will be produced by the IRT vendor. The IRT will generate individual assignments for subject kits of IMP, as appropriate, according to the visit schedule. Subject treatment assignment will be stratified by region and prior biologic exposure (yes/no). The IRT will generate individual assignments for subject kits of IMP, as appropriate, according to the visit schedule. Efforts should be made to limit the enrollment of subjects with prior biologic exposure to approximately 30% of the total study population.

#### Change #27

#### Section 7.10 Randomization and numbering of subjects

#### The following sentence has been deleted:

At Week 24, subjects may be reallocated to a new treatment group based on their PASI response.

#### Change #28

**Section 8 Study Procedures by Visit** 

The following has been deleted from the bulleted list:

The minimum of time between doses should be no less than 21 days and no more than 35 days.

#### Change #29

Sections 8.1 Screening Visit (2 to 4 weeks), 8.2.1 Baseline Visit, 8.2.2 Week 1 (±3 days), 8.2.3 Week 3 ( $\pm 3$  days), 8.2.4 Week 4 ( $\pm 3$  days), 8.2.6 Week 8 ( $\pm 3$  days), 8.2.8 Week 12 ( $\pm 3$  days), 8.2.10 Week 16 (±3 days), 8.3.2 Week 20 (±3 days), 8.3.4 Week 24 (±3 days), 8.3.5 Week 28 (±3 days), 8.3.6 Week 32 (±3 days), 8.3.7 Week 36 (±3 days), 8.3.8 Week 40 (±3 days), 8.3.9 Week 44 (±3 days), 8.3.10 Week 48 (±3 days), 8.3.11 Week 52 (±3 days), 8.3.12 Week 56 (±3 days), and 8.5 Safety Follow-Up Visit (20 weeks after last dose -3/+7 days)

# The following has been added to the bulleted list:

Percentage of BSA

#### Change #30

Section 8.1 Screening Visit (2 to 4 weeks) and Section 8.3.4 Week 24 (±3 days)

#### The following has been added to the bulleted list:

Daily Patient Symptom Diary

#### Change #31

Section 8.2.1 Baseline Visit, Section 8.2.10 Week 16 (±3 days), and Section 8.3.8 Week 40 (±3 days)

- Obtain blood and urine samples for the following analyses prior to dosing:
  - Genomic, proteomic, metabolomics, and candidate biomarker analyses
  - Genetic/epigenetic analyses (for subjects participating in the substudy)

PGADA for subjects with PSA at Baseline

#### Has been changed to:

- Obtain blood and urine samples for the following analyses prior to dosing:
  - Genomic, proteomic, metabolomics, and candidate biomarker analyses (participating subjects only)
  - Genetic/epigenetic analyses (for-participating subjects only participating in the substudy)
- PGADA for subjects with PSA at Baseline

## Change #32

#### **Section 8.2.1 Baseline Visit**

After completion of the above-mentioned procedures, administration of bimekizumab, adalimumab, or placebo will occur.

#### Has been changed to:

After completion of the above-mentioned procedures, administration of bimekizumab, or adalimumab, or placebo will occur.

#### Change #33

#### Section 8.2.2 Week 1 (±3 days)

- Obtain blood samples for the following analyses prior to dosing:
  - Genomic, proteomic, metabolomics, and candidate biomarker analyses

#### Has been changed to:

- As been changed to:

  Obtain blood samples for the following analyses prior to dosing:
  - Genomic, proteomic, metabolomics, and candidate biomarker analyses (participating subjects only)

#### Change #34

#### Section 8.2.6 Week 8 (±3 days)

#### The following has been deleted from the bulleted list:

PGADA for subjects with PsA at Baseline

#### Change #35

#### Section 8.3.2 Week 16 (±3 days)

will occur. After completion of the above-mentioned procedures, administration of bimekizumab or placebo

#### Has been changed to:

After completion of the above-mentioned procedures, the Maintenance Treatment Period will begin with administration of bimekizumab or placebo will occur.

06 Apr 2018 PS0008

#### Change #36

The heading for Section 8.3 Dose-blind Maintenance Treatment Period has been moved to before Week 17 and 19 (±3 days), and the section was renumbered accordingly

#### Change #37

#### The following have been added to the bulleted list:

- Scalp IGA for subjects with scalp involvement at Baseline
- mNAPSI for subjects with nail involvement at Baseline

pp-IGA for subjects with palmoplantar involvement at Baseline

#### Change #38

Section 8.3.10 Week 48 ( $\pm 3$  days)

The following have been deleted from the bulleted list:

- EQ-5D-3L
- SF-36

#### Change #39

Section 8.3.11 Week 52 ( $\pm 3$  days)

#### The following bullet has been added:

... d.3.11 Week 52 (±3 days)

\*\*ollowing bullet has been added:

IGRA tuberculosis test; it is recommended that the QuantiFERON TB GOLD test be performed

#40

Assessment of Efficacy
ing text has been added:

3SA, IGA, scalp IGA, mNAPSI, and pp-IGA shor'
another delegated physician, or an appropr'
based on local requirements) who has been assessments correctly. Preferably
assessment.

asis Area and S

\*\*involve\*\*
nd\*\* The PASI, BSA, IGA, scale Torofoso. The PASI, BSA, IGA, scalp IGA, mNAPSI, and pp-IGA should be performed by the Investigator, another delegated physician, or an appropriately qualified medical professional (based on local requirements) who has had documented training on how to perform these assessments correctly. Preferably the same assessor should evaluate the subject at each assessment.

#### Change #41

# Section 9.1 Psoriasis Area and Severity Index

The percent area of involvement (BSA%) is estimated across 4 body areas; head, upper Has been changed to:

The percent area of involvement (BSA%) is estimated across 4 body areas; head, upper extremities, trunk, and lower extremities. Assessors will enter the degree of involvement for a given region **as a percentage (0 100%) which will then be mapped into a grade** on a scale of 0 **to** 6 (0=none; 1=1% to <10% affected, 2=10% to <30% affected, 3=30% to <50% affected, 4=50% to <70% affected, 5=70% to <90% affected, 6=90% to 100% affected) (Table 9-1).

#### Change #42

#### Section 9.1 Psoriasis Area and Severity Index

The total BSA affected by PSO will be derived based on the regional BSA values provided when assessing the PASI score.

#### Has been changed to:

The total BSA affected by PSO will be entered as a percentage from 0 to 100derived based on the regional BSA values provided when assessing the PASI score.

#### Change #43

#### **Section 9.11 Patient Symptom Diary responses**

UCB developed a new PRO measure that will be used to assess key symptoms relevant to patients with moderate to severe chronic plaque PSO. PS0010 used the draft PRO measure in selected countries to enable psychometric validation of the PRO. Site staff will train the participating subjects on the use of the electronic PRO (ePRO) diary at the Baseline Visit, following which the device will be dispensed to the subject for home use until the Week 16 Visit. The ePRO diary will be administered on a daily basis from Baseline to the Week 16 Visit.

#### Has been changed to:

UCB developed a new PRO measure that will be used to assess key symptoms relevant to patients with moderate to severe chronic plaque PSO. PS0010 used the draft PRO measure in selected countries to enable psychometric validation of the PRO. Site staff will train the participating subjects on the use of the electronic PRO (ePRO) diary at the **ScreeningBaseline** Visit, following which the device will be dispensed to the subject for home use until the Week 16 Visit. The ePRO diary will be administered on a daily basis from **ScreeningBaseline** to the Week 16 Visit.

#### Change #44

#### Section 12.1.1.4 Other safety topics of interest

#### The following paragraph has been deleted:

The following safety topics are prespecified as being of interest for this study, based on findings from the IMP clinical program to date, potential risks generally associated with biologic immunomodulators, or findings from other medicines belonging to the same class of drugs. There are no specific AE reporting requirements for these topics, however special monitoring, additional data collection activities, and/or enhanced signal detection activities (within UCB), are in place.

#### Change #45

#### **Section 12.2** Laboratory measurements

Clinical laboratory assessments consist of serum chemistry, hematology, and urinalysis. A centralized laboratory will be used to supply all laboratory test supplies and analyze all blood and urine samples for hematology, biochemistry, and urinalysis measurements. Any unscheduled laboratory testing should also be collected using the central laboratory. Testing to rule out hepatitis B, hepatitis C, and HIV (see Exclusion Criterion #9, Section 6.2) will be performed at Screening in addition to those measurements listed in Table 12.2.

Specific details regarding the handling and processing of serum chemistry, hematology, and urinalysis samples are provided in the study laboratory manuals.

The following laboratory parameters will be measured:

Table 12-2: Laboratory measurements

| Hematology | Chemistry | Urinalysis dipstick <sup>a</sup> |
|---|---|---|
| Basophils | Calcium | pH |
| Eosinophils | Chloride | Albumin (protein) |
| Lymphocytes | Magnesium | Glucose |
| Atypical lymphocytes | Potassium | Blood |
| Monocytes | Sodium | Leukocyte esterase |
| Neutrophils | Glucose | Nitrite |
| Hematocrit 0 | BUN | Urine dipstick for pregnancy testing <sup>b</sup> |
| Hemoglobin | Creatinine | |
| MCH | ALP | |
| MCHC | AST | |
| MCV | ALT | |
| Platelet count | GGT | |
| RBC count | Total bilirubin | |

# Table 12-2: Laboratory measurements

| Hematology | Chemistry | Urinalysis dipstick <sup>a</sup> |
|---|---|---|
| WBC count | LDH | |
| | Serum pregnancy testing <sup>b</sup> | |

ALP=alkaline phosphatase; ALT=alanine aminotransferase; AST=aspartate aminotransferase; BUN=blood urea nitrogen; ; GGT=gamma glutamyltransferase; LDH=lactate dehydrogenase; MCH=mean corpuscular hemoglobin; MCHC=mean corpuscular hemoglobin concentration; MCV=mean corpuscular volume; RBC=red blood cell; WBC=white blood cell

## Has been changed to:

Clinical laboratory assessments consist of serum chemistry, hematology, urinalysis, and urine drug screen. A centralized laboratory will be used to supply all laboratory test supplies and analyze all blood and urine samples for hematology, biochemistry, and urinalysis measurements. Any unscheduled laboratory testing should also be collected using the central laboratory. Testing to rule out hepatitis B, hepatitis C, and HIV (see Exclusion Criterion #9, Section 6.2) will be performed at Screening in addition to those measurements listed in Table 12-2.

Specific details regarding the handling and processing of serum chemistry, hematology, and urinalysis samples are provided in the study laboratory manuals.

The following laboratory parameters will be measured:

Table 12-2: Laboratory measurements

| Hematology | Chemistry | Urinalysis dipstick <sup>a</sup> |
|---|---|---|
| Basophils | Calcium | pН |
| Eosinophils | Chloride | Albumin (protein) |
| Lymphocytes | Magnesium | Glucose |
| Atypical lymphocytes | Potassium | Blood |
| Monocytes | Sodium | Leukocyte esterase |
| Neutrophils 🛇 | Glucose | Nitrite |
| Hematocrit | BUN | Urine dipstick for pregnancy testing <sup>b</sup> |
| Hemoglobin | Creatinine | Urine drug screen <sup>c</sup> |
| MCH | ALP | |
| MCHC | AST | |
| MCV | ALT | |
| Platelet count | GGT | |

<sup>&</sup>lt;sup>a</sup> A urine microscopic examination will be performed if the result for albumin (protein), leukocyte esterase, blood or nitrite is abnormal. A urine microscopic examination will include: WBC, RBC, epithelial cells (squamous, transitional and renal tubular), hyaline casts, WBC casts, RBC casts, waxy casts, granular casts, calcium oxalate crystals, uric acid crystals, triphosphate crystals, yeast, bacteria, amorphous urates, and amorphous phosphates.

b Pregnancy testing will consist of serum testing at the Screening. The pregnancy test will be urine at all other visits.

| Hematology | Chemistry | Urinalysis dipstick <sup>a</sup> |
|---|---|---|
| RBC count | Total bilirubin | |
| WBC count | LDH | |
| | Serum pregnancy testing <sup>b</sup> | |

ALP=alkaline phosphatase; ALT=alanine aminotransferase; AST=aspartate aminotransferase; BUN=blood urea nitrogen; ; GGT=gamma glutamyltransferase; LDH=lactate dehydrogenase; MCH=mean corpuscular hemoglobin; MCHC=mean corpuscular hemoglobin concentration; MCV=mean corpuscular volume; **PEOT=Premature End of Treatment;** RBC=red blood cell; WBC=white blood cell

#### Change #46

# Section 12.3.1 Assessment and management of TB and TB risk factors, Item d

d. Current or history of NTMB infection despite prior or current therapy.

## Has been changed to:

d. NTMB infection is defined as a clinical infection caused by mycobacterial species other than those belonging to the Mycobacterium tuberculosis complex<del>Current or history of NTMB infection despite prior or current therapy</del>.

#### Change #47

# Section 12.3.1.1 Tuberculosis assessment by IGRA

During conduct of the study, the TB assessment by IGRA (QuantiFERON TB GOLD is recommended) will be performed as described in Table 5-1 for all subjects. The test results will be reported as positive, negative, or indeterminate. Positive TB test results must be reported as an adverse event and appropriately updated once the final diagnosis is known (e.g. active TB, latent TB, or false positive TB test). UCB also recommends that a TB specialist be consulted where TB (latent or active) is suspected or if there are doubts regarding test results. If latent or active TB is identified, subject must undergo appropriate study-specified withdrawal procedures. The retest during Screening must be done during the protocol-defined Screening window.

# Has been changed to:

During conduct of the study, the TB assessment by IGRA (QuantiFERON TB GOLD is recommended) will be performed as described in Table 5-1 for all subjects. The test results will be reported as positive, negative, or indeterminate. Positive **and indeterminate** TB test results must be reported as an adverse event and appropriately updated once the final diagnosis is known (eg, active TB, latent TB, or false positive TB test). UCB also recommends that a TB specialist be consulted where TB (latent or active) is suspected or if there are doubts regarding



<sup>&</sup>lt;sup>a</sup> A urine microscopic examination will be performed if the result for albumin (protein), leukocyte esterase, blood or nitrite is abnormal. A urine microscopic examination will include: WBC, RBC, epithelial cells (squamous, transitional and renal tubular), hyaline casts, WBC casts, RBC casts, waxy casts, granular casts, calcium oxalate crystals, uric acid crystals, triphosphate crystals, yeast, bacteria, amorphous urates, and amorphous phosphates.

b Pregnancy testing will consist of serum testing at the Screening **Visit**. The pregnancy test will be urine at all other visits.

<sup>&</sup>lt;sup>c</sup> Urine drug screen will be performed at Screening Visit and PEOT Visit.
test results. If latent or active TB is identified, subject must undergo appropriate study-specified withdrawal procedures. The retest during Screening must be done during the protocol-defined Screening window.

### Change #48

#### Section 14.1 Definition of analysis sets

#### The following paragraph has been deleted:

The Maintenance Set (MS) will consist of all subjects who receive at least 1 dose of bimekizumab treatment at Week 24 or later.

#### Change #49

Figure 14-1: Sequence of testing





Note: all calculations above are based on the combined Bimekizumab arms with the sample size of 300.

Section 14.3.1.1 Sensitivity analyses In order to obtain reasonal.1

Will be Section 14.3.1.1 Sensitivity analyses

In order to obtain reasonable estimates of variability at a given center, a minimum of 10 subjects will be considered acceptable for a center to be included in the model without pooling. Given the 1:1 randomization allocation scheme, this should provide a minimum of about 5 subjects the bimekizumab arm and 5 subjects in the adalimumab arm. Centers with fewer than 10 subjects will be eligible for pooling,

The following center pooling algorithm will be used for each geographic region:

- If a center has 10 or more subjects, then no pooling will be done for that center.
- Centers with fewer than 10 subjects will be ordered from largest to smallest with pooling proceeding in the following manner:
  - Two or more centers will be combined until the cumulative subject total is at least 10.

Once a pooled center has at least 10 subjects, the process will continue in an iterative fashion for the subsequent centers in the ordered list, where a new pooled center begins each time at least 10 subjects has been reached in the previous pool.

If this iterative process reaches the end of the ordered list of centers where the final pooled center has fewer than 10 subjects, then the subjects from the centers in that pool will be combined with the pooled center formed in the previous iteration.


In order to obtain reasonable estimates of variability at a given center, a minimum of 150 subjects will be considered acceptable for a center to be included in the model without pooling. Given the 1:1:1-randomization allocation scheme, this should provide a minimum of about 5 subjects the bimekizumab Q4W arm, 5 subjects in the bimekizumab Q4W/Q8W arm, and 5 subjects in the adalimumab arm. Centers with fewer than 150 subjects will be eligible for pooling.

The following center pooling algorithm will be used for each geographic region:

- If a center has 150 or more subjects, then no pooling will be done for that center.
- Centers with fewer than 150 subjects will be ordered from largest to smallest with pooling proceeding in the following manner:
  - Two or more centers will be combined until the cumulative subject total is at least 150.
  - Once a pooled center has at least 150 subjects, the process will continue in an iterative fashion for the subsequent centers in the ordered list, where a new pooled center begins each time at least 150 subjects has been reached in the previous pool.
  - If this iterative process reaches the end of the ordered list of centers where the final pooled center has fewer than 150 subjects, then the subjects from the centers in that pool will be combined with the pooled center formed in the previous iteration.

### Change #51

#### Section 14.3.2.1.1 Initial Treatment Period

The secondary efficacy variables for time points during the Initial Treatment Period will be analyzed for all subjects in the RS.

For binary secondary efficacy variables, the stratified CMH test as specified for the primary analysis will be implemented to test for superiority of bimekizumab to adalimumab. As in the primary analysis, NRI will be used to account for missing data.

#### Has been changed to:

The secondary efficacy variables for time points during the Initial Treatment Period will be analyzed for all subjects in the RS.

### For comparisons with adalimumab at Week 16, the 2 bimekizumab arms will be pooled.

For binary secondary efficacy variables, the stratified CMH test as specified for the primary analysis will be implemented to test for superiority of bimekizumab to adalimumab. As in the primary analysis, NRI will be used to account for missing data.

#### Change #52

#### Section 14.3.2.1.2 Maintenance Treatment Period

The only secondary efficacy variables in the Maintenance Treatment Period are PASI90 and IGA at Week 56.

Since all subjects on adalimumab will be switched to bimekizumab at Week 24, the assessment of PASI90 and IGA at Week 56 will be for bimekizumab at the Q4W and Q8W dosing intervals. These summaries will include descriptive statistics by bimekizumab dose regimen for the percentage of responders at Week 56 based on the MS. The summary of PASI90 at Week 56 will be based on subjects who were PASI90 responders at Week 24 (similarly, the summary of IGA responders at Week 56 will be based on Week 24 IGA responders). Subjects with missing data at Week 56 or who discontinue study treatment prior to Week 56 will be imputed via NRI.

#### Has been changed to:

The only secondary efficacy variables in the Maintenance Treatment Period includeare PA\$190. PASI100, and IGA at Week 24 and Week 56.

Since all subjects on adalimumab will be switched to bimekizumab at Week 24, the assessment of PASI90 and IGA at Week 56 will be for bimekizumab at the Q4W and Q8W dosing intervals. These summaries will include descriptive statistics by bimekizumab dose regimens for the percentage of responders at Week 24 and Week 56 based on the MRS. The summary of PASI90 at Week 56 will be based on subjects who were PASI90 responders at Week 24 (similarly, the summary of IGA responders at Week 56 will be based on Week 24 IGA responders). Subjects with missing data at Week 56 or who discontinue study treatment prior to Week 56 will be imputed via NRI.

#### Change #53

# Section 14.3.2.2 Analysis of other efficacy variables

The other efficacy variables in the Initial Treatment Period will be analyzed for all subjects in the RS. For the Maintenance Treatment Period summaries will be based on the MS.

### Has been changed to:

The other efficacy variables in the Initial Treatment Period will be analyzed for all subjects in the RS. For the Maintenance Treatment Period, summaries will be based on the MS.

#### Change #54

#### Section 14.5.1 Safety analyses

Safety variables will be analyzed for all subjects in the SS. Additional summaries focusing on safety during the Maintenance Treatment Period will also be prepared and will be based on the MS.

Adverse events will be coded according to the Medical Dictionary for Regulatory Activities (MedDRA). Adverse events will be summarized descriptively by treatment group, primary system organ class, High Level Term (HLT), and preferred term. Additional tables will summarize AEs by intensity and relationship to IMP, AEs leading to withdrawal from the study, SAEs, and deaths. Adverse Events of Special Monitoring will be summarized and will be described in greater detail in the SAP.

#### Has been changed to:

Safety variables will be analyzed for all subjects in the SS. Additional summaries focusing on safety during the Maintenance Treatment Period will also be prepared and will be based on the MRS.

Adverse events will be coded according to the Medical Dictionary for Regulatory Activities (MedDRA). Adverse events will be summarized descriptively by treatment group, primary system organ class, High Level Term (HLT), and preferred term. Additional tables will summarize AEs by intensity and relationship to IMP, AEs leading to withdrawal from the study, SAEs, and deaths. Adverse Events of Special Monitoring Specific safety topics of interest will be summarized and will be described in greater detail in the SAP.

#### Change #55

#### Section 14.7 Handling of dropouts or missing data

For the secondary endpoints evaluated at Week 56 (based on the MS), all subjects with missing data at Week 56 or who discontinue study treatment prior to Week 56 will be counted as nonresponders.

### Has been changed to:

For the secondary endpoints evaluated at Week 56 (based on the MRS), all subjects with missing data at Week 56 or who discontinue study treatment prior to Week 56 will be counted as

nonresponders.

Change #56

Section 14.9 Determination of sample size

A total of 400 subjects will be randomly assigned in a 7:1 ratio to the following treatment groups: groups:

- Bimekizumab 320mg (200 subjects)
- Adalimumab (200 subjects)

When comparing bimekizumab to adalimumab, the assumed responder rates for PASI90 and IGA at Week 16 for the bimekizumab group are 75% and 85%, respectively. These estimates are based on the results of the Phase 2b PS0010 study. The PASI90 responder rates at Week 16 for adalimumab from the VOYAGE-1 and VOYAGE-2 studies were 50% and 47%, respectively (Blauvelt et al, 2017; Reich et al, 2017). Additionally, the IGA responder rates at Week 16 for adalimumab in VOYAGE-1 and VOYAGE-2 were 66% and 68%, respectively. For the purposes of these sample size calculations at Week 16, we assume a PASI90 responder rate and IGA responder rate for adalimumab of 50% and 68%, respectively.

The testing procedure described in Section 14.3 indicates that the first test will be to demonstrate noninferiority to adalimumab for the co-primary variables of PASI90 and IGA at Week 16. If non-inferiority for both tests is demonstrated, then superiority to adalimumab will be tested.

Because the superiority evaluation is the more stringent test, sample size calculations are based on the testing of superiority to adalimumab for PASI90 and IGA at Week 16. Given these assumptions and a sample size of 200 subjects per treatment group, the power to detect a statistically significant difference between bimekizumab and adalimumab is >99% for PASI90 and 97% for IGA. This assumes a 2-sided significance level of 0.05. Because both co-primary endpoints are highly powered independently, and because PASI and IGA response tend to be

highly correlated, the overall power for achieving superiority on both co-primary endpoints is not calculated here as it is similar to the lower of the individual tests.

A total of 450400 subjects will be randomly assigned in a 1:1:1 ratio to the following treatment groups:

Bimekizumab 320mg Q4W/O8W/ "
bimekizumab 320mg Q4W/O8W/ "
bimekizumab 320mg Q4W/O8W/ " Note that the non-inferiority testing procedure will be based on a 1-sided significance level of

- Adalimumab 80mg administered as an initial dose, followed by 40mg Q2W starting 1 week after the initial dose (ie, adalimumab will be administered according to the labeling recommendations) until Week 24, then bimekizumab 320mg Q4W from Week 24 to Week 52 (150200 subjects)

When comparing bimekizumab to adalimumab, the assumed responder rates for PASI90 and IGA at Week 16 for the bimekizumab group are 75% and 85%, respectively. These estimates are based on the results of the Phase 2b PS0010 study. The PASI90 responder rates at Week 16 for adalimumab from the VOYAGE-1 and VOYAGE-2 studies were 50% and 47%, respectively (Blauvelt et al. 2017; Reich et al. 2017). Additionally, the IGA responder rates at Week 16 for adalimumab in VOYAGE-1 and VOYAGE-2 were 66% and 68%, respectively. For the purposes of these sample size calculations at Week 16, we assume a PASI90 responder rate and IGA responder rate for adalimumab of 50% and 68%, respectively.

The testing procedure described in Section 14.3 indicates that the first test will be to demonstrate noninferiority to adalimumab for the co-primary variables of PASI90 and IGA at Week 16. If non-inferiority for both tests is demonstrated, then superiority to adalimumab will be tested.

Because the superiority evaluation is the more stringent test, sample size calculations are based on the testing of superiority to adalimumab for PASI90 and IGA at Week 16. Given these assumptions and a sample size of 150200 subjects per treatment group in the adalimumab arm and 300 subjects in the pooled bimekizumab arms, the power to detect a statistically significant difference between bimekizumab and adalimumab is >99% for PASI90 response and 97% for IGA response. This assumes a 2-sided significance level of 0.05. Because both coprimary endpoints are highly powered independently, and because PASI and IGA response tend to be highly correlated, the overall power for achieving superiority on both co-primary endpoints is not calculated here as it is similar to the lower of the individual tests.

Note that the non-inferiority testing procedure will be based on a 1-sided significance level of 0.025 and a non-inferiority margin of 10%. The power to demonstrate non-inferiority to adalimumab using the other assumptions described above is >99% for both PASI90 and IGA responses.

#### Change #57

#### **Section 17 REFERENCES**

### The following references have been deleted from the list:

Blauvelt A, et al. Level of efficacy and safety of guselkumab, an anti-interleukin-23 monoclonal antibody, compared with adalimumab for the continuous treatment of moderate-to-severe psoriasis in the phase 3 VOYAGE 1 trial. Annual European Academy of Dermatology and Venereology (EADV 2016); 28 Sept-02 Oct, 2016; Vienna, Austria; VIE16LAT-0080.

Bretz F, Maurer W, Brannath W, Posch M. A graphical approach to sequentially rejective multiple test procedure. Statistics in Medicine. 2009;28:586-604.

Dauden E, Griffiths CE, Ortonne JP, Kragballe K, Molta CT, Robertson D, et al. Improvements in patient-reported outcomes in moderate-to-severe psoriasis patients receiving continuous or paused etanercept treatment over 54 weeks: the CRYSTEL study. J Eur Acad Dermatol Venereol. 2009;23(12):1374-82.

International Menopause Society. Cornwall, UK: Menopause Terminology; 2015. http://www.imsociety.org/menopause\_terminology.php. Accessed 05 Dec 2016.

Langley RG, Feldman SR, Han C, Schenkel B, Szapary P, Hsu MC, et al. Ustekinumab significantly improves symptoms of anxiety, depression, and skin-related quality of life in patients with moderate-to-severe psoriasis: Results from a randomized, doubleblind, placebo-controlled phase III trial. J Am Acad Dermatol. 2010;63(3):457-65.

Menter A, Tyring SK, Gordon K, Kimball AB, Leonardi CL, Langley RG, et al. Adalimumab therapy for moderate to severe psoriasis: A randomized, controlled phase III trial. J Am Acad Dermatol 2008;58:106-15.

Saurat JH, Stingl G, Dubertret L, Papp K, Langley RG, Ortonne JP, et al. Efficacy and safety results from the randomized controlled comparative study of adalimumab vs. methotrexate vs. placebo in patients with psoriasis (CHAMPION). Brit J Dermatol. 2008;158:558–66.

### 18.2 Protocol Amendment 2

### Rationale for the amendment

The purpose of this amendment was the following:

- Extend the duration of the Screening Period, and therefore the overall study duration, by 1 week
- Update list of current treatment for PSO to reflect changes in labeling and approved countries
- Update list of completed and ongoing bimekizumab studies to reflect completion of study UP0042
- Clarify calculation of PASI responder rates

Remove references to PD assessments as they will not be conducted in this study

• Update Schedule of study assessments to include a hematology and biochemistry sample at Week 28, and to modify the visits at which the TB questionnaire, body weight, physical examination, and ECG are assessed

- Clarify that all visits from first dose to Week 24 would have a  $\pm 3$  day visit window, while all visits from Week 28 to end of study would have a ±7 day window

- Modify exclusion criteria pertaining to history of malignancy, systemic disease, and major depression

  Add new withdrawal criteria for nonresponders and for subject.

  Clarify withdrawal criteria for out.

- Correct information pertaining to how adalimumab is supplied
- Update prohibited concomitant medications to include tildrakizumab and risankizumab
- Corrected discrepancies between Section 8 Study procedures by visit and Table 5-1 Schedule of study assessments Updated laboratory measurements to be performed.

  Provide additional details for requirements.

  Defined a BK7 c

- Provide additional details for requirements for IMP rechallenge in the event of PDILI
- Clarify regions for analyses
- Update the sequence testing and analysis of secondary efficacy variables

In addition, minor spelling, editorial, and formatting changes were made, and the List of abbreviations was updated.

#### Change #1

### Section 1 Summary second and third paragraphs

The study population consists of adult subjects (≥18 years of age) with a diagnosis of moderate to severe chronic plaque PSO (Baseline Psoriasis Area and Severity Index [PASI] > 12 and body surface area [BSA] affected by PSO ≥10% and Investigator's Global Assessment [IGA] score ≥3 [on a 5-point scale]) who are candidates for adalimumab or for systemic PSO therapy and/or phototherapy and/or photochemotherapy.

Approximately 600 subjects will be screened in order to have a total of 450 subjects randomized in the study. For each subject, the study will last a maximum of 76 weeks and will consist of 4 periods, a Screening Period (2 to 4 weeks), a double-blind, active comparator-controlled Initial Treatment Period (16 weeks), a dose-blind Maintenance Treatment Period (40 weeks), and a Safety Follow-Up (SFU) Period (20 weeks after the last dose of the investigational medicinal product [IMP]).

The study population consists of adult subjects (≥18 years of age) with a diagnosis of moderate to severe chronic plaque PSO (Baseline Psoriasis Area and Severity Index [PASI] ≥12 and body

Approximately 600 subjects will be screened in order to have a total of 450 subjects randomized in the study. For each subject, the study will last a maximum of 76-77 weeks and will consist of 4 periods, a Screening Period (2 to 4-5 weeks), a double-blind active a Safety Follow II. a Safety Follow-Up (SFU) Period (20 weeks after the last final dose of the investigational id any exter medicinal product [IMP]).

### Change #2

### Section 2.1.2 Current treatments for psoriasis, 1st paragraph

Therapy for patients with PSO varies according to the severity of disease. Limited or mild disease is often treated with topical therapies such as corticosteroids and vitamin D analogs. Patients with more severe disease are often treated with photochemotherapy, methotrexate, cyclosporine, the oral phosphodiesterase 4 (PDE4) inhibitor apremilast, or biologic agents, such as tumor necrosis factor (TNF) antagonists, interleukin (IL)-12/23 inhibitors, IL-23p19 inhibitors and IL-17A inhibitors. The effectiveness of TNF inhibitors in the treatment of PSO has been demonstrated in many Phase 3 clinical studies and has led to the approval of multiple TNF inhibitors for use in patients with moderate to severe PSO. Interleukin inhibitors approved for this indication include the IL-12/23 antagonist ustekinumab, the IL-23p19 antagonist guselkumab (in the US only) the IL-17A inhibitors secukinumab and ixekizumab, and the IL-17 receptor antagonist brodalumab.

### Has been changed to:

Therapy for patients with PSO varies according to the severity of disease. Limited or mild disease is often treated with topical therapies such as corticosteroids and vitamin D analogs. Patients with more severe disease are often treated with photochemotherapy phototherapy, methotrexate, cyclosporine, the oral phosphodiesterase 4 (PDE4) inhibitor apremilast, or biologic agents, such as tumor necrosis factor (TNF) antagonists, interleukin (IL)-12/23 inhibitors, IL-23p19 inhibitors and IL-17A inhibitors. The effectiveness of TNF inhibitors in the treatment of PSO has been demonstrated in many Phase 3 clinical studies and has led to the approval of multiple TNF inhibitors for use in patients with moderate to severe PSO. Interleukin inhibitors approved for this indication include the IL-12/23 antagonist ustekinumab, the IL-23p19 antagonist guselkumab (in the US only), the IL-17A inhibitors secukinumab and ixekizumab, Change #3
Section and the IL-17 receptor antagonist brodalumab.

#### Section 2.1.2 Current treatments for psoriasis, third bullet

Chemophototherapy is a frequent option for moderate to severe patients, but the inconvenience of multiple treatment visits and varying efficacy limits its use in the market.

**Phototherapy** is a frequent option for moderate to severe patients, but the inconvenience of multiple treatment visits and varying efficacy limits its use in the market.

### Change #4

### Section 2.1.2 Current treatments for psoriasis, last bullet, second and fourth sub-bullets

- Ustekinumab has been approved in the US and the EU for the treatment of adult patients with moderate to severe plaque PSO who are candidates for phototherapy or systemic therapy. Ustekinumab is a human immunoglobulin (Ig) G1k monoclonal antibody that binds with specificity to the p40 protein subunit used by both the IL-12 and IL-23 cytokines, naturally occurring cytokines that are involved in inflammatory and immune responses, such as natural killer cell activation and CD4+ T-cell differentiation and activation.
- Guselkumab has been approved in the US for the treatment of adult patients with moderate to severe plaque PSO who are candidates for systemic therapy or phototherapy. It is a human monoclonal IgG1 $\lambda$  antibody that selectively binds to the p19 subunit of interleukin 23 (IL-23) and inhibits its interaction with the IL-23 receptor. IL-23 is a naturally occurring cytokine that is involved in normal inflammatory and immune responses. Guselkumab inhibits the release of proinflammatory cytokines and chemokines.

### Has been changed to:

- chemokines.

  s been changed to:

  Ustekinumab has been approved in the US and the EU for the treatment of adult patients with moderate to severe plaque PSO who are candidates for phototherapy or systemic therapy. Ustekinumab is a human immunoglobulin (Ig) G1k monoclonal antibody that binds with specificity to the p40 protein subunit used by both the IL-12 and IL-23 cytokines, naturally occurring cytokines that are involved in inflammatory and immune responses, such as natural killer cell activation and CD4+ T-cell differentiation and activation.
- Guselkumab has been approved in the US and the EU for the treatment of adult patients with moderate to severe plaque PSO who are candidates for systemic therapy or phototherapy. It is a human monoclonal IgG1λ antibody that selectively binds to the p19 subunit of interleukin 23 (IL-23) and inhibits its interaction with the IL-23 receptor. IL-23 is a naturally occurring cytokine that is involved in normal inflammatory and immune responses. Guselkumab inhibits the release of proinflammatory cytokines and chemokines.

Section 2.2.1.1 Completed studies
Four clinical et al. Four clinical studies of bimekizumab have been completed: UP0008 in 39 subjects with mild to moderate plaque PSO, RA0124 in 30 healthy volunteers, PA0007 in 53 subjects with PsA, and UP0031 in 12 healthy volunteers.

Four Five clinical studies of bimekizumab have been completed: UP0008 in 39 subjects with mild to moderate plaque PSO, RA0124 in 30 healthy volunteers, PA0007 in 53 subjects with PsA, and UP0031 in 12 healthy volunteers, and UP0042 in 48 healthy volunteers.

### And the following paragraph has been added:

UP0042 was a randomized double-blind, placebo-controlled, single-dose, parallel-group study to evaluate the safety, tolerability, and pharmacokinetics of bimekizumab administered as subcutaneous injection to Japanese and Caucasian healthy subjects. This study demonstrated that the PK profiles following single administration of 80mg, 160mg, and 320mg with sc injection were dose proportional with a linear elimination in both Japanese and Caucasian subjects and that the PK profiles of Japanese and Caucasian subjects were considered to be generally similar. A single dose of bimekizumab (80mg, 160mg, or 320mg) administered as sc injection was generally safe and well tolerated in healthy Japanese and Caucasian subjects and no major differences in safety findings were observed between Japanese and Caucasian subjects.

#### Change #6

### **Section 2.2.1.2 Ongoing studies**

Four additional studies of bimekizumab in the treatment of PSO and 1 study in healthy volunteers are ongoing.

- PS0010 is a Phase 2b, double-blind, placebo-controlled, dose ranging study to evaluate the safety, efficacy, PK, and pharmacodynamics (PD) of bimekizumab in adult subjects with moderate to severe chronic plaque PSO.
- PS0011 is a long-term extension study for subjects who completed PS0010 to assess the long-term safety, tolerability, and efficacy of bimekizumab.
- PS0016 is a Phase 2a, subject-blind, Investigator-blind study to evaluate the time course of PD response, safety, and PK of bimekizumab in adult subjects with moderate to severe chronic plaque PSO.
- PS0018 is a long-term extension study for eligible subjects from PS0016 to assess the safety, tolerability, and efficacy of bimekizumab.
- UP0042 is a Phase 1 study designed to evaluate the safety, tolerability, and PK of bimekizumab administered as an sc injection of 80mg, 160mg, or 320mg to Japanese and Caucasian healthy subjects.

# Has been changed to:

Four additional studies of bimekizumab in the treatment of PSO and 1 study in healthy volunteers are ongoing.

• PS0010 is a Phase 2b, double-blind, placebo-controlled, dose ranging study to evaluate the safety, efficacy, PK, and pharmacodynamics (PD) of bimekizumab in adult subjects with moderate to severe chronic plaque PSO.

- PS0011 is a long-term extension study for subjects who completed PS0010 to assess the long-term safety, tolerability, and efficacy of bimekizumab.
- PS0016 is a Phase 2a, subject-blind, Investigator-blind study to evaluate the time course of PD response, safety, and PK of bimekizumab in adult subjects with moderate to severe chronic plaque PSO.
- PS0018 is a long-term extension study for eligible subjects from PS0016 to assess the safety, tolerability, and efficacy of bimekizumab.
- UP0042 is a Phase 1 study designed to evaluate the safety, tolerability, and PK of bimekizumab administered as an sc injection of 80mg, 160mg, or 320mg to Japanese and Caucasian healthy subjects.

Section 4.3 Other variables

The following text has been added:

The other variables are listed below and will be evaluated according to the planned assessments Table 5-1.

Change #8

Section 4.3.1 Other efficacy variables, last sentence in second paragraph

Note that PASI responder rates will always be calculated relative to the Baseline (first dose) Visit.

Has been changed to:

Note that Unless otherwise stated PASI responder rates will always be calculated relative to the Baseline (first dose) Visit.

Change #9

Section 4.4 Pharmacokinetic variable

Section 4.5 Pharmacogenomic variables

Section 4.6 Immunological variable

Have been changed to:

Section 4.4 4.3.3 Pharmacokinetic variable

Section 4.5 4.3.4 Pharmacogenomic variables

Section 4.6 4.3.5 Immunological variable

Section 5.1 Study description
PS0008 is a Pi PS0008 is a Phase 3, multicenter study consisting of a 16-week, randomized, double-blind, parallel-group, active-comparator-controlled Initial Treatment Period followed by a 40-week, Maintenance Treatment Period to evaluate the efficacy and safety of bimekizumab in adult subjects with moderate to severe chronic plaque PSO. To be eligible to participate in this study. subjects must be adults with a diagnosis of moderate to severe PSO (Baseline PASI ≥12 and BSA affected by PSO  $\geq$ 10% and IGA score  $\geq$ 3 [on a 5-point scale]) who are candidates for systemic PSO therapy and/or phototherapy and/or photochemotherapy. Adalimumab will be

rS0008 is a Phase 3, multicenter study consisting of a 16-week, randomized, double-blind, parallel-group, active-comparator-controlled Initial Treatment Period followed by a 40-week, Maintenance Treatment Period to evaluate the efficacy and safety of bimekizumab in adultation subjects with moderate to severe chronic plaque PSO. To be eligible to post subjects must be adults with a diagnosis of moderate to systemic PSO > 10% and IC systemic PSO therapy and/or phototherapy and/or photoehemotherapy. Adalimumab will be administered per the local label. Up to 30% of subjects may have been previously exposed to a biologic therapy (see Exclusion Criterion #23, Section 6.2).

### Change #11

#### Section 5.2 Study periods

This study will include 4 periods, a Screening Period (2 to 4 weeks), an Initial Treatment Period (16 weeks), a Maintenance Treatment Period (40 weeks), and a SFU Period (20 weeks after the last dose of IMP).

### Has been changed to:

This study will include 4 periods, a Screening Period (2 to 4-5 weeks), an Initial Treatment Period (16 weeks), a Maintenance Treatment Period (40 weeks), and a SFU Period (20 weeks after the **last final** dose of IMP).

Section 5.2.1 Screening Period The Screening Period will last 2 weeks, but can be extended up to a total of 4 weeks.

# Has been changed to:

The Screening Period will last 2 weeks, but can be extended up to a total of 4-5 weeks in cases where a laboratory assessment needs to be repeated or to allow washout of prohibited medications. This document cannot be

### Section 5.3 Study duration per subject

For each subject, the study will last a maximum of up to 76 weeks, as follows:

• Screening Period: 2 to 4 weeks

### Has been changed to:

For each subject, the study will last a maximum of up to <del>76-</del>77 weeks, as follows:

• Screening Period: 2 to 4-5 weeks

### Change #14

#### Section 5.5 Anticipated regions and countries

• The regions planned for study conduct are Europe, Canada, and the US, with possible extension to other regions and countries.

### Has been changed to:

The regions planned for study conduct are **North America**, **Western** Europe, **Canada**, and the US Central/Eastern Europe, and Asia/Australia, with possible extension to other regions and countries.

#### Change #15

### Section 5.6 Schedule of study assessments

The schedule of study assessments for all subjects enrolled in the study is presented in Table 5-1.

#### Has been changed to:

The schedule of study assessments for all subjects enrolled in the study is presented in Table 5-1. At each visit, all study assessments should be performed prior to administration of IMP.



Table 5-1: Schedule of study assessments

| Table 5-1: | Sch | edul | le of | stud | y ass | sessi | ment | S | | | | | | | | | | | | aiiaii | ) S | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit <sup>a</sup> /<br>Week | Screening | | | Doub | | | al Trea<br>er first | | Period | | | | I | Dose-bli | nd Ma<br>(wee | intena<br>ks afte | ance T | reatn | nent P | | | | W56/PEOT | SFIIb |
| Protocol activity | | Baseline<br>(first dose) | 1 | 3 | 4 | 5,<br>7 | 8 | 9,<br>11 | 12 | 13,<br>15 | 16 | 17,<br>19 | 20 | 21, 23 | 242 | 28 | 32 | 36 | 40 | 44 | 48 | 52 | 56 | |
| Informed consent <sup>c</sup> | X | | | | | | | | | | | | | tion | | | | | | | | X <sup>d</sup> | | |
| Inclusion/exclusion | X | X | | | | | | | | | | | olic | ,0 | | | | | | | | | | |
| Urine drug screen | X | | | | | | | | | | ر م | ? | 36, | | | | | | | | | | X | |
| Demographic data | X | | | | | | | | | /< | ) 1 | ijo, | | | | | | | | | | | | |
| Psoriasis history | X | | | | | | | | | $\mathcal{C}^{\vee}$ | Oil | | | | | | | | | | | | | |
| Significant past<br>medical history and<br>concomitant<br>diseases | X | Xe | | | | | | < | ZEDP<br>Zejir | O all | | | | | | | | | | | | | | |
| Physical examination <sup>f,g</sup> | X | | | | | | | 1/1/8 | X | | X | | | | X | | | X | | | X | | X | X |
| Height | | X | | | | | X | | | | | | | | | | | | | | | | | |
| Body weight | | X | | | | 5 | 30/ | | | | X | | | | X | | | X | | | X | | X | |
| Vital signs <sup>h</sup> | X | X | X | X | X | \$ | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Hematology and biochemistry | X | X | X | X | X) | | X | | X | | X | | X | | X | | X | | X | | X | | X | X |
| Urinalysis | X | X | | OS, | | | | | | | X | | | | X | | X | | X | | X | | X | X |
| ECG | X | | | ~ | | | | | | | X | | | | X | | | X | | | X | | X | |
| Pregnancy testing <sup>1</sup> Confidential | X | XC | 31, | | X | | X | | X | | X | | X | | X | X | X | X | X | X | X | X | X | X |

Table 5-1: Schedule of study assessments

| UCB<br>Clinical Study Prot | ocol | [ | | | | | | | I | Bimeki | zumab | | | | | | | | | | , S | 062 | Apr 20<br>PS00 | )18 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Table 5-1: | Sch | edu | le of | stud | y ass | sessr | nent | S | | | | | | | | | | | . ( | ailail | ,<br>, | | | |
| Visit <sup>a</sup> /<br>Week | Screening | | | Doul | ble-blin<br>(wee | d Initia | | | Period | | | | ] | Dose-bli | | aintena<br>eks aft | | reatn | o`<br>ient P | | | | W56/PEOT | $\mathbf{SFU}^{\mathrm{b}}$ |
| Protocol activity | | Baseline<br>(first dose) | 1 | 3 | 4 | 5,<br>7 | 8 | 9,<br>11 | 12 | 13,<br>15 | 16 | 17,<br>19 | 20 | 21, 23 | 247 | 28 | 32 | 36 | 40 | 44 | 48 | 52 | 56 | |
| Hepatitis B and C testing <sup>j</sup> | X | | | | | | | | | | | | | dion | | | | | | | | | | |
| HIV testing <sup>k</sup> | X | | | | | | | | | | | 7 | 66/1 | | | | | | | | | | | |
| Chest x-ray <sup>l</sup> | X | | | | | | | | | | 0 | 100 | | | | | | | | | | | | |
| IGRA Tuberculosis<br>test | X | | | | | | | | | | 01/12 | | | | | | | | | | | X | | |
| Tuberculosis<br>questionnaire | X | X | | | | | | | EDP | ali | X | | | | X | | | X | | X | | X | X | X |
| Blood sample for<br>bimekizumab<br>plasma<br>concentrations <sup>m</sup> | | X | X | X | X | | X | 100 | X | | X | | X | | X | | | X | | | X | | X | X |
| Blood sample for<br>anti-bimekizumab<br>antibodies <sup>m</sup> | | X | | | X | • | X | 7 | X | | X | | X | | X | | | X | | | X | | X | X |
| Blood sample<br>genomic,<br>proteomic, and<br>metabolomics, and<br>candidate<br>biomarker<br>analyses <sup>c,m</sup> | | X | X | LOC V | sedic | SUR | X | | X | | X | | | | | | | | | | | | X | |

Table 5-1: Schedule of study assessments

| Clinical Study Prot Table 5-1: | | | lo of | otud | | | mont | | | 31meki | zumab | | | | | | | | | اند | 37S | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit <sup>a</sup> / Week | Screening | | ie oi | | y ass | | ıl Trea | tment | Period | | | | 1 | Dose-bli | nd Ma<br>(wee | nintena<br>eks aft | ance T | reatn | nent P | | | | W56/PEOT | SFUb |
| Protocol activity | | Baseline<br>(first dose) | 1 | 3 | 4 | 5,<br>7 | 8 | 9,<br>11 | 12 | 13,<br>15 | 16 | 17,<br>19 | 20 | 21, 23 | 242 | 28 | 32 | 36 | 40 | 44 | 48 | 52 | 56 | |
| Blood sample<br>genetic/epigenetic<br>analyses <sup>c,m</sup> | | X | | | | | | | | | | _1 | dic | dilon | | | | | | | | | X | |
| PASI | X | X | X | X | X | | X | | X | | X | | X | | X | X | X | X | X | X | X | X | X | X |
| IGA | X | X | X | X | X | | X | | X | | X | ijor | X | | X | X | X | X | X | X | X | X | X | X |
| Percentage of BSA | X | X | X | X | X | | X | | X | | XIV | | X | | X | X | X | X | X | X | X | X | X | X |
| DLQI | | X | X | X | X | | X | | X | | Χ | | X | | X | | X | | X | | X | | X | |
| PHQ-9 | X | X | | | X | | X | < | X | (9) | X | | X | | X | X | X | X | X | X | X | X | X | |
| eC-SSRS | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Patient Symptom<br>Diary (daily) | X | X | X | X | X | X | X | X,C | X | X | X | X | X | X | X | | | | | | | | | |
| scalp IGA | | X | Xn | Xn | Xn | | Xa. | | Xn | | Xn | | Xn | | Xn | | X <sup>n</sup> | | Xn | | Xn | | Xn | |
| mNAPSI | | X | | | Xº | JIP | Xº | | Xº | | Xº | | Xº | | Xº | | Xº | | Xº | | Xº | | Xº | |
| pp-IGA | | X | | | Xp | ) | X <sup>p</sup> | | Xp | | X <sup>p</sup> | | Xp | | X <sup>p</sup> | | X <sup>p</sup> | | Xp | | X <sup>p</sup> | | Xp | |
| EQ-5D-3L | | X | | | X | | X | | X | | X | | | | X | | | | X | | | | X | |
| SF-36 | | X | | be | X | _ | X | | X | | X | | | | X | | | | X | | | | X | |
| Patient global<br>assessment of<br>psoriasis <sup>q</sup> | | | anno | | | | | | | | | | | | X | | X | | X | | X | | X | |

Table 5-1: Schedule of study assessments

| Visit <sup>a</sup> /<br>Week | Screening | | | Dou | ble-blir<br>(we | ıd Initi<br>eks afte | | | Period | | | | I | Oose-blii | | | | Treatn | | eriod | | | W56/PEOT | $\mathbf{SFU}^{\mathrm{b}}$ |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Protocol activity | | Baseline<br>(first dose) | 1 | 3 | 4 | 5,<br>7 | 8 | 9,<br>11 | 12 | 13,<br>15 | 16 | 17,<br>19 | 20 | 21,<br>23 | 242 | 28 | 32 | 36 | 40 | 44 | 48 | 52 | 56 | |
| PASE | | X | | | | | | | | | | | | ijon | | | | | | | | | X | |
| PGADA <sup>r</sup> | | X | | | X | | | | X | | X | 1 | -Olic | 0 | X | | X | | X | | X | | X | |
| WPAI-SHP V2.0 | | X | | | | | | | | | XO | | 16, | | X | | | | X | | | | X | |
| Concomitant medication | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Adverse events | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| IRT <sup>s</sup> | X | X | X | X | X | X | X | X | X) | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Bimekizumab,<br>adalimumab, or<br>placebo<br>administration <sup>s</sup> | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | | |

BSA=Body Surface Area; CV=cardiovascular; DLQI=Dermatology Life Quality Index; ECG=electrocardiogram; eCRF=electronic Case Report Form; eC-SSRS=electronic Columbia Suicide Severity Rating Scale; EQ-5D-3L=Euro-Quality of Life 5-Dimensions 3 Levels; GI=gastrointestinal; HCV=hepatitis C virus; HIV=human immunodeficiency virus; ICF=Informed Consent Form; IGA=Investigator's Global Assessment; IGRA=interferon-gamma release assay; IMP=investigational medicinal product; IRT=interactive response technology; mNAPSI=Modified Nail Psoriasis Severity Index Score; PASE=Psoriatic Arthritis Screening and Evaluation; PASI=psoriasis area severity index; PD=pharmacodynamic; PEOT=Premature End of Treatment Visit; PGADA=Patient Global Assessment of Disease Activity; PHQ-9=Patient Health Questionnaire-9; pp-IGA=palmoplantar Investigator's Global Assessment; PsA=psoriatic arthritis; SF-36=Short Form 36-item Health Survey; SFU=Safety Follow-Up; scalp IGA=scalp-specific Investigator's Global Assessment; TB=tuberculosis; WPAI-SHP=Work Productivity and Activity Impairment Questionnaire-specific health problem

<sup>&</sup>lt;sup>a</sup> Visit windows of ±3 days from the first dose at all visits except SFU. The SFU Visit window is -3 and +7 days from last dose.

<sup>&</sup>lt;sup>b</sup> The SFU Visit will occur 20 weeks after the last dose for subjects who do not enroll in the open-label study.

<sup>&</sup>lt;sup>c</sup> A separate ICF will be required for subjects who decide to participate in the genomics, genetics, and proteomics substudy. The ICF must be signed prior to collecting any samples for the substudy. The samples will be stored at -80°C at the central biorepository for up to 20 years.

<sup>&</sup>lt;sup>d</sup> A separate ICF is required to be completed for the open-label study.

**Table 5-1:** Schedule of study assessments

| Visit <sup>a</sup> /<br>Week | Screening | | Dou | ble-blin<br>(we | ıd Initia<br>eks afte | | | Period | | | | j | Dose-bli | nd Mainten<br>(weeks aft | , | | | eriod | | | W56/PEOT | SFU <sup>b</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Protocol activity | | Baseline<br>(first dose) | 3 | 4 | 5,<br>7 | 8 | 9,<br>11 | 12 | 13,<br>15 | 16 | 17,<br>19 | 20 | 21, 23 | 242 28 | 32 | 36 | 40 | 44 | 48 | 52 | 56 | |

- <sup>e</sup> Ensure no significant changes in medical history.
- f Includes evaluation of signs and symptoms of active TB and risk for exposure to TB.
- g The physical examination will include examination of the following systems: eyes, hair, and skin; respiratory; CV; and GI.
- h Vital signs (sitting systolic and diastolic blood pressure, pulse rate, and body temperature) are to be measured prior to blood sampling, and prior to dosing, where applicable.
- i Pregnancy testing will consist of serum testing at the Screening. The pregnancy test will be urine at all other visits.
- Subjects who have evidence of or test positive for hepatitis B by any of the following criteria: 1) positive for hepatitis B surface antigen (HBsAg+); 2) positive for anti-hepatitis B core antibody (HBcAb+) are excluded. A positive test for HCV is defined as: 1) positive for hepatitis C antibody (anti-HCV Ab), and 2) positive via a confirmatory test for HCV (for example, HCV polymerase chain reaction) are also excluded. Subjects will also be tested for anti-hepatitis B surface antibody.
- Screening chest x-ray must occur within 3 months prior to Screening Visit.

  Mall blood samples taken prior to dosing
- <sup>n</sup> The scalp IGA will only be assessed for those subjects with scalp involvement (scalp IGA score >0) at Baseline.
- <sup>o</sup> The mNAPSI will be assessed only in subjects with nail involvement (mNAPSI score >0) at Baseline.
- <sup>p</sup> The pp-IGA will only be assessed in subjects with palmoplantar involvement (pp-IGA score >0) at Baseline.
- <sup>q</sup> The Patient Global Assessment of psoriasis will be performed as part of the patient symptoms diary on a weekly basis from Screening through the Initial Treatment Period with a +3 day completion window. During the Maintenance Treatment Period this assessment will be completed at each clinic visit specified with a  $\pm 3$  day completion window.
- The PGADA is assessed for all subjects at Baseline. At all subsequent visits, the PGADA is only for subjects with PsA at Baseline (defined as a past medical history of PsA or PASE  $\geq$ 47).
- <sup>s</sup> IMP administration is based on randomization.

Table 5-1: Schedule of study assessments

| UCB<br>Clinical Study Prot | tocol | | | | | | | | Е | Bimeki | zumab | | | | | | | | | | S | 06 A | Apr 20<br>PS00 | )18<br>)08 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Has been chan | ged | to: | | | | | | | | | | | | | | | | | | idi | O, | | | |
| Table 5-1: | Sch | edu | le of | stud | y ass | sessi | nent | s | | | | | | | | | | | Or V | 91, | | | | |
| Visit <sup>a</sup> /<br>Week | Screening | | | Doul | | d Initia | | | Period | | | | I | Dose-bli | | | ance I | 10/1 | nent P | | | | W56/PEOT | $\mathbf{SFU}^{\mathrm{b}}$ |
| Protocol activity | | Baseline (first dose) | 1 | 3 | 4 | 5,<br>7 | 8 | 9,<br>11 | 12 | 13,<br>15 | 16 | 17,<br>19 | 20 | 21, 23 | 24 | 28 | 32 | 36 | 40 | 44 | 48 | 52 | 56 | |
| Informed consent <sup>c</sup> | X | | | | | | | | | | | 1 | olic | ,0 | | | | | | | | X <sup>d</sup> | | |
| Inclusion/exclusion | X | X | | | | | | | | | ر م | | 3,9% | | | | | | | | | | | |
| Urine drug screen | X | | | | | | | | | / | ) 1 | 110, | | | | | | | | | | | X | |
| Demographic data | X | | | | | | | | | CV. | Oil | | | | | | | | | | | | | |
| Psoriasis history | X | | | | | | | | COP | QUI | | | | | | | | | | | | | | |
| Significant past<br>medical history and<br>concomitant<br>diseases | X | Xe | | | | | | . ~ | Keil | (2) | | | | | | | | | | | | | | |
| Physical examination <sup>f,g</sup> | X | X | | | | | X | H | X | | X | | | | X | | | X | | | X | | X | X |
| Height | | X | | | | 5 | 0, | | | | | | | | | | | | | | | | | |
| Body weight | | X | | | | SUL | | | X | | X | | | | X | | | X | | | X | | X | |
| Vital signs <sup>h</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Hematology and biochemistry | X | X | X | X | X | | X | | X | | X | | X | | X | X | X | | X | | X | | X | X |
| Urinalysis | X | X | NO | > | | | | | | | X | | | | X | | X | | X | | X | | X | X |
| ECG | X | ~ | $\sim$ | | | | | | X | | X | | | | X | | | X | | | X | | X | |
| Confidential | JUM | S, | | | | | | | Pa | ıge 164 | l of 19 | 0 | | | | | | | | | | | | |

**Table 5-1:** Schedule of study assessments

| UCB<br>Clinical Study Prot | tocol | | | | | | | | I | Bimeki | zumab | | | | | | | | | . ( | 075 | 062 | Apr 20<br>PS00 | )18 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Table 5-1: | Sch | edu | le of | stud | y ass | sessr | nent | S | | | | | | | | | | | ,( | ai lail | | | | |
| Visit <sup>a</sup> /<br>Week | Screening | | | Doul | ble-blin<br>(wee | d Initia | | | Period | | | | ] | Dose-bli | nd Ma<br>(wee | ks aft | ance T | reatn | nent P | | | | W56/PEOT | SFUb |
| Protocol activity | | Baseline<br>(first dose) | 1 | 3 | 4 | 5,<br>7 | 8 | 9,<br>11 | 12 | 13,<br>15 | 16 | 17,<br>19 | 20 | 21, 23 | 242 | 28 | 32 | 36 | 40 | 44 | 48 | 52 | 56 | |
| Pregnancy testing <sup>i</sup> | X | X | | | X | | X | | X | | X | | X | tion | X | X | X | X | X | X | X | X | X | X |
| Hepatitis B and C<br>testing <sup>j</sup> | X | | | | | | | | | | | 7 | Oblic | | | | | | | | | | | |
| HIV testing <sup>k</sup> | X | | | | | | | | | | 0 | :01 | <i>y</i> . • | | | | | | | | | | | |
| Chest x-ray <sup>l</sup> | X | | | | | | | | | | 173 | ). · | | | | | | | | | | | | |
| IGRA Tuberculosis<br>test | X | | | | | | | | 10, | | 00, | | | | | | | | | | | X | | |
| Tuberculosis<br>questionnaire | X | X | | | | | | < | X | 0 | X | | | | X | | | X | | X | X | X | X | X |
| Blood sample for<br>bimekizumab<br>blasma<br>concentrations <sup>m</sup> | | X | X | X | X | | X | HINE | X | | X | | X | | X | | | X | | | X | | X | X |
| Blood sample for anti-bimekizumab antibodies <sup>m</sup> | | X | | | X | SUP | X | | X | | X | | X | | X | | | X | | | X | | X | X |
| Blood sample genomic, proteomic, and metabolomics, and candidate piomarker unalyses <sup>c,m</sup> | | X | X | loe i | Sedi | | X | | X | | X | | | | | | | | | | | | X | |

Table 5-1: Schedule of study assessments

| Table 5-1: | 3ch | edul | le of | stud | y ass | sessi | nent | s | | | | | | | | | | | \G | ailail | ) S | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit <sup>a</sup> /<br>Week | Screening | | | Douk | | d Initia | | | Period | | | | I | Oose-blii | nd Ma<br>(wee | intena<br>ks aft | ance T | reatn | o`<br>ient P | | | | W56/PEOT | SFIJ |
| Protocol activity | | Baseline<br>(first dose) | 1 | 3 | 4 | 5,<br>7 | 8 | 9,<br>11 | 12 | 13,<br>15 | 16 | 17,<br>19 | 20 | 21,<br>23 | 240 | 28 | 32 | 36 | 40 | 44 | 48 | 52 | 56 | |
| Blood sample<br>genetic/epigenetic<br>analyses <sup>c,m</sup> | | X | | | | | | | | | | 1 | dic | dilon | | | | | | | | | X | |
| PASI | X | X | X | X | X | | X | | X | | X | | X | | X | X | X | X | X | X | X | X | X | X |
| IGA | X | X | X | X | X | | X | | X | / | X | io | X | | X | X | X | X | X | X | X | X | X | X |
| Percentage of BSA | X | X | X | X | X | | X | | X | <u>~</u> | XIV | | X | | X | X | X | X | X | X | X | X | X | X |
| DLQI | | X | X | X | X | | X | | X | ali ali | Χ | | X | | X | | X | | X | | X | | X | |
| PHQ-9 | X | X | | | X | | X | < | X | 0 | X | | X | | X | X | X | X | X | X | X | X | X | |
| eC-SSRS | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Patient Symptom<br>Diary (daily) | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | | | | | | | | | |
| scalp IGA | | X | Xn | X <sup>n</sup> | X <sup>n</sup> | | $X_{\sigma}$ | | X <sup>n</sup> | | Xn | | X <sup>n</sup> | | Xn | | X <sup>n</sup> | | Xn | | Xn | | Xn | |
| mNAPSI | | X | | | Xº | CUR | $X_{o}$ | | Xº | | Xº | | Xº | | Xº | | Xº | | Xº | | Xº | | Xº | |
| pp-IGA | | X | | | Xp | ) | Xp | | Xp | | Xp | | Xp | | X <sup>p</sup> | | X <sup>p</sup> | | $X^p$ | | Xp | | Xp | |
| EQ-5D-3L | | X | | | X | | X | | X | | X | | | | X | | | | X | | | | X | |
| SF-36 | | X | | Sol Sol | X | | X | | X | | X | | | | X | | | | X | | | | X | |
| Patient global assessment of psoriasis <sup>q</sup> Confidential | | . C | anno | | | | | | | | | | | | X | | X | | X | | X | | X | |

Table 5-1: Schedule of study assessments

| Visit <sup>a</sup> /<br>Week | Screening | | | Dou | ble-blin<br>(we | ıd Initis<br>eks afto | | | Period | | | | Г | Oose-bli | | | | Treatn | | eriod | | | W56/PEOT | $\mathbf{SFU}^{\mathbf{b}}$ |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Protocol activity | | Baseline<br>(first dose) | 1 | 3 | 4 | 5,<br>7 | 8 | 9,<br>11 | 12 | 13,<br>15 | 16 | 17,<br>19 | 20 | 21,<br>23 | 242 | 28 | 32 | 36 | 40 | 44 | 48 | 52 | 56 | |
| PASE | | X | | | | | | | | | | | | ijon | | | | | | | | | X | |
| PGADA <sup>r</sup> | | X | | | X | | | | X | | X | 1 | -Olic | 0 | X | | X | | X | | X | | X | |
| WPAI-SHP V2.0 | | X | | | | | | | | | XO | | 367 | | X | | | | X | | | | X | |
| Concomitant medication | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Adverse events | X | X | X | X | X | X | X | X | X | X X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| IRT <sup>s</sup> | X | X | X | X | X | X | X | X | X) | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Bimekizumab,<br>adalimumab, or<br>placebo<br>administration <sup>s</sup> | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | | |

BSA=Body Surface Area; CV=cardiovascular; DLQI=Dermatology Life Quality Index; ECG=electrocardiogram; eCRF=electronic Case Report Form; eC-SSRS=electronic Columbia Suicide Severity Rating Scale; EQ-5D-3L=Euro-Quality of Life 5-Dimensions 3 Levels; GI=gastrointestinal; HCV=hepatitis C virus; HIV=human immunodeficiency virus; ICF=Informed Consent Form; IGA=Investigator's Global Assessment; IGRA=interferon-gamma release assay; IMP=investigational medicinal product; IRT=interactive response technology; mNAPSI=Modified Nail Psoriasis Severity Index Score; PASE=Psoriatic Arthritis Screening and Evaluation; PASI=psoriasis area severity index; PD=pharmacodynamic; PEOT=Premature End of Treatment Visit; PGADA=Patient Global Assessment of Disease Activity; PHQ-9=Patient Health Questionnaire-9; pp-IGA=palmoplantar Investigator's Global Assessment; PsA=psoriatic arthritis; SF-36=Short Form 36-item Health Survey; SFU=Safety Follow-Up; scalp IGA=scalp-specific Investigator's Global Assessment; TB=tuberculosis; WPAI-SHP=Work Productivity and Activity Impairment Questionnaire-specific health problem


<sup>&</sup>lt;sup>a</sup> Visit windows of ±3 days from the first dose at all visits except SFU. Visit windows of ±3 days from the first dose to the Week 24 visit. Visit windows of ±7 days from the Week 28 visit to the Week 52 visit. The SFU Visit window is -3 and +7 days from last final dose.

<sup>&</sup>lt;sup>b</sup> The SFU Visit will occur 20 weeks after the last final dose for subjects who do not enroll in the open-label study.

<sup>&</sup>lt;sup>c</sup> A separate ICF will be required for subjects who decide to participate in the genomics, genetics, and proteomics substudy. The ICF must be signed prior to collecting any samples for the substudy. All genomic, proteomic, and metabolomics samples will be stored at -80°C at the central biorepository

### Table 5-1: Schedule of study assessments

| Visit <sup>a</sup> /<br>Week | Screening | | Doul | ble-blin<br>(wee | d Initia | | | Period | | | | I | Dose-blii | nd Mainten<br>(weeks aft | | | | eriod | | | W56/PEOT | $\mathbf{SFU}^{\mathrm{b}}$ |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Protocol activity | | Baseline<br>(first dose) | 3 | 4 | 5,<br>7 | 8 | 9,<br>11 | 12 | 13,<br>15 | 16 | 17,<br>19 | 20 | 21, 23 | 242 28 | 32 | 36 | 40 | 44 | 48 | 52 | 56 | |

for up to 20 years.

- <sup>d</sup> A separate ICF is required to be completed for the open-label study.
- <sup>e</sup> Ensure no significant changes in medical history.
- f Includes evaluation of signs and symptoms of active TB and risk for exposure to TB.
- g The physical examination will include examination of the following systems: eyes, hair, and skin; respiratory; CV; and GI be performed as per Section 12.3.5.
- h Vital signs (sitting systolic and diastolic blood pressure, pulse rate, and body temperature) are to be measured prior to blood sampling, and prior to dosing, where applicable.
- i Pregnancy testing will consist of serum testing at the Screening. The pregnancy test will be urine at all other visits.
- Subjects who have evidence of or test positive for hepatitis B by any of the following criteria: 1) positive for hepatitis B surface antigen (HBsAg+); 2) positive for anti-hepatitis B core antibody (HBcAb+) are excluded. A positive test for HCV is defined as: 1) positive for hepatitis C antibody (anti-HCV Ab), and 2) positive via a confirmatory test for HCV (for example, HCV polymerase chain reaction) are also excluded. Subjects will also be tested for anti-hepatitis B surface antibody.
- <sup>k</sup> The HIV test results will not be recorded in the eCRF.
- <sup>1</sup> Screening chest x-ray must occur within 3 months prior to Screening Visit.
- <sup>m</sup> All blood samples taken prior to dosing.
- <sup>n</sup> The scalp IGA will only be assessed for those subjects with scalp involvement (scalp IGA score >0) at Baseline.
- ° The mNAPSI will be assessed only in subjects with nail involvement (mNAPSI score >0) at Baseline.
- <sup>p</sup> The pp-IGA will only be assessed in subjects with palmoplantar involvement (pp-IGA score >0) at Baseline.
- <sup>q</sup> The Patient Global Assessment of psoriasis will be performed as part of the patient symptoms diary on a weekly basis from Screening through the Initial Treatment Period with a +3 day completion window at the specified clinic visits. During the Maintenance Treatment Period this assessment will be completed at each clinic visit specified with a ±3 day completion window at the specified clinic visits.
- The PGADA is assessed for all subjects at Baseline. At all subsequent visits, the PGADA is only for subjects with PsA at Baseline (defined as a past medical history of PsA or PASE ≥47).
- s IMP administration is based on randomization. The dosing window is ±3 days relative to the scheduled dosing visit through Week 24. The dosing window is ±7 days from Week 28 through the end of the study.


### Section 5.7 Schematic diagram

Section 6.1 Inclusion criteria

To be eligible to participate in this study, all of the following criteria must be met at Screening and be reconfirmed at the Baseline Visit:

6. Subject is a candidate for systemic PSO therapy and/or phototherapy and/or photochemotherapy.

Have been changed to:

i o be eligible to participate in this study, all of the following criteria must be met at Screening and be reconfirmed at the Baseline Visit:

6. Subject is a candidate for systemic PSO therapy and/or phototherapy and/or photochemotherapy.

Have been changed to:

i o be eligible to participate and be reconfirmed at the Baseline Visit:

and be reconfirmed at the Baseline Visit:

6a. Subject is a candidate for systemic PSO therapy and/or phototherapy-and/or photochemotherapy.

### Change #18

#### **Exclusion criteria** Section 6.2

- 3. Subject previously participated in another study of a medication (systemic) under investigation within the 12 weeks or at least 5 half-lives prior to the Screening Visit, whichever is greater, or is currently participating in another study of a medication (systemic) under investigation.
- 4. Subject previously participated in another study of a topical medication under investigation within the 4 weeks prior to the Screening Visit, or is currently participating in another study of a topical medication under investigation.
- 5. Subject previously participated in another study of a medical device under investigation within the 4 weeks prior to the Screening Visit, or is currently participating in another study of a medical device under investigation.
- 14. Subject has any active malignancy or history of malignancy within 5 years prior to the Screening Visit EXCEPT treated and considered cured cutaneous squamous or basal cell
- diabetes) considered by the Investigator to be uncontrolled, unstable, or likely to progress to a clinically significant degree during the course of the study.

  27. Subject has presence of severe degree.
  - screening PHO-9. Medication used to treat depression should be stable for 4 weeks prior to Baseline.

#### Have been changed to:

- 3a. Subject previously participated in another study of a medication (systemic) under investigation within the 12 weeks or at least 5 half lives prior to the Screening Visit, whichever is greater, or is currently participating in another study of a medication (systemic) under investigation. Subject must be washed out of the medication for 12 weeks or at least 5 half-lives prior to the Baseline Visit, whichever is greater.
- 4a. Subject previously participated in another study of a topical medication under investigation within the 4 weeks prior to the Screening Visit, or is currently participating in another study of a topical medication under investigation. Subject must be washed out of the medication for 4 weeks prior to the Baseline Visit.
- 5a. Subject previously participated in another study of a medical device under investigation within the 4 weeks prior to the Screening Visit, or is currently, or was within the 4 weeks prior to the Baseline Visit, participating in another study of a medical device under investigation.
- 14a. Subject has any active malignancy or history of malignancy within 5 years prior to the Screening Visit EXCEPT treated and considered cured cutaneous squamous or basal cell carcinoma, or in situ cervical cancer, or ductal carcinoma in situ of the breast.
- 17a. Subject has any systemic disease (eg, renal failure, heart failure, hypertension, liver disease, diabetes ie, cardiovascular, neurological, renal, liver, metabolic, gastrointestinal, hematological, immunological, etc.) considered by the Investigator to be uncontrolled, unstable, or likely to progress to a clinically significant degree during the course of the study.
- 27a. Subject has presence of **moderately severe major depression or** severe **major** depression, indicated by a score of ≥15 using the screening PHQ-9. Medication used to treat depression should be stable for **4-8** weeks prior to Baseline.

Section 6.2 Exclusion criteria

The following text has been added:

30. Subject is taking or has taken prohibited psoriasis medications without meeting the mandatory washout period relative to the Baseline Visit (Table 7–2).

Change #20

Section 6.3 Withdrawal criteria

The following withdrawal criteria have been added, modified, and/or renumbered:

- 8. At Week 28 and all following visits, subjects on continuous treatment with the same IMP for at least 12 weeks with a persistent IGA score ≥3 over at least a 4-week period are defined as nonresponders and should discontinue IMP.
- There is confirmation of a pregnancy during the study, as evidenced by a positive pregnancy test (see Section 12.1.4 for more information regarding pregnancies).
- 10. A subject considered as having either a suspected new LTB infection or who develops active TB or NTMB infection during the study (including but not limited to, conversion demonstrated by IGRA or other diagnostic means) must be immediately discontinued from

IMP and a PEOT Visit must be scheduled as soon as possible, but not later than the next regular visit.

The subject must be permanently withdrawn if further examinations result in a diagnosis of active TB, or if the subject is diagnosed with latent TB infection (LTBI) with no initiation of prophylactic treatment, prematurely discontinues prophylactic treatment, or, in the opinion of the Investigator or Sponsor, is noncompliant with prophylactic TB therapy.

Confirmed active TB is an SAE and must be captured on an SAE Report Form and provided to the Sponsor in accordance with SAE reporting requirements. As with all SAEs, periodic following reports should be completed as per protocol requirements until such time as the TB infection resolves.

Additional information on TB policies is provided in Section 12.3.1.

- 11. Subjects with newly diagnosed inflammatory bowel disease (IBD) or with IBD flares during the study must:
- Be referred, as appropriate, to a health care professional treating IBD, such as a gastroenterologist
- Discontinue IMP and be followed-up until resolution of active IBD symptoms

If IBD flares increase in severity or frequency during the study, the Investigator should use clinical judgement in deciding whether the subject should continue in the study and contact the Medical Monitor and UCB study physician to confirm the subject's suitability for continued participation in the study.

- 12. Subjects **must be referred** immediately to a mental health care professional and may be withdrawn from the study based upon the Investigator's judgment of benefit/risk-for either of the following:
- Active suicidal ideation as indicated by a positive response ("Yes") to Questions 4 or 5 or to the suicidal behavior questions of the "Since Last Visit" version of the eC-SSRS.
- Moderately severe **major** depression as indicated by a PHQ-9 score of 15 to 19 if this represents an increase of 3 points compared to last visit.
- 13. Subjects must be referred immediately to a mental healthcare professional and must be withdrawn in case of
- Active suicidal ideation as indicated by a positive response ("Yes") to Question 5 of the "Since Last Visit" version of the eC-SSRS
- Any suicidal behavior since last visit.
- Severe **major** depression as indicated by a PHQ-9 score  $\geq$ 20.

The mental health consultation will be documented must be recorded in source documentation.

### Section 7.1 Description of investigational medicinal product(s)

### Has been changed to:

Adalimumab is commercially available and will be supplied as a PFS for sc injection (at a concentration of 40mg/0.8mL or 40mg/0.4mL depending on regional availability) in single-use syringein a 1mL PFS at a concentration of 40mg/0.8ml injection. mjectio, availability)
or 10mg/0.4ml,
or 10mg/0.4ml,
and any other birth of the product of the production of the product




**Table 7-1: Dosing scheme** 

| | | | | Initia | l Trea | tment | | | | | | | Mai | ntena | ance T | reatn | ent | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Week<br>Dose Assignment | 0 | 1, | 4 | 5,<br>7 | 8 | 9,<br>11 | 12 | 13,<br>15 | 16 | 17,<br>19 | 20 | 21,<br>23 | 24 | 28 | 32 | 36 | 40 | 44 | 48 | 52 |
| bimekizumab 320mg<br>Q4W/Q4W | •• | 0 | •• | 0 | •• | 0 | •• | 0 | •• | 0 | •• | 0 | •• | et c | •• | •• | •• | •• | •• | •• |
| bimekizumab 320mg<br>Q4W/Q8W | •• | 0 | •• | 0 | •• | 0 | •• | 0 | •• | 0 | 00 | oil | 36 | 00 | •• | 00 | •• | 00 | •• | 00 |
| adalimumab 40mg | <b>A A</b> | <b>A</b> | 00 | <b>A</b> | 00 | <b>A</b> | 00 | <b>A</b> | 00 | <b>A</b> | 00 | 0/7 | •• | •• | •• | •• | •• | •• | •• | •• |

Q+w=every 4 weeks; Q8W=every 8 weeks

Notes: A bimekizumab 160mg injection is depicted by a black circle (•). A placebo injection is depicted by a white circle (○). An adalimumab 40mg injection is depicted by a black triangle (▲)

Has been changed to:

Table 7-1: Dosing scheme

| Week<br>Dose Assignment | 0 | 1, | 4 | 5,<br>7 | 8 | 9,<br>11 | 212 | 13,<br>15 | 16 | 17,<br>19 | 20 | 21,<br>23 | 24 | 28 | 32 | 36 | 40 | 44 | 48 | 52 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| bimekizumab 320mg<br>Q4W/Q4W | • | 0 | •• | 0 | •• | on | | 0 | • | 0 | • | 0 | • | • | • | • | • | • | •• | • |
| bimekizumab 320mg<br>Q4W/Q8W | •• | 0 | •• | 0 | OIX. | | •• | 0 | •• | 0 | 00 | 0 | •• | 00 | •• | 00 | •• | 00 | •• | 00 |
| adalimumab<br>40mg/bimekizumab<br>320mg Q4W | <b>A A</b> | <b>A</b> | 00 | <b>4</b> 50 | 200 | <b>A</b> | 0 | <b>A</b> | 00 | <b>A</b> | 00 | <b>A</b> | • | • | •• | •• | • | •• | •• | • |

Q4W=every 4 weeks; Q8W=every 8 weeks

Notes: A bimekizumab 160mg injection is depicted by a black circle (•). A placebo injection is depicted by a white circle (o). An adalimumab 40mg injection is Notes: A bimekizumab 160mg injection depicted by a black triangle (▲).


### **Section 7.6 Drug Accountability**

Blinded study staff may be delegated the responsibility to receive, inventory, and destroy the used kits. The packaging identifies each kit by a unique number that does not correlate to the contents and therefore, does not unblind study site staff. Unblinded study staff will be responsible for preparation (breaking tamper proof sticker on kit, etc) of the clinical study material, including recording the administration information on source documents.

### Has been changed to:

Unblinded study staff will be delegated the responsibility to receive, inventory and destroy the used kits. The packaging identifies each kit by a unique number, but due to the commercial packaging of the comparator, the unblinded study staff will be responsible in order to maintain the blind. Blinded study staff may be delegated the responsibility to receive, inventory, and destroy the used kits. The packaging identifies each kit by a unique number that does not correlate to the contents and therefore, does not unblind study site staff. Unblinded study staff will be responsible for preparation (breaking tamper proof sticker on kit, etc) of the clinical study material, including recording the administration information on source documents.

#### Change #24

# Section 7.8.2 Prohibited concomitant treatments (medications and therapies), Table 7-2

Table 7-2: Prohibited psoriasis medications

| Drug P H | Washout period relative to Baseline Visit |
|---|---|
| Topicals except for those permitted (Section 7.8 f.1) | 2 weeks |
| Systemic retinoids | 3 months |
| Systemic treatment (nonbiological): systemic immunosuppressant agents (eg, methotrexate, cyclosporine, azathioprine, thioguanine) fumaric acid esters specifically used for the treatment of PSO systemic corticosteroids phototherapy or photochemotherapy | 1 month |
| Anti-TNFs: | |
| adatimumab (including biosimilar) | Any exposure to adalimumab |
| etanercept (including biosimilar) | 1 month for etanercept |
| infliximab (including biosimilar), golimumab, certolizumab pegol | 3 months for infliximab (including biosimilar), golimumab, certolizumab pegol |
| Other biologics and other systemic therapies, eg: | |
| apremilast, tofacitinib | 2 weeks for apremilast and tofacitinib |

**Table 7-2: Prohibited psoriasis medications** 

| Drug | Washout period relative to Baseline Visit |
|---|---|
| alefacept, efalizumab, guselkumab | 3 months for alefacept, efalizumab, and guselkumab |
| ustekinumab, briakinumab | 6 months for ustekinumab and briakinumab |
| rituximab | 12 months for rituximab |
| Anti-IL-17 therapy: | 3 months |
| brodalumab | (bimekizumab is excluded per exclusion |
| ixekizumab | criteria) |
| secukinumab | delle |
| Any other antipsoriatic agent (systemic) under | 3 months or 5 half-lives, whichever is greater |
| investigation (or approved after the protocol is approved) | 7 3/2 |
| Any other antipsoriatic agent (topical) under | 1 month |
| investigation | aliv |

IL-17=interleukin 17; PSO=psoriasis; TNF=tumor necrosis factor

| investigation | |
|---|---|
| IL-17=interleukin 17; PSO=psoriasis; TNF=tumor necrosis | factor |
| IL-17=interleukin 17; PSO=psoriasis; TNF=tumor necrosis Has been changed to: Table 7-2: Prohibited psoriasis medication Drug Topicals except for those permitted (Section 7.8.D.1) | OPT 20P |
| Table 7-2: Prohibited psoriasis medication | ons |
| Drug | Washout period relative to Baseline Visit |
| Topicals except for those permitted (Section 7.8.1.1) | 2 weeks |
| Systemic retinoids | 3 months |
| Systemic treatment (nonbiological): systemic immunosuppressant agents (eg, methotrexate, cyclosporine, azathioprine, thioguanine) fumaric acid esters specifically used for the treatment of PSO systemic corticosteroids phototherapy or photochemotherapy | 1 month |
| Anti-TNFs: | |
| adalimumab (including biosimilar) etanercept (including biosimilar) infliximab (including biosimilar), golimumab, certolizumab pegol | Any exposure to adalimumab 1 month for etanercept 3 months for infliximab (including biosimilar), golimumab, certolizumab pegol |
| Other biologics and other systemic therapies, eg: | |
| apremilast, tofacitinib | 2 weeks for apremilast and tofacitinib |
| alefacept, efalizumab, guselkumab | 3 months for alefacept, efalizumab, and guselkumab |

Table 7-2: Prohibited psoriasis medications

| Drug | Washout period relative to Baseline Visit |
|---|---|
| tildrakizumab, risankizumab | 5 months for tildrakizumab and risankizumab |
| ustekinumab, briakinumab | 6 months for ustekinumab and briakinumab |
| rituximab | 12 months for rituximab |
| Anti-IL-17 therapy: brodalumab ixekizumab secukinumab | 3 months (bimekizumab is excluded per exclusion criteria) |
| Any other antipsoriatic agent (systemic) under investigation (or approved after the protocol is approved) | 3 months or 5 half-lives, whichever is greater |
| Any other antipsoriatic agent (topical) under investigation | 1 month |

IL-17=interleukin 17; PSO=psoriasis; TNF=tumor necrosis factor

#### Change #25

# Section 7.10 Randomization and numbering of subjects, first paragraph

An IRT will be used for assigning eligible subjects to a treatment regimen based on a predetermined production randomization and/or packaging schedule provided by UCB (or designee). The randomization schedule will be produced by the IRT vendor. The IRT will generate individual assignments for subject kits of IMP, as appropriate, according to the visit schedule. Subject treatment assignment will be stratified by region and prior biologic exposure (yes/no). The IRT will generate individual assignments for subject kits of IMP, as appropriate, according to the visit schedule.

### Has been changed to:

An IRT will be used for assigning eligible subjects to a treatment regimen based on a predetermined production randomization and/or packaging schedule provided by UCB (or designee). The randomization schedule will be produced by the IRT vendor. The IRT will generate individual assignments for subject kits of IMP, as appropriate, according to the visit schedule. Subject treatment assignment will be stratified by region (North America, Western Europe, Central/Eastern Europe and Asia/Australia) and prior biologic exposure (yes/no). The IRT will generate individual assignments for subject kits of IMP, as appropriate, according to the visit schedule.

#### **Change #26**

#### Section 8 STUDY PROCEDURES BY VISIT, first bullet

• Visit windows of  $\pm 3$  days on either side of the scheduled dosing are permitted; however, the Investigator should try to keep the subjects on the original dosing schedule. The window of

- $\pm 3$  days is relative to Baseline and applicable for all subsequent visits. Changes to the dosing schedule outside of the 3-day window must be discussed with the Medical Monitor.
- For the SFU Visit (20 weeks after the last dose), the visit should occur no more than 3 days

- From the Week 1 Visit to the Week 24 visit, Visit visit windows of ±3 days on either side of the scheduled dosing are permitted; however, the Investigator should try to keep the subjects on the original dosing schedule. The window of ±3 days in applicable for all subsequent visits. From the windows are ±7 days of the subsequent visits. discussed with the Medical Monitor.
- The dosing window is  $\pm 3$  days relative to the scheduled dosing visit through Week 24. The dosing window is  $\pm 7$  days relative to the scheduled dosing visit from Week 28 through the end of the study.
- For the SFU Visit (20 weeks after the last final dose), the visit window is  $\pm 7$  days relative to the scheduled visit date. should occur no more than 3 days prior to the scheduled visit date and within 7 days after the scheduled visit date ( 3 days/+7 days).

Change #27

Section 8.1 Screening Visit (2 to 4 weeks)

Has been changed to:

Section 8.1 Screening Visit (2 to 4-5 weeks

Change #28

Section 8.1 Screening Visit (2 to 4 weeks)

IGRA tuberculosis test; it is recommended that the QuantiFERON TB GOLD test be performed

### Has been changed to:

IGRA tuberculosis test; it is recommended that the QuantiFERON TB GOLD test be performed

Change #29 ©

Sections 8.2.1 Baseline Visit

The following has been added to the bulleted list:

Physical examination including evaluation of signs and symptoms of active TB and risk for exposure to TB

Sections 8.2.8 Week 12 ( $\pm 3$  days)

days), and 8.3.12 Week 56 (±3 days)

Has been changed to:

Sections 8.3.5 Week 28 ( $\pm 3 \pm 7$  days), 8.3.6 Week 32 ( $\pm 3 \pm 7$  days), 8.3.7 Week 36 ( $\pm 3 \pm 7$ (days), 8.3.8 Week 40 ( $\pm 3\pm 7$  days), 8.3.9 Week 44 ( $\pm 3\pm 7$  days), 8.3.10 Week 48 ( $\pm 3\pm 7$  days), 8.3.11 Week 52 ( $\pm 3$ - $\pm 7$  days), and 8.3.12 Week 56 ( $\pm 3$ - $\pm 7$  days)

#### Sections 8.3.11 Week 52 ( $\pm 3$ days)

IGRA tuberculosis test; it is recommended that the QuantiFERON TB GOLD test be performed

### Has been changed to:

extensions or variations thereof. IGRA tuberculosis test; it is recommended that the QuantiFERON TB GOLD test be performed

#### Change #37

Section 8.5 Safety Follow Up Visit (20 weeks after last dose  $\pm$ -3/+7 days)

Has been changed to:

Section 8.5 Safety Follow Up Visit (20 weeks after last final dose  $\pm 3/\sqrt[4]{3}$ 

Change #38

#### **Section 9 ASSESSMENT OF EFFICACY**

The PASI, BSA, IGA, scalp IGA, mNAPSI, and pp-IGA should be performed by the Investigator, another delegated physician, or an appropriately qualified medical professional (based on local requirements) who has had documented training on how to perform these assessments correctly. Preferably, the same assessor should evaluate the subject at each assessment.

#### Has been changed to:

The PASI, BSA, IGA, scalp IGA, mNAPSI, and pp-IGA should be performed by the Investigator, another delegated physician, or an appropriately qualified medical professional (based on local requirements) who has had documented training on how to perform these assessments correctly. Preferably, the The same assessor should evaluate the subject at each assessment.

#### Change #39

### Section 9.10 Patient Global Assessment of psoriasis, second and third paragraphs

The Patient Global Assessment of PSO will be performed as part of the patient symptoms diary from baseline through the Initial Treatment Period; the assessment is to completed within a +3 day completion window at each of the visits specified in Table 5-1.

During the double-blind Maintenance Treatment Period, this assessment will be completed within a +3 day completion window at the visits specified in Table 5-1.

Has been changed to:
The Patient C1 The Patient Global Assessment of PSO will be performed as part of the patient symptoms diary from baseline Screening through the Initial Treatment Period; the assessment is to be completed within a +3 day completion window at each of the visits specified in Table 5 1.

During the double-blind Maintenance Treatment Period, this assessment will be completed within a +3 day completion window at the visits specified in Table 5-1.

appropriate anchor items at the end of every study week. The ePRO diary software will be programmed such that the subjects will be given a window of opportunity to complete the ePRO diaryeach evening. The data collected on the ePRO diary will be uploaded to a central server database and will be 21 CFR Part 11 compliant. Appropriate GCP process

Has been charmal.

### Has been changed to:

The ePRO diary will also administer the patient global assessment of PSO as noted above appropriate anchor items at the end of every study week. The ePRO diary software will be programmed such that the subjects will be given a window of opportunity to complete the ePRO diary each evening. The data collected on the ePRO diary will be uploaded to a central server database and will be 21 CFR Part 11 compliant. Appropriate GCP procedures (including subject/site training and testing) will be performed at the study sites.

### Change #41

### Section 9.12 PASE questionnaire

Standardized responses are based on 5 categories relating to agreement (strongly agree [1], agree [2], no idea [3], disagree [4], and strongly disagree [5]). The total maximum score is 75 points (symptom score: 35 points and function score: 40 points).

#### Has been changed to:

Standardized responses are based on 5 categories relating to agreement (strongly agree [1-5], agree [2-4], no idea [3], disagree [4-2], and strongly disagree [5-1]). The total maximum score is 75 points (symptom score: 35 points and function score: 40 points).

#### Change #42

#### Section 12.1.4 Pregnancy

A pregnancy becomes an SAE in the following circumstances: miscarriage, abortion (elective or spontaneous), unintended pregnancy after hormonal contraceptive failure (if the hormonal contraceptive was correctly used), ectopic pregnancy, fetal demise, or any congenital anomaly/birth defect of the baby.

#### Has been changed to:

A pregnancy becomes an SAE in the following circumstances: miscarriage, abortion (elective or spontaneousel elective-abortion when medically indicated (e.g. when pregnancy is endangering life or health of woman or when fetus will be born with severe abnormalities), unintended pregnancy after hormonal contraceptive failure (if the hormonal contraceptive was correctly used), ectopic pregnancy, fetal demise, or any congenital anomaly/birth defect of the baby.

### **Section 12.2 Laboratory measurements**

Table 12-2: Laboratory measurements

| Hematology | Chemistry | Urinalysis dipstick <sup>a</sup> |
|---|---|---|
| Basophils | Calcium | рН |
| Eosinophils | Chloride | Albumin (protein) |
| Lymphocytes | Magnesium | Glucose |
| Atypical lymphocytes | Potassium | Blood |
| Monocytes | Sodium | Leukocyte esterase |
| Neutrophils | Glucose | Nitrite |
| Hematocrit | BUN | Urine dipstick for pregnancy testing <sup>b</sup> |
| Hemoglobin | Creatinine | Urine drug screen <sup>d</sup> |
| MCH | ALP | ajijo |
| MCHC | AST | Spire |
| MCV | ALT | 8 |
| Platelet count | GGT LD 12th | |
| RBC count | Total bilirubin | |
| WBC count | LDH LO BULL | |
| _ | Serum pregnancy testing <sup>b</sup> | |

# Has been changed to:

Table 12-2: Laboratory measurements

| Hematology | Chemistry | Urinalysis dipstick <sup>a</sup> |
|---|---|---|
| Basophils | Calcium | pН |
| Eosinophils | Chloride | Albumin (protein) |
| Lymphocytes | Magnesium | Glucose |
| Atypical lymphocytes | Potassium | Blood |
| Monocytes | Sodium | Leukocyte esterase |
| Neutrophils | Glucose | Nitrite |
| Hematocrit | BUN | Urine dipstick for pregnancy testing <sup>b</sup> |
| Hemoglobin | Creatinine | Urine drug screen <sup>d</sup> |
| MCH | ALP | |
| MCHC | AST | |

### **Table 12-2: Laboratory measurements**

| Hematology | Chemistry | Urinalysis dipstick <sup>a</sup> |
|---|---|---|
| MCV | ALT | |
| Platelet count | GGT | |
| RBC count | Total bilirubin | , and the second |
| WBC count | LDH | Jalio |
| | Serum pregnancy testing <sup>b</sup> | or |

Change #44

Section 12.2.1 Evaluation of PDILI

Rechallenge with a substance potentially causing drug-induced liver injury is dangerous, may be fatal, and must not occur. fatal, and must not occur.

### Has been changed to:

Rechallenge with a substance potentially causing drug induced liver injury is dangerous, may be fatal, and must not occur.

#### Change #45

# Section 12.2.1.2.1 IMP restart/rechallenge (if applicable)

Rechallenge with a substance potentially causing drug-induced liver injury is dangerous, may be fatal, and must not occur.

### Has been changed to:

### Section 12.2.1.2.1 IMP restart/rechallenge (if applicable)

Rechallenge with a substance potentially causing drug induced liver injury is dangerous, may be fatal, and must not occur. Rechallenge with IMP can occur only if ALL of the following requirements are met:

- The results of additional testing and monitoring described in Section 12.2.1.3 and Section 12.2.1.4 confirm a nondrug-related cause for the abnormal hepatic laboratory parameters and any associated symptoms (ie, a subsequent alternative diagnosis fully explains the hepatic findings).
- The subject has shown clear therapeutic benefit from the IMP.
- Subject's ALT or AST elevations do not exceed ≥5xULN.
- Subject's total bilirubin is <2xULN.
- Subject has no signs or symptoms of hypersensitivity or hepatitis.
- The rechallenge is approved by the UCB responsible physician, DMC, and a hepatologist. The hepatologist must be external to UCB but may be a member of the


### DMC. It is recommended that the hepatologist be a local hepatology expert or the hepatologist treating the subject.

At Screening, all subjects will have an IGRA test (QuantiFERON TB GOLD is recommended), action chest x-ray (unless already performed within 3 months of Screening) and examination for signor and symptoms of TB.

Change #47

### Section 12.3.1 Assessment and management of TB and TB risk factors

- b. High risk of acquiring TB infection:
  - Known exposure to another person with active TB infection within the 3 months prior to Screening.

#### Has been changed to:

- b. High risk of acquiring TB infection:
  - Known close exposure to another person with active TB infection within the 3 months prior to Screening.

### Has been changed to:

At Screening, all subjects will have an IGRA test (QuantiFERON TB GOLD test is recommended), a chest x-ray (unless already performed within 3 months of Screening) and examination for signs and symptoms of TB.

#### Change #48

### Section 12.3.1.1 Tuberculosis assessment by IGRA

During conduct of the study, the TB assessment by IGRA (QuantiFERON TB GOLD is recommended) will be performed as described in Table 5-1 for all subjects.

### Has been changed to:

During conduct of the study, the TB assessment by IGRA (QuantiFERON TB GOLD test is recommended) will be performed as described in Table 5-1 for all subjects.

# Change #49

#### Section 12.3.1.3 Tuberculosis questionnaire, last paragraph

Has been deleted: Subjects with a latent or active TB infection must be withdrawn from the study.

Subjects with a latent or active TB infection must be withdrawn from the study.

#### Change #50

#### Section 12.3.1.4 Tuberculosis management, second paragraph

During the study, subjects who develop evidence of LTB infection or active TB must immediately stop further administration of IMP and will be referred to an appropriate TB Indicate the state of the state specialist (pulmonologist or infectious disease specialist) for further evaluation. Evidence of

specialist (pulmonologist or infectious disease specialist) for further evaluation. Evidence of LTB infection is defined as subject's IGRA test converts to positive or indeterminate (and confirmed indeterminate on repeat), or the subject's questionnaire or history and physical indicates that TB infection or exposure may have occurred. Evidence of active TB includes, in addition to the aforementioned tests, signs and symptoms of organ involvement. In either situation, the subject should be carefully assessed by a TB specialist for active TB. Subjects diagnosed with active TB or LTB infection should be withdrawn from the study and receive appropriate TB or prophylaxis therapy.

Change #51

Section 12.3.2 Pregnancy testing

A negative urine pregnancy test result should be obtained immediately prior to each

administration of IMP and at all subsequent postdosing visits.

### Has been changed to:

A negative urine pregnancy test result should be obtained immediately prior to each administration of IMP and at all subsequent postdosing visits at the visits specified in **Table 5-1**.

#### Change #52

Section 14.1 Definition of analysis sets

The following analysis set has been added:

The Bimekizumab Set (BKZ Set) will consist of all subjects who have received at least 1 dose of bimekizumab in this study.

Section 14.1 Definition of analysis sets

The Full Analysis C The Full Analysis Set (FAS) will consist of all randomized subjects that receive at least 1 dose of the IMP and have a valid measurement of the primary efficacy variable at Baseline.

The Full Analysis Set (FAS) will consist of all randomized subjects that receive at least 1 dose of Has been changed to:

The hypotheses (H<sub>1</sub>, H<sub>2</sub>, H<sub>3</sub>, H<sub>4</sub>, H<sub>5</sub>, H<sub>6</sub>, H<sub>7</sub>, H<sub>8</sub>, H<sub>9</sub>, H<sub>10</sub>, H<sub>11</sub> and H<sub>12</sub>) comparing bimekizumab vs. adalimumab will be tested at a 2-sided alpha level of 0.05.

Change #55

Section 14.2 General statistical considerations

Figure 14-1: Sequence of testing

Image: Sequence of testing



Note: all calculations above are based on the combined Bimekizumab arms with the sample size of 300.

Figure 14-1: Sequence of testing



Note: Calculations for  $H_1$ - $H_2$  are based on the combined Bimekizumab arms with the sample size of 300. \* in  $H_{10}$ - $H_{12}$  indicated calculations are based on the Bimekizumab Q4W/Q4W arm only with sample size of 150.

### Change #56

# Section 14.3.2.1.2 Maintenance Treatment Period

The secondary efficacy variables in the Maintenance Treatment Period include PASI90, PASI100, and IGA at Week 24 and Week 56.

## Has been changed to:

The secondary efficacy variables in the Maintenance Treatment Period include PASI90, PASI100, and IGA at Week 24 and Week 56.

In order to differentiate between subjects remaining on Q4W dosing from those switching to Q8W dosing at Week 16, the treatment comparisons at Week 24 for PASI100, PASI90

and IGA will be performed in 2 different ways using the following randomized treatment arms:

- 1. Bimekizumab Q4W and bimekizumab Q4W/Q8W combined vs adalimumab (testing H<sub>7</sub>, H<sub>8</sub>, and H<sub>9</sub>)
- 2. Bimekizumab Q4W only vs adalimumab (testing H<sub>10</sub>, H<sub>11</sub>, and H<sub>12</sub>)

#### Change #57

#### Section 14.4 Subgroup analyses

Subgroup analyses will be performed on the primary and secondary efficacy variables that are part of the fixed sequence testing procedure described in Section 14.3. The following variables for subgroup analyses will be defined: age, gender, disease duration, region, weight, body mass index (BMI), prior systemic chemotherapy or photochemotherapy, prior biologic exposure, prior systemic therapy of any kind, Baseline disease severity, and antibody positivity. These summaries will be based on imputed data (NRI) and will include descriptive statistics only.

### Has been changed to:

Subgroup analyses will be performed on the primary and secondary efficacy variables that are part of the fixed sequence testing procedure described in Section 14.3. The following variables for subgroup analyses will be defined: age, gender, disease duration, region, weight, body mass index (BMI), prior systemic chemotherapy or photochemotherapy phototherapy, prior biologic exposure, prior systemic therapy of any kind, Baseline disease severity, and antibody positivity. These summaries will be based on imputed data (NRI) and will include descriptive Section 14.5.2 Pharmacokinetic analyses

The following text has been directly and the second of the

The relationship between efficacy response (PASI/IGA) and bimekizumab plasma concentration will be explored via graphical and a model based approach to quantify the time course of dose/exposure response. In addition, the relationship between safety and exposure will also be explored. The data will be combined with that from other bimekizumab trials in PSO for a pooled, cross trial analysis. The details of this analysis will be described in a data analysis plan, and the analysis itself will be reported separately from the Clinical Study Report (CSR). The details of the model and the approach will be specified in a data analysis plan.

Change #59

### **Section 14.6 Handling of protocol deviations**

Important protocol deviations are deviations from the protocol which potentially could have a meaningful impact on study conduct, or on the primary efficacy, key safety, or PK/PD outcomes for an individual subject.

. omes

A state of the state of


### 19 DECLARATION AND SIGNATURE OF INVESTIGATOR

I confirm that I have carefully read and understood this protocol and agree to conduct this clinical study as outlined in this protocol, according to current Good Clinical Practice and local laws and requirements.

I will ensure that all subInvestigators and other staff members read and understand all aspects of this protocol.

I have received and read all study-related information provided to me.

The objectives and content of this protocol as well as the results deriving from it will be treated confidentially, and will not be made available to third parties without prior authorization by UCB.

All rights of publication of the results reside with UCB, unless other agreements were made in a separate contract.

| Investigator: | eation and all. |
|---|---|
| Printed name | Date/Signature |
| et any mar | ELV de la company de la compan |
| , be used to suppor | |
| Printed name Printed name Printed name Any mail This document cannot be used to support any mail | |

This document compate bearing to support any manual respectively.


# **Approval Signatures**

| Version: | 1.0 | |
|---|---|---|
| Document Number: | CLIN-000116785 | 6 |
| Title: | PS0008 Protocol Amendme | ent 2 yajiahle |
| Approved Date: | 11 Apr 2018 | ent 2 The Approvals |
| | | exensi |
| | | adand |
| | | tion are |
| | Documen | t Approvals |
| Approval | | Name Christopher Cioffi |
| Verdict: Approved | | Date of Signature: 11-Apr-2018 12:41:40 GMT+0000 |
| Approval | SUPPORT any marketing aut | Name: Nancy Cross<br>Capacity: Clinical |
| verdict. Approved | aketh | Date of Signature: 11-Apr-2018 12:57:27 GMT+0000 |
| Approval<br>Verdict: Approved | and mic | Name: Jackie Thirlwell<br>Capacity: Clinical |
| V616.101.14 | ~0/X,0. | Date of Signature: 11-Apr-2018 13:43:25 GMT+0000 |
| *( | ENK, | |
| ised to | | |
| * PE | | |
| allino | | |
| - Olit Co | | |
| cume | | |
| ) | | |